#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma

Compound Number : GSK3772847

Effective Date : 27-MAR-2019

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2017N311825 02.
- This RAP is intended to describe the Efficacy, Safety, PK, PD and Biomarker analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the End of Treatment Phase (ETP) and Statistical Analysis Complete (SAC) deliverable.
- This study does have an internal safety review committee (iSRC) and all details of iSRC deliverable are documented in a separate iSRC RAP.

#### Author's Name and Functional Area:

| Approver | | Date |
|------------------|--------------------------------------------|--------------|
| PPD | | 20.34.7.2010 |
| Principal Statis | stician (Respiratory, Clinical Statistics) | 20-MAR-2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations** (Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Investigation Lead (Respiratory, HUP Clinical | 20-MAR-2019 |
| Development) | |
| Principal Programmer (Respiratory, Clinical Programming) | 22-MAR-2019 |
| PPD PPD | |
| Clinical Development Physician (Respiratory, MDC Global Clinical) | 25-MAR-2019 |
| PPD | |
| Scientist (Respiratory, Patient Centred Outcomes, Value Evidence and Outcomes) | 22-MAR-2019 |
| PPD | 20-MAR-2019 |
| Director (Respiratory, Value Evidence and Outcomes) | 20-WAK-2019 |
| Senior Director (Respiratory, Clinical Pharmacology Modelling and Simulation) | 22-MAR-2019 |
| PPD | |
| Director of Clinical Development (Respiratory, MDC Global Clinical) | 26-MAR-2019 |
| Senior Scientific Director (Respiratory, RD AI DPU Head) | 25-MAR-2019 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---------------------------------------------------------------|-------------|
| Senior Statistics Director (Respiratory, Clinical Statistics) | 27-MAR-2019 |
| Programming Manager (Respiratory, Clinical Programming) | 27-MAR-2019 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUC | TION | 6 |
| 2. | SUMMARY | OF KEY PROTOCOL INFORMATION | 7 |
| ۷. | | nges to the Protocol Defined Statistical Analysis Plan | |
| | | Amendments | |
| | 2.3. Study | y Objective(s) and Endpoint(s) | 11 |
| | 2.4. Study | y Design | 14 |
| | | stical Hypotheses | |
| | | ple Size Calculations | |
| 3. | PI ANNED A | NALYSES | 16 |
| ٥. | | of Treatment Phase Analyses | |
| | | Analyses | |
| 4. | ANIAI VOIC I | POPULATIONS | 17 |
| 4. | | ocol Deviations | |
| | 4.1. PIOIC | Deviations | 10 |
| 5. | | ATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | DNS | |
| | | y Treatment & Sub-group Display Descriptors | |
| | | line Definitions | |
| | | centre Studies | |
| | | nination of Covariates, Other Strata and Subgroups | |
| | 5.4.1 | | |
| | | ple Comparisons and Multiplicity | 22 |
| | | r Considerations for Data Analyses and Data Handling rentions | 22 |
| 6. | STUDY POF | PULATION ANALYSES | <mark>23</mark> |
| | 6.1. Over | view of Planned Study Population Analyses | 23 |
| | 6.2. Dispo | osition | <mark>23</mark> |
| | 6.3. Medi | cal Conditions | 23 |
| | 6.4. Cond | comitant Medications | 23 |
| 7. | EFFICACY A | ANALYSES | 24 |
| • • | | ary Efficacy Analyses | |
| | 7.1.1 | , , , | |
| | 7.1.2 | · | |
| | 7.1.3 | | |
| | 7.1.4 | · | |
| | 7.1.5 | • | |
| | 7.1.0 | 7.1.5.1. Statistical Methodology Specification | 25 |
| | 7.2. Seco | ndary Efficacy Analyses | |
| | 7.2.1 | | 29 |
| | 7.2.2 | | |
| | 7.2.3 | • | |
| | 7.2.4 | | |
| | 1.2.7 | 7 2 4 1 Statistical Methodology Specification | |

| 8. SAFETY ANALYSES 36 8.1. Adverse Events Analyses 36 8.2. Adverse Events of Special Interest Analyses 36 8.3. Vital Signs, Electrocardiogram (ECG) and Holter 36 8.4. Clinical Chemistry, Haematology and Cardiac Markers 36 8.5. Antibodies 37 8.6. Clinical Laboratory Analyses 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2.1. Endpoint / Variables <td< th=""><th></th><th></th><th>CONFIDENTIAL</th><th>207597</th></td<> | | | CONFIDENTIAL | 207597 |
|---|---|---|---|---|
| 8.1. Adverse Events Analyses 36 8.2. Adverse Events of Special Interest Analyses 36 8.3. Vital Signs, Electrocardiogram (ECG) and Holter 36 8.4. Clinical Chemistry, Haematology and Cardiac Markers 36 8.5. Antibodies 37 8.6. Clinical Laboratory Analyses 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endopint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2.1 Endpoint / Variables 40 10.2.2 Summary Measure 40 10.2.1 Endpoint / Variables 40 10.2.2 Summary Measure 40 10.2.3 Population of Interest 40 | 8. | SAFE | TY ANALYSES | 36 |
| 8.2. Adverse Events of Special Interest Analyses 36 8.3. Vital Signs, Electrocardiogram (ECG) and Holter 36 8.4. Clinical Chemistry, Haematology and Cardiac Markers 36 8.5. Antibodies 37 8.6. Clinical Laboratory Analyses 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1. Eccondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.4. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.1. Endpoint / Variables 40 10.2.2. Suma | 0. | | | |
| 8.3. Vital Signs, Electrocardiogram (ECG) and Holter 36 8.4. Clinical Chemistry, Haematology and Cardiac Markers 36 8.5. Antibodies 37 8.6. Clinical Laboratory Analyses 37 9. PHARMACOKINETIC ANALYSES 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1. Endpoint / Variables 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Stati | | - | | |
| 8.4. Clinical Chemistry, Haematology and Cardiac Markers | | | | |
| 8.5. Antibodies 37 8.6. Clinical Laboratory Analyses 37 9. PHARMACOKINETIC ANALYSES 37 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1.1 Secondary Pharmacodynamic Analyses 38 10.1.2 Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2.1 Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.2. | | | | |
| 8.6. Clinical Laboratory Analyses | | | | |
| 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2. Exploratory Biomarker Analyses / Methods 38 10.2. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.1. Appendix 2: Schedule of Activities 43 12.2. Appendix 3: Assessment Windows 49 12.3. Appendix 4: Study Phases and Treatment Emergent Adverse Events 50 | | | | |
| 9.1. Secondary Pharmacokinetic Analyses 37 9.1.1. Endpoint / Variables 37 9.1.2. Population of Interest 37 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2. Exploratory Biomarker Analyses / Methods 38 10.2. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.1. Appendix 2: Schedule of Activities 43 12.2. Appendix 3: Assessment Windows 49 12.3. Appendix 4: Study Phases and Treatment Emergent Adverse Events 50 | 9 | PHAR | RMACOKINETIC ANALYSES | 37 |
| 9.1.1. Endpoint / Variables | ٥. | | | |
| 9.1.2. Population of Interest | | 0 | · | |
| 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events 37 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Events 40 10.2.3. Population of Intercurrent (Post-Randomisation) Events 40 10.2.4. Strategy for Intercurrent (Post-Randomi | | | | |
| 9.1.4. Statistical Analyses / Methods 37 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES 38 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.2. Exploratory Biomarker Analyses / Methods 38 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.1. Appendix 2: Schedule of Activities 43 12.2. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 < | | | | |
| 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1 Endpoint / Variables 38 10.1.2 Summary Measure 38 10.1.3 Population of Interest 38 10.1.4 Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5 Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1 Endpoint / Variables 40 10.2.2 Summary Measure 40 10.2.3 Population of Interest 40 10.2.4 Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5 Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.1 Appendix 2: Schedule of Activities 43 12.2.1 Protocol Defined Schedule of Events 43 12.3.1 Definitions of Assessment Windows 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1 Study Phases 50 | | | | |
| 10.1. Secondary Pharmacodynamic Analyses 38 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. Appendix 1: Protocol Deviation Management 42 12.1. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3.1. Definitions of Assessment Windows 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | 10 | ДЦΛД | MACODYNAMIC AND BIOMARKER ANALYSES | 38 |
| 10.1.1. Endpoint / Variables 38 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | 10. | | | |
| 10.1.2. Summary Measure 38 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | 10.1. | | |
| 10.1.3. Population of Interest 38 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | | · | |
| 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events 38 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2. Appendix 3: Assessment Windows 49 12.3. Appendix 3: Assessment Windows 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | | | |
| 10.1.5. Statistical Analyses / Methods 38 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | | | |
| 10.2. Exploratory Biomarker Analyses 40 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | | · | |
| 10.2.1. Endpoint / Variables 40 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | 10.2 | · | |
| 10.2.2. Summary Measure 40 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases 50 | | 10.2. | · | |
| 10.2.3. Population of Interest 40 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events 40 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events 50 12.4.1. Study Phases 50 | | | The state of the s | |
| 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events. 40 10.2.5. Statistical Analyses / Methods. 40 11. REFERENCES. 41 12. APPENDICES. 42 12.1. Appendix 1: Protocol Deviation Management. 42 12.2. Appendix 2: Schedule of Activities. 43 12.2.1. Protocol Defined Schedule of Events. 43 12.3. Appendix 3: Assessment Windows. 49 12.3.1. Definitions of Assessment Windows for Analyses. 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse 50 12.4.1. Study Phases. 50 | | | • | |
| 10.2.5. Statistical Analyses / Methods 40 11. REFERENCES 41 12. APPENDICES 42 12.1. Appendix 1: Protocol Deviation Management 42 12.2. Appendix 2: Schedule of Activities 43 12.2.1. Protocol Defined Schedule of Events 43 12.3. Appendix 3: Assessment Windows 49 12.3.1. Definitions of Assessment Windows for Analyses 49 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events 50 12.4.1. Study Phases 50 | | | • | |
| 12. APPENDICES4212.1. Appendix 1: Protocol Deviation Management4212.2. Appendix 2: Schedule of Activities4312.2.1. Protocol Defined Schedule of Events4312.3. Appendix 3: Assessment Windows4912.3.1. Definitions of Assessment Windows for Analyses4912.4. Appendix 4: Study Phases and Treatment Emergent Adverse5012.4.1. Study Phases50 | | | | |
| 12.1. Appendix 1: Protocol Deviation Management4212.2. Appendix 2: Schedule of Activities4312.2.1. Protocol Defined Schedule of Events4312.3. Appendix 3: Assessment Windows4912.3.1. Definitions of Assessment Windows for Analyses4912.4. Appendix 4: Study Phases and Treatment Emergent Adverse5012.4.1. Study Phases50 | 11. | REFEI | RENCES | 41 |
| 12.1. Appendix 1: Protocol Deviation Management4212.2. Appendix 2: Schedule of Activities4312.2.1. Protocol Defined Schedule of Events4312.3. Appendix 3: Assessment Windows4912.3.1. Definitions of Assessment Windows for Analyses4912.4. Appendix 4: Study Phases and Treatment Emergent Adverse5012.4.1. Study Phases50 | 40 | ۸۰۰۰۰ | NDICEC | 40 |
| 12.2. Appendix 2: Schedule of Activities4312.2.1. Protocol Defined Schedule of Events4312.3. Appendix 3: Assessment Windows4912.3.1. Definitions of Assessment Windows for Analyses4912.4. Appendix 4: Study Phases and Treatment Emergent Adverse5012.4.1. Study Phases50 | 12. | 40.4 | | |
| 12.2.1. Protocol Defined Schedule of Events | | | | |
| 12.3. Appendix 3: Assessment Windows | | 12.2. | | |
| 12.3.1. Definitions of Assessment Windows for Analyses | | 40.0 | | |
| 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events | | 12.3. | | |
| Events | | 10.4 | | 49 |
| 12.4.1. Study Phases50 | | 1∠.4. | | 50 |
| • | | | | |
| 17.4.1.1 Study Phases for Concomitant Medication 51 | | | 12.4.1.1 Study Phases for Concomitant Medication | |
| 12.4.2. Treatment Emergent Flag for Adverse Events51 | | | | |

Appendix 5: Data Display Standards & Handling Conventions.......52

Appendix 6: Derived and Transformed Data ......54

Appendix 7: Reporting Standards for Missing Data......59

General 54
Study Population 54

Efficacy......56

Safety ......57

Premature Withdrawals......59

12.5.

12.6.

12.5.1.

12.5.2.

12.6.1.

12.6.2. 12.6.3.

12.6.4.

12.7.1.


| | 1272 | Handling of Missing Data | 50 |
|---|---|---|---|
| | 12.1.2. | 12.7.2.1. Handling of Missing and Partial Dates | |
| 12.8. | Annendi | x 8: Values of Potential Clinical Importance | |
| 12.9. | | x 9: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 12.10. | | x 10: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | 12.10.6. | Efficacy Figures | 70 |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | |
| | 12.10.9. | Pharmacodynamic and Biomarker Tables | <b>7</b> 8 |
| | 12.10.10 | ).Pharmacokinetic Figures | <b>7</b> 9 |
| | | Pharmacodynamic and Biomarker Figures | |
| | | 2.ICH Listings | |
| | 12.10.13 | B. Non-ICH Listings | 85 |
| 12 11 | Annendi | v 11. Evample Mock Shells for Data Displays | 99 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 207597:

| Protocol Revision Chronology: | | |
|---|---|---|
| 2017N311825_00 | 2017-MAR-06 | Original |
| 2017N311825_01 | 2017-JUN-02 | To address clarifications regarding the aim of the study, the eligibility criteria, the schedule of activities, the clinical assessments, and the recording of lab data and adverse events. The benefit: risk section was also updated based on the Part 2 results from study CNTO7160ASH1001. Also, a few typographical errors were corrected. |
| 2017N311825_02 | 2017-SEP-13 | To add more information on the risk: benefit section and the study design justification sections. To address clarifications regarding the unblinding of treatment in case of emergency. To clarify that rechallenge is not allowed once the treatment discontinuation criteria are met. Also, a few typographical errors were corrected. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Modified Intent to Treat population. | Modified Intent to Treat (Loss of Control), Modified Intent to Treat and Safety excluding GCP noncompliant subjects populations. | The Modified Intent to Treat (Loss of Control) was added to account for the intercurrent event when participants receive the wrong study treatment. Whilst the data from GCP noncompliant participants should not be used in the efficacy analysis, the participants were dosed with GSK3772847 or Placebo so all safety data (AEs, SAEs, ECGs etc.) should be reported. |
| Section 10.4.1 of the protocol describes a sensitivity analysis where data is analysed as missing and worst case (loss of control) for participants who withdraw from the study for reasons other than loss of asthma control. | A primary and secondary estimand have been defined to capture where data is analysed as missing and worst case (loss of control) for various intercurrent events where participants withdraw from the study for reasons other than loss of asthma control. | The protocol was approved before the ICH E9 addendum on estimands. The RAP is performing the same planned analysis as detailed in the Protocol however the terminology has been updated in accordance with ICH E9. |
| Statistical analysis would be performed for each screening eosinophil strata separately. | Bayesian analysis will include screening eosinophil strata as a covariate instead of performing split analysis models. In addition, an exploratory analysis using fractional polynomials was added to examine the relationship between loss of control and screening eosinophils (continuous), IgE and FeNO. | Bayesian analysis will now include the same covariates as the frequentist analysis. By modelling eosinophils as a continuous endpoint, it will provide more information on the impact of varying screening eosinophil levels on the treatment effect. It will also provide additional information on the role of IgE and FeNO on loss of asthma control. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Mixed model repeated measures will be used to analyse the following endpoints. The baseline value of each endpoint will be included along with baseline*visit and treatment*visit interactions. Treatment differences, 95% confidence intervals and p-values will be presented. Change from baseline in ACQ-5 absolute score Change from baseline in SGRQ total score Change from baseline in Pre-bronchodilator FEV <sub>1</sub> Change from baseline in FeNO | FEV <sub>1</sub> and FeNO will only be analysed up until Week 4 (down titration of ICS), all data post Week 4 will be summarised descriptively only. In addition, an exploratory analysis using fractional polynomials was added to examine the relationship between FEV <sub>1</sub> at Week 4 with screening eosinophils (continuous), IgE and FeNO. Continuous ACQ-5 and SGRQ will only be summarised and will not be analysed. | FEV <sub>1</sub> and FeNO are impacted by ICS, so including change from baseline post-down titration of ICS would be confounding change due to study treatment with change due to ICS. To better explore the data prior to down titration, the fractional polynomial analysis has been added to examine the relationship between FEV <sub>1</sub> at Week 4 with screening eosinophils (continuous), IgE and FeNO. FEV1, FeNO, ACQ-5 and SGRQ analysed using an MMRM would be assuming that |
| | | data is missing at random. In fact, participants could have withdrawn due to loss of asthma control which is related to study treatment, so the analysis assumptions would not have been valid. |
| Secondary endpoints listed as: Serum concentrations of GSK3772847 at weeks 2, 4, 8, 12, 16, 20, 24 and 28. Free and total soluble ST2 levels at weeks 2, 4, 8, 12, 16, 20, 24 and 28. | Secondary endpoints listed as: Serum concentrations of GSK3772847 by nominal time. Free and total soluble ST2 levels in serum by nominal time. | Endpoint updated to use nominal time so that all data collected is summarised. |
| Proportion of participants with loss of asthma control assessed over Weeks 0-16 only. | Proportion of participants with loss of asthma control assessed over Weeks 0-16 and over Weeks 0-6. | An additional endpoint assessing loss of control between Weeks 0 and 6 was added to help support the time to loss of asthma control analysis. |
| The posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.5 and 0.2 (i.e. more than a 0%, 25%, 50% and 80% reduction) will be produced. | The posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.7, 0.5 and 0.2 (i.e. more than a 0%, 25%, 30%, 50% and 80% reduction), and greater than 0.6 (i.e. less than a 40% reduction) will be produced. | The additional posterior probabilities of the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo being <0.70 (more than a 30% reduction) and >0.60 (less that a 40% reduction) were added to assist internal decision making. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| <ul> <li>Proportion of participants with a ≥0.5 point ACQ-5 score increase from baseline.</li> <li>Proportion of participants who have pre-bronchodilator FEV1 decrease from baseline (measured at the end of Run-in) &gt;7.5 %.</li> <li>Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the pre-defined schedule.</li> <li>Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).</li> <li>Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule</li> <li>Proportion of participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16.</li> <li>Proportion of St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16.</li> </ul> | Endpoints to be summarised and not analysed. | Due to participants being withdrawn after they reach one component of loss of control, there is no information available for the other components/ ACQ-5/SGRQ after this date. As a result the numbers of the subjects who have useable data are very small, and any estimates will be biased, so informative decisions can't be made. The data must still be summarised to comply with disclosure rules for pre-specified secondary endpoints. |
| The minimum detectable effect for the sample size calculations is reported as 31% corresponding to a proportion with loss of control on GSK3772847 of 28%. | The minimum detectable effect for the sample size calculations is reported as 36% corresponding to a proportion with loss of control on GSK3772847 of 28%. | A typographical error in the protocol which meant that minimum detectable effect was incorrectly reported as 31%, this has been corrected in the RAP. |

# 2.2. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Pla | Reporting and Analysis Plan_207597_Final_V01 [20-DEC-2018] |
| Reporting and Analysis Pla | n_207597_Amendment_Final_V01 |
| Analysis of components of loss of asthma control and responder analysis | Analysis of components of loss of asthma control and responder analysis were removed as explained in Section 2.1. |
| | Additional information provided on the Bayesian logistic regression including starting values, set seeds and thinning options. |
| Bayesian Analysis | The posterior probabilities of the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo being <0.70 (more than a 30% reduction) and >0.40 (less that a 40% reduction) were added to assist internal decision making. |
| Repeated Measures<br>Analysis | Information on the variance-covariance matrix and use of the OM option added. |
| Treatment Discontinuation Date | Derivation added for treatment discontinuation date |
| Sample Size | A typographical error in the protocol which meant that minimum detectable effect was incorrectly reported as 31%, this has been corrected in the RAP amendment. |
| Tables, Listings and Figures | Minor clarification/typographical errors in output titles and associated RAP text were added. |

# 2.3. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of GSK3772847, compared with placebo, administered intravenously every 4 weeks for 12 weeks (Week 0 – Week 12, 4 doses in total) in participants with moderately severe asthma. | <ul> <li>Primary – Proportion of participants with loss of asthma control over Weeks 0-16 where 'loss of asthma control' is defined as at least one of the following: <ul> <li>Asthma Control Questionnaire (ACQ-5) score increase from baseline (measured at the end of Run-in) ≥ 0.5 point or</li> <li>Pre-bronchodilator Forced expiratory volume in 1 second (FEV1) decrease from baseline (measured at the end of Run-in) &gt;7.5 % or</li> <li>Inability to titrate inhaled corticosteroid according to the pre-defined schedule or</li> <li>A clinically significant asthma exacerbation (requiring oral corticosteroid [OCS] and/or hospitalisation).</li> </ul> </li> </ul> |
| Secondary | / |
| To evaluate other aspects of efficacy of GSK3772847 compared with placebo in participants with moderately severe asthma. | <ul> <li>Other efficacy endpoints (at or by Week 16):</li> <li>Proportion of participants with a ≥0.5 point ACQ-5 score increase from baseline.</li> <li>Proportion of participants who have prebronchodilator FEV1 decrease from baseline (measured at the end of Run-in) &gt;7.5 %.</li> <li>Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the pre-defined schedule.</li> <li>Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).</li> <li>Proportion of participants with loss of asthma control over Weeks 0-6</li> <li>Time to loss of asthma control.</li> <li>Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule</li> <li>The incidence, mean rate, and total number per participant of hospitalisations or Emergency Room (ER) visits during the study treatment period.</li> <li>Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.</li> <li>Proportion of participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to</li> </ul> |

| Objectives | Endpoints |
|---|---|
| - | Week 16. |
| | <ul> <li>Change from baseline in SGRQ total score at<br/>Weeks 4, 8, 12 and 16.</li> </ul> |
| | <ul> <li>Proportion of St. George's Respiratory<br/>Questionnaire (SGRQ) responders (at least a<br/>4 unit improvement from baseline) at Weeks<br/>4, 8, 12 and 16.</li> </ul> |
| | • Change from baseline in pre-bronchodilator FEV1 at Weeks 2, 4, 6, 8, 10, 12, 14, 16. |
| | Change from baseline in mean morning peak expiratory flow (PEF) and mean evening PEF over each four weeks of the 16 week treatment period. |
| | Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period. |
| | <ul> <li>Change from baseline in rescue medication<br/>use (albuterol/salbutamol): mean number of<br/>inhalations per day over each four weeks of<br/>the 16 week treatment period.</li> </ul> |
| | Changes from baseline in night-time awakenings due to asthma symptoms |
| | requiring rescue medication use over each four weeks of the 16 week treatment period. |
| | Change from baseline in fractional exhaled nitric oxide (FeNO) at each week measured. |
| <ul> <li>To evaluate the safety and tolerability of<br/>GSK3772847, compared with placebo<br/>administered intravenously every 4 weeks</li> </ul> | <ul> <li>Incidence and frequency of adverse events<br/>(AEs) and serious adverse events (SAEs).</li> <li>Change from baseline in vital signs at weeks</li> </ul> |
| for 12 weeks (Week 0-12, 4 doses in total) in | 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24 and 28. |
| participants with moderately severe asthma. | <ul> <li>Change between post-dose and pre-dose in<br/>vital signs at weeks 0, 4, 8 and 12.</li> </ul> |
| | <ul> <li>Change from baseline in 12-lead<br/>electrocardiogram (ECG) measurements at<br/>weeks 4, 8, 12 and 16.</li> </ul> |
| | <ul> <li>Change between post-dose and pre-dose in<br/>12-lead ECG measurements at weeks 0, 4,<br/>8 and 12.</li> </ul> |
| | <ul> <li>Change from baseline in 24 hours Holter<br/>measurements at weeks 4 and 12.</li> </ul> |
| | Change from baseline in clinical chemistry at weeks 2, 4, 8, 12, 16 and 28. |
| | <ul> <li>Change from baseline in haematology and<br/>cardiac markers at weeks 1, 2, 4, 6, 8, 10,<br/>12, 14, 16 and 28.</li> </ul> |
| | <ul> <li>Incidence of and titres of anti- GSK3772847<br/>antibodies at weeks 2, 4, 8, 12, 16, 20, 24<br/>and 28.</li> </ul> |


| | Objectives | Endpoints |
|---|---|---|
| • | To evaluate the pharmacokinetics (PK) of GSK3772847 in participants with moderately severe asthma. | Serum concentrations of GSK3772847 by nominal time. |
| • | To evaluate the pharmacodynamics (PD) of GSK3772847 in participants with moderately severe asthma. | Free and total soluble ST2 levels in serum by nominal time. |
| Exp | oloratory | |
| • | To compare the effect of GSK3772847 with placebo on biomarkers in serum and sputum. | <ul> <li>Changes from baseline in induced<br/>sputum biomarkers (subset) at weeks 8<br/>and 16.</li> </ul> |
| | | <ul> <li>Changes from baseline in exploratory<br/>serum markers at weeks 8 and 16.</li> </ul> |

# 2.4. Study Design



| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Interim | The End of Treatment Phase Analysis will take place after all subjects have |
| Analysis | completed the week 16 visit, and will be considered an interim analysis for both efficacy and safety. There will be no modifications to dosing regimens, sample size or any other aspects of the trial based on this data, as all study assessments, apart from follow-up, will have already been completed. |

# 2.5. Statistical Hypotheses

The primary null hypothesis ( $H_0$ ) for this study is that the ratio of the proportions of subjects with loss of asthma control from randomisation to Week 16 between GSK3772847 and placebo is unity.

$$H_0$$
:  $\frac{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ GSK3772847}{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ Placebo}=1$ 

The alternative hypothesis ( $H_1$ ) for this study is that the ratio of the proportions of subjects with loss of asthma control from randomisation to Week 16 between GSK3772847 and placebo is not unity.

$$H_1$$
:  $rac{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ GSK3772847}{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ Placebo} 
eq 1$ 

# 2.6. Sample Size Calculations

With 70 evaluable participants per arm and assuming the true proportion with loss of control on placebo is 44%, the smallest observed difference that would lead to rejection of the null hypothesis (minimum detectable effect) is 36% corresponding to a proportion with loss of control on GSK3772847 of 28%.

As detailed in Section 2.1, there was a typographical error in the protocol which meant that minimum detectable effect was incorrectly reported as 31%, this has been corrected above.

#### 3. PLANNED ANALYSES

# 3.1. End of Treatment Phase Analyses

The End of Treatment Phase Analysis will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the Week 16 visit or the Early Withdrawal visit
- 2. All required database cleaning activities have been completed and database release has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

Due to an inability to lock log forms used for collection of exacerbation data, the end of treatment phase analysis will be considered an interim analysis for both efficacy and safety. Any safety data collected for participants who have completed clinic visits after Week 16 will also be cleaned and included in the analysis.

All participants will have completed the active treatment phase of the study by the time of the interim, so no modifications will be made to the study as a result of the End of Treatment Phase Analysis. The Final Analysis is intended to be an analysis of safety data collected in the Post-treatment Follow-Up phase.

The sponsor will be unblinded to the results of the analysis.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- All subjects have completed the study.
- All required database cleaning activities for data after Week 16/ Early Withdrawal as well as data collected on log pages have been completed.
- Final database release and database freeze has been declared by Data Management.

No unblinding will take place as part of the final analysis as all participants will have already been unblinded during the End of Treatment Phase Analysis.

# 4. ANALYSIS POPULATIONS

Some participants are being excluded from the efficacy analyses due to a failure at their site to follow GCP. As these participants received GSK3772847 or placebo during their period of participation, all safety data will be reported.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | The All Subjects Enrolled (ASE) population<br>will consist of all participants who sign the<br>ICF. | Study population Reason for withdrawal prior to randomisation |
| Randomised | The randomised population will consist of all participants who were randomised. A participant who is recorded as a screen or run-in failure and also randomised will be considered to be randomised in error provided they have not performed any study assessments. | No formal analysis will<br>be performed on this<br>population |
| Modified Intent-to-<br>Treat excluding<br>GCP non-<br>compliant<br>subjects (Loss of<br>Control) | The Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of Control) (mITT_LoC) will consist of all randomised participants who take at least 1 dose of study treatment, excluding participants where an investigation by GSK has shown that good clinical practice has not been followed. Any participants excluded from this population will be identified as protocol deviations and listed in a separate output. Participants will be analysed according to the treatment they receive >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. For loss of asthma control, participants will be analysed according to the treatment they were receiving at the time of loss of control. | •Efficacy (loss of control) |
| Modified Intent-to-<br>Treat excluding<br>GCP non-<br>compliant<br>subjects | The Modified Intent-to-Treat excluding GCP non-compliant subjects (mITT) population will consist of all randomised participants who take at least 1 dose of study treatment, excluding participants where an investigation by GSK has shown that good clinical practice has not been followed. Any participants excluded from this population will be identified as protocol deviations and listed in a separate output. Participants will be analysed according to the treatment they receive | •Efficacy (all except loss of control) |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. | |
| Safety including<br>GCP non-<br>compliant<br>subjects | The Safety (SAFF_ALL) population will consist of all randomised participants who take at least 1 dose of study treatment. Participant will be analysed according to the treatment they receive >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. | Study population Inclusion, exclusion and randomisation criteria deviations Participant disposition Safety |
| Pharmacokinetic | The PK population will consist of all randomised participants who received at least one dose of study medication, and for whom at least one pharmacokinetic sample was obtained, analysed and was measurable. | ●PK |

#### NOTES:

- 1. Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.
- 2. If a participant is inadvertently given both study treatments they will be analysed according to the treatment that they received the more frequently.

#### 4.1. Protocol Deviations

All important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [21-Aug-2017 (Version 1) or later].

- ➤ Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- ➤ This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Note: Inclusion and exclusion criteria deviations are always reported as important.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|------|----------------------------------------|-----------------------|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description Order [1] | |
| G | GSK3772847 10 mg/kg | GSK3772847 | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

• Order represents treatments being presented in TFL, as appropriate.

Treatment comparisons will be displayed as follows using the descriptors as specified:

• GSK3772847 vs Placebo

There were four strata used for the randomisation depending on the participants baseline blood eosinophil count and whether they consented to the sputum sub-study:

- Sputum sub-study and screening blood eosinophils < 150 cells/μL
- Sputum sub-study and screening blood eosinophils  $\geq$ =150 cells/ $\mu$ L
- Not sputum sub-study and screening blood eosinophils < 150 cells/μL
- Not sputum sub-study and screening blood eosinophils  $\geq 150 \text{ cells/}\mu\text{L}$

Displays will be presented by combining data across all four strata to give the overall estimate of GSK3772847 versus placebo.

Sputum sub-study will not be accounted for within the statistical analysis as the sputum sub-study strata was for monitoring recruitment only.

An additional exploratory analysis using fractional polynomials has been added to further investigate the relationship between loss of control and screening eosinophils and summary statistics on eosinophils will also be provided.

# 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Pre-<br>Screening | Screen<br>Run-in | Day 1<br>(Pre-Dose) | |
| Loss of Asthma Control | | | | |
| Pre-bronchodilator Forced expiratory volume in 1 second (FEV <sub>1</sub> ) | | X | Х | Day 1 |
| Asthma Control Questionnaire (ACQ-5) score | | Χ | Х | Day 1 |
| Other Patient Reported Outcomes | 3 | | | |
| St. George's Respiratory<br>Questionnaire (SGRQ) | | | Х | Day 1 |
| Peak Expiratory Flow (PEF) | | | | |
| Mean morning peak expiratory flow (PEF) | | Χ | X | Run-in [1] |
| Mean evening peak expiratory flow (PEF) | | Χ | Х | Run-in [1] |
| Fractional Exhaled Nitric Oxide (F | eNO) | | | |
| Fractional Exhaled Nitric Oxide (FeNO) | | | Х | Day 1 |
| Symptom Scores | | | | |
| Mean daytime asthma symptom score | | Х | Х | Run-in [1] |
| Night-time awakenings due to asthma symptoms requiring rescue medication | | X | Х | Run-in [1] |

| Parameter | Study Assessments<br>Considered As Baseline | | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Pre-<br>Screening | Screen<br>Run-in | Day 1<br>(Pre-Dose) | |
| Rescue Medication | | | | |
| Rescue medication use | | Х | Х | Run-in [1] |
| Mean number of inhalations per day over each four weeks | | Х | Х | Run-in [1] |
| Safety | | | | |
| Vital Signs | | Х | Х | Day 1 |
| 12-lead Electrocardiogram (ECG) measurements | | Х | Х | Day 1 |
| 24 hours Holter measurements | | Х | | Screen/Run in |
| Clinical laboratory tests (haematology and chemistry) | | Х | Х | Day 1 |
| Biomarkers | | | | |
| Induced sputum biomarkers | | | Х | Day 1 |
| Serum biomarkers | | | Х | Day 1 |
| Exploratory serum markers | | | Х | Day 1 |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- [1] Mean over the last 7 days of the run-in period prior to V2. Participants must have at least 4 full days of data (morning and evening) in the last 7 days of run-in to be eligible.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site, country, and regions.

| Region | Countries |
|----------------|-----------------------------|
| North America | United States, Canada |
| Latin America | Mexico |
| Eastern Europe | Ukraine, Russian Federation |
| Oceania | Australia |

# 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Covariates |
|---|---|
| Screening eosinophils | At randomisation participants are stratified according to their screening peripheral blood eosinophil count. Screening eosinophils will be included in both primary and secondary analysis as a categorical variable (<150 cells/µL, >=150 cells/µL). |
| | If the analysis models are unable to converge due to low number of participants with screening blood eosinophils <150 cells/µL, then screening eosinophil will be re-categorised according to a cut point of 300 cells/µL instead i.e. <300 cells/µL and >=300 cells/µL |

# 5.5. Multiple Comparisons and Multiplicity

As there is a single primary treatment comparison, no adjustment is required for primary comparisons. No adjustments will be made for multiplicity for other endpoints.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety Population including GCP non-compliant subjects population (SAFF\_ALL), unless specified to be on the All Subjects Enrolled (ASE) population.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

# 6.2. Disposition

The study population summary will use the All Subjects Enrolled (ASE) population and show the number of subjects overall who were enrolled, the number of screen failures and the number with each reason for screen failure. It will also show the number of subjects who were randomised and who were in the modified Intent-to-treat (Loss of Control), modified Intent-to-treat, Safety including GCP non-compliant subjects, and PK populations.

For the Safety including GCP non-compliant subjects, reasons for withdrawal summary will show the number and percentage of subjects who completed the study, who withdrew prematurely from the study and who reported each primary and sub-reason for withdrawal.

#### 6.3. Medical Conditions

The number and percentage of subjects reporting each current medical condition will be presented. This table will include a subheading of 'Cardiovascular Disorders,' which will summarise the information taken from the cardiac disorders page in the eCRF. All medical conditions must be summarised on this table regardless of frequency. This will be repeated for past medical conditions.

#### 6.4. Concomitant Medications

Non-Asthma medications will be summarised by Anatomical-Therapeutic-Chemical (ATC) level 1 and ingredient. Asthma medications will be summarised by the latest version of the Respiratory Medication Class (RMC), and will be derived for each asthma concomitant medication. Multi-ingredient medications will be presented according to their combination ATC classification rather than the classifications of the ingredients.

Asthma and non-asthma medications will be listed separately. A listing of the relationship between ATC Level 1, ingredient and verbatim text will be produced for non-asthma medications only.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint

- Proportion of participants with loss of asthma control over Weeks 0-16
- Proportion of participants with loss of asthma control over Weeks 0-6 (Secondary)

## 7.1.2. Summary Measure

Bayesian Method (Primary): The posterior median and 95% credible interval. In addition, the posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.7, 0.5 and 0.2 (i.e. more than a 0%, 25%, 30%, 50% and 80% reduction), and greater than 0.6 (i.e. less than a 40% reduction).

Frequentist Method (Supportive): Odds Ratio. The odds of having experienced loss of asthma control on GSK3772847 compared to the odds of having experienced loss of asthma control on placebo.

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the modified Intent to Treat (Loss of Control) population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomisation) Events

| Intercurrent Event | Primary Estimand | Secondary Estimand |
|---|---|---|
| Study treatment<br>discontinuation due to an<br>AE/SAE | Excluded from analysis | Set as loss of asthma control (i.e. worst case scenario). |
| Death | Excluded from analysis | Set as loss of asthma control (i.e. worst case scenario). |
| Prohibited/ Concomitant medications that could impact patients' asthma control | Use data as is. | Set as loss of asthma control (i.e. worst case scenario). |
| Non-compliance with FP/SAL, FP or study titration | Use data as is. | Set as loss of asthma control (i.e. worst case scenario). |
| Missing data * | Excluded from analysis | Set as loss of asthma control (i.e. worst case scenario). |

#### Notes:

\* Missing data is not an intercurrent event, however missing values will be imputed according to the estimand under investigation.

- If the intercurrent event occurs after loss of asthma control then all information on loss of asthma control will be used.
- Prohibited/ concomitant medications will be identified as protocol deviations within the prohibited/ concomitant medications category and will have text that start with "LoAC"
- Non-compliance FP/SAL, FP or study titration will be identified as compliance <80%, compliance
  ≥ 120% or protocol deviations within the other deviations related to wrong study
  treatment/administration/dose sub-category and will have text that starts with "TIT"</li>

If any of the following intercurrent events occurs, then all data will be accepted:

Pregnancy
 Accidental unblinding

Whilst it's possible that site staff were unable to administer study drug as they were unable to find a suitable vein, the team felt this would not be caused by the randomised study treatment and the visit would be rescheduled. Therefore, if this occurs all data will be accepted and treated as any other out of window assessment.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Proportion of participants with loss of asthma control over Weeks 0-16
- Proportion of participants with loss of asthma control over Weeks 0-6 (Secondary)

#### **Model Specification**

• The primary endpoint proportion of subjects with loss of asthma control will be analysed for the Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of Control) population using both Bayesian (primary) and Frequentist (supportive) methods.

Bayesian Method (Primary):

- A logistic regression model within proc MCMC will be used to generate the posterior distribution of the ratio of GSK/Placebo.
- The analysis model will include categorical variables for treatment and screening eosinophil strata, with each coefficient (including the intercept) having a non-informative normal(mean=0,var=1x10<sup>6</sup>) prior.
- Odds ratios generated from the model will be back-transform to produce the probability of experiencing loss of asthma control on both GSK3772847 and Placebo. From these estimates the ratio of loss of asthma control on GSK/Placebo will be calculated within the proc MCMC call.

• Three Markov chain Monte Carlo (MCMC) chains will be run, with all parameters in the model being assessed for convergence. This is done to ensure that the results are not sensitive to the initial values selected. The chain with the lowest deviance information criteria (DIC) will be used for the analysis output. Each chain will have 100,000 simulations, with a thinning of 10 and a burn-in of 500, in order to generate 10,000 samples per chain. This may be adjusted if the chains fail to converge. The starting seeds and initial values for all three chains are given below:

| | Set Seed | Starting Value |
|---------|----------|----------------|
| Chain 1 | 2075971 | -2 |
| Chain 2 | 2075972 | 0 |
| Chain 3 | 2075973 | 2 |

- The posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.7, 0.5 and 0.2 (i.e. more than a 0%, 25%, 30%, 50% and 80% reduction), and greater than 0.6 (i.e. less than a 40% reduction) will be calculated, along with the estimated median ratio and associated 95% credible interval. The 95% credible interval will use the highest posterior density where possible, and if this isn't possible then the 2.5% and 97.5% credible intervals will be reported.
- In addition to summary tables a plot of the cumulative probabilities from the posterior distribution for the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo will be generated.
- This analysis will be repeated for loss of asthma control between Weeks 0 and 6.

#### Frequentist Method (Supportive):

 The proportion of participants with loss of asthma control will be analysed using logistic regression allowing for screening eosinophils strata. It will include fixed effects terms for treatment and screening eosinophil strata.

Fractional Polynomials (Exploratory Analysis for Loss of Control Over Weeks 0-16):

- Screening blood eosinophil count will be transformed using a first order fractional polynomial term, and then a second order fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by transformed eosinophil covariate interaction will also be included in the model to allow the magnitude of the treatment difference to differ by screening eosinophil count.
- The impact of extreme observations are a well-known problem with fraction polynomial modelling. To address this a two-step transformation to "pull-in" extremes and shift the origin away from zero will be used (Royston and Sauerbrei, 2007). The formula to achieve this is given below:

$$g\delta(x) = \delta + (1 - \delta) \frac{g(x) - g(x_{(2)})}{g(x_{(n)}) - g(x_{(2)})}$$

where 
$$g(x) = \left[ \ln \left( \frac{\emptyset\left(\frac{(x-\overline{x})}{s}\right) + \varepsilon}{1 - \emptyset\left(\frac{(x-\overline{x})}{s}\right) + \varepsilon} \right) + \varepsilon^* \right] / (2\varepsilon^*)$$

with: 
$$0 < \delta < 1$$

$$s = 0.01$$

$$s^* = -\ln\left[s/(1+s)\right]$$

$$\bar{x} = n^{-1} \sum x_i$$

$$s = (n-1)^{-1} \sum_{i} \left(x_{(i)} - \bar{x}\right)^2$$

As recommended we shall use  $\varepsilon = 0.01$  and  $\delta = 0.2$ .

- All models (first and second order) will be evaluated and the best fitting model will be selected based on the Akaike information criterion (AIC).
- The selected best fitting model will be used to predict the probability of loss of control by treatment arm along with the corresponding predicted odds ratio by screening eosinophil count. This model will include the observed margins (OM) option which will use the analysis dataset.
- The fit of the model to the raw data will be assessed visually by overlaying a plot of the
  treatment estimates and differences estimated in groups defined by quartiles of screening
  eosinophil counts. Estimates will be plotted against the mean eosinophil count within each
  subgroup.
- The role of baseline immunoglobulin E (IgE) and baseline FeNO (separately) on the
  effectiveness of GSK3772847 with respect to loss of asthma control will be investigated in a
  similar way.

# **Model Checking & Diagnostics**

Bayesian Method (Primary):

- The Markov chain standard error (MCSE) should be compared to the standard deviation of the distribution (SD) to make sure that MCSE/SD ≤ 0.01 for all parameters in the mode.
- The Geweke diagnostic test will be used to check whether the mean estimates have converged by comparing means from the early and later part of the Markov chain using a z-score t-test. Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.
- Gelman & Rubin diagnostic checks should be used to assess if the Markov chains have mixed.
- Visual checks on diagnostic plots will be performed to assess:

- Has the Markov chain settled down?
- Are sufficient simulations being run?
- o Is there sufficient burn-in?
- o Is the effective sample size large enough?

## Frequentist Method (Supportive):

None.

#### **Model Results Presentation**

#### Bayesian Method (Primary):

• The proportions of participants experience loss of asthma control on GSK3772847, Placebo and the ratio of GSK3772847/Placebo will be presented along with their 95% credible interval.

#### Frequentist Method (Supportive):

 The proportion of participants experiencing loss of asthma control on GSK3772847, Placebo and the odds ratio will be presented along with the 95% confidence intervals and p-value. This will be presented for all participants combined.

#### Fractional Polynomials (Exploratory Analysis):

 A plot of the relationship between the probability of experiencing loss of control on each treatment as well as the odds ratio versus continuous eosinophils will be produced.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Endpoint and Summary Measure

| Endpoint | Summary Measure |
|---|---|
| <ul> <li>Individual Components of Loss of Asthma Control: <ul> <li>Proportion of participants with a ≥0.5 point. ACQ-5 score increase from baseline.</li> <li>Proportion of participants who have prebronchodilator FEV1 decrease from baseline (measured at the end of Run-in) &gt;7.5 %.</li> </ul> </li> <li>Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the pre-defined schedule.</li> <li>Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).</li> <li>Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule</li> </ul> | Number and percentage of participants experiencing each component of loss of asthma control (summary statistics only). |
| Time to loss of asthma control. | Mean, median, lower and upper quartiles of time to loss of asthma control, along with probability of experiencing loss of asthma control at each dosing visit. |
| The incidence, mean rate, and total number per participant of Asthma Related hospitalisations or Emergency Room (ER) visits during the study treatment period. | Summary statistics and study treatment exposure (no statistical analysis required). |
| <ul> <li>Responders:</li> <li>Proportion of participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16.</li> <li>Proportion of St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16.</li> </ul> | Number and percentage of participants (summary statistics only) |
| Change from Baseline Analysis: Change from baseline in pre-bronchodilator FEV1 Change from baseline in fractional exhaled nitric oxide (FeNO) | Mean change from baseline (summary statistics only) |

| Endpoint | Summary Measure |
|---|---|
| <ul> <li>Change from Baseline:</li> <li>Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.</li> <li>Change from baseline in SGRQ total score at Weeks 4, 8, 12 and 16.</li> </ul> | Mean change from baseline (summary statistics only) |
| <ul> <li>Change from baseline in mean morning peak expiratory flow (PEF) and mean evening PEF for each four week period of the overall 16 week treatment period.</li> <li>Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period.</li> <li>Changes from baseline in night-time awakenings due to asthma symptoms requiring rescue medication use over each four weeks of the 16 week treatment period.</li> <li>Change from baseline in rescue medication use (albuterol/salbutamol): mean number of inhalations per day over each four weeks of the 16 week treatment period.</li> </ul> | Change from baseline (summary statistics only) |

#### 7.2.2. Population of Interest

The secondary efficacy analyses will be based on the modified Intent to Treat population, unless otherwise specified.

### 7.2.3. Strategy for Intercurrent (Post-Randomisation) Events

For the analysis of time to loss of asthma control, both primary and secondary estimands (Section 7.1.4) will be examined. It is important to assess both estimands as data is missing after withdrawal or loss of asthma control. This could produce biased estimates, as loss of control and therefore missing data is related to study treatment, and so the secondary estimand where missing data is set as non-responders must also be considered.

For all other endpoints, only the primary estimand will be examined. This estimand uses all data as collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.

Once participants experience loss of asthma control and/or withdraw from study treatment they immediately restart their standard of care medication (ICS/LABA). As a

result, any data collected past this point will have been impacted by the standard of care medications and any estimates produced biased by the additional use of ICS/LABA. For this reason, data post withdrawal from study treatment is not included in the on-treatment efficacy analysis.

### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Time to loss of asthma control.

#### Strategy for Intercurrent (Post-Randomisation) Events

Both primary and secondary estimands (Section 7.1.4) will be examined. It is important to
assess both estimands as data is missing after withdrawal or loss of asthma control. This could
produce biased estimates, as loss of control and therefore missing data is related to study
treatment, and so the secondary estimand where missing data is set as non-responders must
also be considered.

#### **Model Specification**

- Time to loss of asthma control will be analysed on the Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of Control) population using Kaplan-Meier analysis (Proc lifetest).
   Within the Kaplan Meier plot participants will either be counted as an event or they will be censored.
- A log rank test will be performed to test for difference between the time to loss of asthma control on Placebo compared with GSK3772847

#### Primary Estimand:

- Events: Participants who experience loss of asthma control during the study
- Censoring: Participants who discontinue investigational product for reasons other than loss of asthma control will be censored at the date of early withdrawal from study treatment.
   Participants who successfully complete the 16 week treatment period will be censored at 113 days (16 weeks + 1 day).

#### Secondary Estimand:

- Events: Participants who experience loss of asthma control during the study or who
  discontinue investigational product for reasons other than loss of asthma control (date of event
  will be set to date of early withdrawal from study treatment).
- Censoring: Participants who successfully complete the 16 week treatment period will be censored at 113 days (16 weeks + 1 day).

Time to event/censoring = Date of event/censoring—Treatment start date + 1. If participants experience multiple reasons for loss of control then the earliest date will be used as described in Section 0.

#### **Model Checking & Diagnostics**

None

#### Model Results Presentation

- Kaplan-Meier plots of the probability of a participant experiencing loss of asthma control by treatment will be produced.
- In addition, a summary table will be produced showing the probability of experiencing loss of asthma control by 4, 8, 12 and 16 weeks along with the median, upper and lower quartiles of time to loss of asthma control on both treatment arms (this will be NA if <50% of participants on a treatment lose control).

#### **Endpoint / Variables**

• Change from baseline in pre-bronchodilator FEV<sub>1</sub> at Weeks 2, 4, 6, 8, 10, 12, 14, 16.

#### Strategy for Intercurrent (Post-Randomisation) Events

Primary estimand only.

#### **Model Specification**

Only data until Week 4 (down titration of ICS) will be analysed, all data post Week 4 will be summarised descriptively only.

Data up to and include Week 4 (down titration of ICS):

A repeated measures model with terms for baseline FEV<sub>1</sub>, treatment, visit and screening eosinophil strata. The model will also include baseline FEV<sub>1</sub> by visit, visit by treatment and screening eosinophil strata by visit interactions.

#### Model Structure:

- The variance-covariance matrix will be assumed unstructured.
- Kenward Roger (KR) method will be used for calculating degrees of freedom. If the analysis
  does not run using the KR method then the residual method will be used instead.
- An observed margins (OM) dataset will be used to derive the LS means using coefficients
  which are based on the subjects used in the analysis. This is a dataset with a row for every
  subject-visit combination that contains all of the covariates. The OM will be at the average
  baseline FEV<sub>1</sub>.

FEV<sub>1</sub> at Weeks 4 Only - Fractional Polynomials (Exploratory Analysis):

 Screening blood eosinophil count will be transformed using a first order fractional polynomial term, and then a second order fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by transformed eosinophil covariate interaction will also be included in the model to allow the magnitude of the treatment difference to differ by screening eosinophil count.

• The impact of extreme observations are a well-known problem with fraction polynomial modelling. To address this a two-step transformation to "pull-in" extremes and shift the origin away from zero will be used (Royston and Sauerbrei, 2007). The formula to achieve this is given below:

$$g\delta(x) = \delta + (1 - \delta) \frac{g(x) - g(x_{(1)})}{g(x_{(n)}) - g(x_{(1)})}$$

where 
$$g(x) = \left[ \ln \left( \frac{\emptyset \left( \frac{(x-\overline{x})}{s} \right) + \varepsilon}{1 - \emptyset \left( \frac{(x-\overline{x})}{s} \right) + \varepsilon} \right) + \varepsilon^* \right] / (2\varepsilon^*)$$

with:  $0 < \delta < 1$ 

$$\varepsilon = 0.01$$

$$\varepsilon^* = -\ln \left[ \varepsilon/(1+\varepsilon) \right]$$

$$\bar{x} = n^{-1} \sum_i x_i$$

$$s = (n-1)^{-1} \sum_{} \left(x_{(i)} - \bar{x}\right)^2$$

As recommended we shall use  $\varepsilon = 0.01$  and  $\delta = 0.2$ .

- All models (first and second order) will be evaluated and the best fitting model will be selected based on the AIC.
- The selected best fitting model will be used to predict FEV<sub>1</sub> by treatment arm along with the
  corresponding predicted difference in FEV<sub>1</sub> by screening eosinophil count. This model will
  include the OM option which will use the analysis dataset.
- The fit of the model to the raw data will be assessed visually by overlaying a plot of the
  treatment estimates and differences estimated in groups defined by quartiles of screening
  eosinophil counts. Estimates will be plotted against the mean eosinophil count within each
  subgroup.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by

obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

• The estimates of the mean and difference for each treatment group from the model will be produced, along with 95% confidence intervals and p-values for treatment comparisons.

#### **Endpoint / Variables**

- Change from baseline in fractional exhaled nitric oxide (FeNO).
- Change from baseline in blood eosinophils

# Strategy for Intercurrent (Post-Randomisation) Events

Primary estimand only.

#### **Model Specification**

Only data until Week 4 (down titration of ICS) will be analysed, all data post Week 4 will be summarised descriptively only. Both FeNO and eosinophils have the ratio of post-baseline values to baseline values log transformed prior to analysis. For FeNO where multiple measurements can be taken at a visit, the data will be log transformed (using the natural logarithm (ln) hereby referred to as log) and the average log transformed value used as the visit value.

#### FeNO Analysis Model:

A repeated measures model with terms for log(baseline FeNO), treatment, visit, screening eosinophil strata and interaction terms for log(baseline FeNO) by visit, treatment by visit and screening eosinophil strata by visit.

#### Eosinophil Analysis Model:

A repeated measures model with terms log(baseline eosinophils), treatment, visit and interaction terms for log(baseline eosinophils) by visit and treatment by visit.

#### Model Structure:

- The variance-covariance matrix will be assumed unstructured.
- Kenward Roger (KR) method will be used for calculating degrees of freedom. If the analysis
  does not run using the KR method then the residual method will be used instead.
- An observed margins (OM) dataset will be used to derive the LS means using coefficients
  which are based on the subjects used in the analysis. This is a dataset with a row for every
  subject-visit combination that contains all of the covariates. The OM will be at the average
  logarithm of baseline FeNO or average logarithm of baseline eosinophils dependent on the
  model.

Due to a large amount of FeNO data being outside the normal range, further analysis of FeNO may be explored.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model

respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

- The estimated treatment ratios together with 95% CIs (back-transformed from the differences on the log-scale) will be produced for each treatment group along with the treatment comparisons and p-values.
- In addition the percentage change from baseline will also be presented where this is calculated as:
  - % change from baseline = (ratio-1)\*100

The following endpoints will be summarised descriptively only. No analysis will be performed and all data will be reported as collected excluding data after which participants had reached loss of asthma control/withdrawn early from study treatment and restarted their standard of care medication (Primary Estimand only), using the modified Intent to Treat population:

- Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.
- Participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16.
- Change from baseline in SGRQ total score at Weeks 4, 8, 12 and 16.
- St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16.
- Change from baseline in mean morning peak expiratory flow (PEF) and mean evening PEF over each four weeks of the 16 week treatment period. Note: Each PEF is taken in triplicate with the maximum value being used.
- Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period.
- Changes from baseline in night-time awakenings due to asthma symptoms requiring rescue medication use over each four weeks of the 16 week treatment period. Note: This is the change from baseline in the average number of nights a participant woke up at least once and had to use their rescue medication.
- Change from baseline in rescue medication use (albuterol/salbutamol): mean number of inhalations per day over each four weeks of the 16 week treatment period.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety including GCP non-compliant subjects population, unless otherwise specified. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and Adverse Events of Special Interest (AESIs) will be based on GSK Core Data Standards.

### 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.

# 8.3. Vital Signs, Electrocardiogram (ECG) and Holter

Summary statistics for vital signs at baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24 and 28 will be produced along with change from baseline summaries for each post baseline timepoint. In addition, the change between post-dose and pre-dose vital signs measurements will be summarised at weeks 0, 4, 8 and 12.

Similar 12-lead electrocardiogram (ECG) measurements at baseline, weeks 4, 8, 12 and 16 will be produced along with change from baseline summaries for each post baseline timepoint, and changes between post-dose and pre-dose in 12-lead ECG measurements at weeks 0, 4, 8 and 12.

24 hour Holter measurements collected at baseline, weeks 0, 4 and 12 will be summarised along with change from baseline at weeks 0, 4 and 12. Only participants with at least 16hrs worth of data will be included in any tables however all data will be listed.

# 8.4. Clinical Chemistry, Haematology and Cardiac Markers

Summaries of clinical chemistry results at baseline, weeks 2, 4, 8, 12, 16 and 28 along with change from baseline for all post-baseline measurements will be produced.

Similarly, haematology and cardiac markers at baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28 along with change from baseline for all post-baseline measurements will also be produced.
#### 8.5. Antibodies

Summaries of the incidence of and titres of anti- GSK3772847 antibodies at weeks 0\*, 2, 4\*, 8\*, 12\*, 16, 20, 24 and 28.

#### 8.6. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of liver function tests will be based on GSK Core Data Standards.

#### 9. PHARMACOKINETIC ANALYSES

Due to the time required to analyse PK samples, no PK outputs will be included in the end of treatment phases analysis.

#### 9.1. Secondary Pharmacokinetic Analyses

#### 9.1.1. Endpoint / Variables

Serum concentrations of GSK3772847 by nominal time.

#### 9.1.2. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

#### 9.1.4. Statistical Analyses / Methods

- No statistical analysis will be performed.
- Serum concentration will be summarised descriptively with summary figures being produced.
- Scatter plots of trough serum concentration vs FeNO, trough serum concentration vs blood eosinophils, and trough serum concentration vs IgE at Week 4 only will also be produced.

<sup>\* =</sup> Pre-dose only

#### 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

#### 10.1. Secondary Pharmacodynamic Analyses

#### 10.1.1. Endpoint / Variables

Free and total soluble ST2 levels in serum

#### 10.1.2. Summary Measure

Free soluble ST2: Summary statistics and percentage change from baseline Total soluble ST2: Summary statistics and percentage change from baseline

Only pre-dose trough sST2 will be used for analysis. Post-dose trough sST2 will be summarised only.

#### 10.1.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the modified Intent to Treat population, unless otherwise specified.

#### 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

#### 10.1.5. Statistical Analyses / Methods

#### **Endpoint / Variables**

- Percentage change from baseline in free sST2 (On-treatment)
- Percentage change from baseline in free sST2 (Post-treatment)
- Percentage change from baseline in total sST2 (On-treatment)
- Percentage change from baseline in total sST2 (Post-treatment)

#### **Strategy for Intercurrent (Post-Randomisation) Events**

No intercurrent events are considered for this endpoint. All data will be used as collected.

#### **Model Specification**

- The ratio of post-baseline sST2 values to baseline sST2 values will be log transformed prior to analysis. Note: Log(post baseline sST2 /baseline sST2) is equivalent to log(post baseline sST2) – log(baseline sST2).
- A repeated measures model with terms for treatment, visit, visit by treatment, the logarithm of baseline sST2, the logarithm of baseline sST2 by visit and screening eosinophil strata will be fitted.

#### Model Structure:

- The variance-covariance matrix will be assumed unstructured.
- Kenward Roger (KR) method will be used for calculating degrees of freedom. If the analysis does not run using the KR method then the residual method will be used instead.

An observed margins (OM) dataset will be used to derive the LS means using coefficients
which are based on the subjects used in the analysis. This is a dataset with a row for every
subject-visit combination that contains all of the covariates. The OM will be at the average
baseline of free sST2 (either On-treatment or Post-treatment according to the model).

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

 The estimated treatment ratios together with 95% CIs (back-transformed from the differences on the log-scale).

#### Fractional Polynomials (Exploratory Analysis)

The role of free sST2 on the effectiveness of GSK3772847 with respect to loss of asthma control will be investigated, using the modified intent to treat (loss of control) population. The number of participants experiencing loss of control will be predicted at each level of baseline free sST2 based on a model including a free sST2 main effect term and an interaction with treatment term.

Baseline free sST2 will be transformed using a first order fractional polynomial term, and then a second order fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by transformed free sST2 covariate interaction will also be included in the model to allow the magnitude of the treatment difference to differ by baseline free sST2.

The impact of extreme observations are a well-known problem with fraction polynomial modelling. To address this a two-step transformation to "pull-in" extremes and shift the origin away from zero will be used (Royston and Sauerbrei, 2007). The formula to achieve this is given below:

$$g\delta(x) = \delta + (1 - \delta) \frac{g(x) - g(x_{(1)})}{g(x_{(n)}) - g(x_{(1)})}$$
where 
$$g(x) = \left[ \ln \left( \frac{\emptyset\left(\frac{(x - \overline{x})}{s}\right) + \varepsilon}{1 - \emptyset\left(\frac{(x - \overline{x})}{s}\right) + \varepsilon} \right) + \varepsilon^* \right] / (2\varepsilon^*)$$
with:  $0 < \delta < 1$ 

$$\varepsilon = 0.01$$

$$\varepsilon^* = -\ln \left[ \varepsilon / (1 + \varepsilon) \right]$$

$$\bar{x} = n^{-1} \sum x_i$$
 $s = (n-1)^{-1} \sum (x_{(i)} - \bar{x})^2$ 

As recommended we shall use  $\varepsilon = 0.01$  and  $\delta = 0.2$ .

All models (first and second order) will be evaluated and the best fitting model will be selected based on the AIC.

The selected best fitting model will be used to predict the probability of loss of control by treatment arm along with the corresponding predicted odds ratio by baseline free sST2. This model will include the OM option which will use the analysis dataset.

The fit of the model to the raw data will be assessed visually by overlaying a plot of the treatment estimates and differences estimated in groups defined by quartiles of baseline free sST2 counts. Estimates will be plotted against the mean baseline free sST2 count within each subgroup.

#### 10.2. Exploratory Biomarker Analyses

#### 10.2.1. Endpoint / Variables

- Changes from baseline in induced sputum biomarkers (subset) at weeks 8 and 16.
- Changes from baseline in exploratory serum markers at weeks 8 and 16.

#### 10.2.2. Summary Measure

Change from baseline

#### 10.2.3. Population of Interest

The exploratory biomarker analyses will be based on the modified Intent to Treat population, unless otherwise specified.

#### 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

#### 10.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Induced sputum biomarkers and exploratory serum markers at weeks 8 and 16 will be summarised using descriptive statistics, including the geometric mean and CV as well as listed.

No statistical analysis will be performed on this data.

#### 11. REFERENCES

Charter for the Internal Safety Review Commitee (iSRC), Protocol 207597 Title: A randomised, double-blind, parallel group, multicenter, stratified study assessing the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with severe asthma, 26 June 2017

GlaxoSmithKline Document Number 2017N311825\_02, Protocol: A randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma, 13 September 2017

Internal Safety Review Commitee (iSRC) Reporting and Analysis Plan for a randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma, 20 July 2018

Protocol Deviation Management Plan (PDMP), Version 01, 21 August 2017

Royston and Sauerbrei, Improving the robustness of fractional polynomial models by preliminary covariate transformation: A pragmatic approach, Computational Statistics & Data Analysis, Volume 51, Issue 9, 15 May 2007, Pages 4240-4253 doi.org/10.1016/j.csda.2006.05.006

Winthrop et al, 2015, Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance, Annals of the Rheumatoid Arthritis Disease, doi: 10.1136/annrheumdis-2015-207841. Epub 2015 Sep 22

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management

The full list of protocol deviations collected on the eCRF is in the PDMP. Please refer to this document for current guidance.

There is no per protocol population in this study.

# 12.2. Appendix 2: Schedule of Activities

#### 12.2.1. Protocol Defined Schedule of Events

| Procedure | Pre-<br>Screen | Scree | | | | Tr | eatme | nt Per | riod | | | | Follo | w-up P | eriod <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ing <sup>1</sup> | n Run-<br>in | 1 | 2 day | s | | | | ± 3 da | ays | | | (± 3 days) | | | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | Pre-screening and screening can occur on the same day FU period to start 4 weeks after ETP or EW visit. |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | 11 J. |
| Informed consent<br>(ICF) | х | | | | | | | | | | | | | | | |
| Genetic ICF | | X | | | | | | | | | | 1.0 | | 4 | | |
| ICF for sputum | | X | 07 | | | | | | | | | | | | | ļ |
| Inclusion and exclusion criteria | | Х | | | | | | | | | | | | | | |
| Randomisation<br>Criteria | | | Х | | | | | | | | | 50 | | | | |
| Demography | X | | | | Ĩ | i i | | | | | | | | | | 1 |
| Full physical exam<br>including height and<br>weight | | х | | | | | | | | | | | | | | |
| Medical history<br>(includes substance<br>abuse) | | х | | | | | | | | | | | | | | Substances [Drugs, Alcohol,<br>tobacco] and family history of<br>premature CV disease]):<br>[including cardiovascular<br>medical history] |

| 2111 | Pre- | Scree | | | | Tr | eatme | nt Pe | iod | | | | Follo | w-up P | eriod <sup>2</sup> | 93.50 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screen<br>ing <sup>1</sup> | n Run- | ± | 2 day | s | | ±3 days | | | | | | | ± 3 day | | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | Pre-screening and screening can occur on the same day FU period to start 4 weeks after ETP or EW visit. |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | <i>j.</i> |
| Laboratory<br>assessments | | X1,2 | יא | x | Χı | Χ¹ | х | Χ¹ | x | Χ¹ | х | X1 | | | Χ¹ | Haematology (including eosinophil count) and cardiac markers measured at all clinic visits. 1. Clinical chemistry (including liver chemistry). 2. Routine urinalysis at screening (Visit 1) |
| Pregnancy test <sup>1</sup> | х | 2 | Хз | | | X3 | | Х3 | | X <sub>3</sub> | | х | Х | х | х | Test for women with child bearing potential. Serum pregnancy test at V0/V1. Test to be performed predose during the treatment period. |
| [HIV, Hep B and Hep<br>C screen] | | х | | | | | | | | | | | | | | A confirmatory negative Hepatitis C RNA test must be obtained, to be able to enrol participants with positive Hepatitis C antibody due to prior resolved disease. If test has been performed within 3 months prior to first dose of study treatment, testing at screening is not required. |

| 400 5 700 | Pre- | Scree | | | | Tr | eatme | nt Pe | riod | | | | Follo | ow-up l | Period <sup>2</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screen<br>ing <sup>1</sup> | n Run- | 1 | 2 day | s | | | | ± 3 da | iys | | | 4 | (± 3 da | | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | 1.Pre-screening and screening can occur on the same day 2. FU period to start 4 weeks after ETP or EW visit. |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | ir). |
| Genetic blood sample<br>– Pre dose | | | | 7 | | | - | х | | | | =5,5 | | | | Pharmacogenetic sample may<br>be drawn any time from Visit 2<br>onwards. Informed consent for<br>optional substudies e.g.<br>genetics must be obtained<br>before collecting a sample |
| Sputum sample collection | | | X | | | | | x | | | | х | | | | Pre-dose collection and in a<br>sub-set of participants (~50 %)<br>at selected sites; also collected<br>for EW participants |
| PK, target<br>engagement and<br>immunogenicity<br>assessments | | | X | х | х | х | | x | | х | | х | Х | x | X | See SoA Table 2 for details |
| Exploratory<br>Biomarkers | | | X | | | | | X | | | | Х | | | | Pre dose collection |
| Efficacy | | - | (i ) | | | | | i i | - 1 | | 35 | ÿ | | <u> </u> | ğ | <u> </u> |
| Spirometry | | Х | Χ | | Х | Х | Х | X | Х | χ | Х | Х | | | | Test to be performed pre-dose<br>during the Treatment period |
| Reversibility | | X | | | 3 | | | | | | | | | | | |
| FeNO | | | X | Х | Х | Х | Χ | X | Χ | X | Х | Х | | | 8 | Test to be performed pre-dose |
| Review loss of<br>asthma control<br>criteria | | | | х | х | х | Х | х | Х | х | Х | х | | | | It will include review of data to<br>determine loss of asthma<br>control. See Section 9.1.5. |
| Dispense eDiary | | Х | | | | | | | - | | 2 | * | 0. | | | |

| Procedure | Pre-<br>Screen | Scree<br>n Run- | - | | | Tr | eatme | nt Per | riod | | | | Follo | ow-up | Period <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ingf | in | <u>, </u> | 2 day | s | | 0 | 90 - 915 | ± 3 da | ays | 53 | 53 | | ±3 da | ys) | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | 1.Pre-screening and screening can occur on the same day 2. FU period to start 4 weeks after ETP or EW visit. 3. Visit 3 - Day 4 /feet doos of |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | 11-7. |
| Collect eDiary | | | | 1 3 | 1 | | | 1 3 | 8 | | | X | | | | |
| Review eDiary | | | X | X | X | Х | Х | X | Х | Х | Х | X | | | | |
| Safety | | | | | | | • | | 111370 | | 201 | 200 | | 411 | | |
| 12-lead ECG | | х | Χ¹ | | | X1 | | X1 | | X¹ | | х | | | | Test to be performed pre-<br>dose and post-dose within 30<br>mins after end of infusion. |
| 24 hrs Holter | | х | Χ¹ | | | Χ¹ | | | | Χ¹ | | | | | | Holter monitor needs to be returned to clinic at end of 24-hour recording (i.e. the next day). 1. Place the Holter 30-60 mins prior to dosing. |
| Vital signs | | х | χ¹ | х | Х | Χ1 | х | Χı | Х | X1 | Х | х | Х | x | х | Test to be performed pre-<br>dose prior to spirometry and<br>post-dose prior the 12 -lead<br>ECG. |
| Dispense paper<br>Medical<br>Problems/Medication<br>s Taken worksheet | | х | Х | X | X | х | х | x | Х | х | Х | X | Х | х | | |
| Review paper<br>Medical<br>Problems/Medication<br>s Taken worksheet | | | х | х | х | х | Х | х | х | х | х | х | х | х | х | |

| Procedure | Pre-<br>Screen | Scree<br>n Run- | | | | Tr | eatme | nt Per | riod | | | | Follo | ow-up l | Period <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ing <sup>1</sup> | in | ± 2 days ± 3 days | | | | | | | | | ±3 da | ys) | | | |
| Visit 0 | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | Pre-screening and screening can occur on the same day FU period to start 4 weeks after ETP or EW visit. |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | IF). |
| AE/SAE review | X¹ | Χ¹ | | <b>←===</b> | | | | | | | | <b>&gt;</b> | х | х | х | At V0 and V1 collect only<br>SAEs considered as related to<br>study participation. |
| Concomitant<br>medication review | Х | Х | | <b>←===</b> | | | | | | | | <b>→</b> | Х | X | Х | |
| Questionnaires | | 8 3 | | | | | | | | | | | 66 | 165<br>10. | is a | ë |
| ACQ-5 | | х | | | | | ) | K | | | | | | | | After randomization, ACQ5 will<br>be completed by the<br>participants every 7 days. |
| SGRQ | | | X | | | X | | X | | X | 8 | Х | | | | |
| Study Treatment | | | | | | | | | | | | -01 | 500 | AU | - | <u> </u> |
| Double blind Study<br>Treatment (IP) | | | Х | | | х | | х | | Х | | | | | | Patients will remain in the clinic<br>for monitoring for at least 2<br>hours after the end of infusion. |
| FP/Sal (500/50)<br>dispensing | | Х | Х | | | | | | | | | | | | | |
| FP (mcg) dispensing | | | | | 500 | 250 | 100 | 50 | , | | | | 0.0 | | | |
| Dispense albuterol<br>(as needed) | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | 802 | |

| | | | | | Treatn | nent Peri | od | | | | F | ollow-up | ) <sup>2</sup> | 3.7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ± 2 days ± 3 days | | | | | | | | | (± 3 days) | | | Notes | |
| Visit | 21 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or EW) | 12 | 13 | 14 | Visit 2 = Day 1 (first dose of IP). FU period to start |
| Week | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 4 weeks after ETP or<br>EW visit. |
| Study Day | 1 | 8 | 15 | 29 | 43 | 49 | 71 | 85 | 99 | 113 | | | | EVV VISIL |
| Double blind<br>Study<br>Treatment<br>(IP) | X | | | x | | х | | x | | | | | | |
| PK sample | X2 | X | X | Х3 | | Х3 | | X1 | | X | X | X | X | 1. Pre dose and |
| Free and total<br>sST2 | X¹ | Х | Х | X3 | | X3 | | χ1 | | X | Х | X | X | post dose. 2. Post dose only. |
| Immunogenicit<br>y sam <mark>p</mark> le | X3 | | X | Хз | | Хз | | Х3 | | x | х | х | х | 3. Pre dose only. Pre-dose samples within 2 hours from the planned dosing time. Post-dose samples as soon as possible after end of infusion but must be taken within 4 hours. |

# 12.3. Appendix 3: Assessment Windows

# 12.3.1. Definitions of Assessment Windows for Analyses

Nominal visits will be used and no windowing will be applied for analysis.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

| Study Phase for all data except efficacy | Definition |
|---|---|
| Pre-treatment | Date ≤ Study Treatment Start Date |
| On-treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 28 days |
| Post-treatment | Date > Study Treatment Stop Date + 28 days |

| Study Phase for efficacy | Definition |
|---|---|
| Pre-treatment | Date ≤ Study Treatment Start Date |
| On-treatment | Study Treatment Start Date < Date ≤ Date of discontinuation from study treatment |
| | Or if the participant did not discontinue early from study treatment |
| | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 28 days |
| Post-treatment | Date > Study Treatment Stop Date + 28 days |

Once participants withdraw from study treatment they immediately restart their standard of care medication (ICS/LABA). As a result, any data collected past this point will have been impacted by the standard of care medications and any estimates produced biased by the additional use of ICS/LABA. For this reason, data post withdrawal from study treatment is not included in the on-treatment efficacy analysis.

The post treatment definition is the same for efficacy and safety analysis.

Completion of study epoch's will be defined as the following:

| Study Phase | Definition of Completion |
|---|---|
| Run-in | Randomised into study and received first dose of study treatment |
| Treatment | Completed Week 16 visit or withdrew from treatment phase due to loss of asthma control |
| Follow up | Completed 12 week follow-up period |

#### 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| Pre-treatment | <ul> <li>Conmed Start Date &lt; Study Treatment First Dose Date</li> <li>Conmed End Date &lt; Study Treatment First Dose Date</li> <li>CMSTRF = "BEFORE"</li> <li>Randomisation date is missing i.e. subject was not randomised</li> </ul> |
| On-treatment | <ul> <li>Study Treatment First Dose Date &lt;= Conmed Start Date &lt;= Study Treatment Last Dose Date + 28</li> <li>Study Treatment First Dose Date &lt;= Conmed End Date &lt;= Study Treatment Last Dose Date + 28</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (CMENRF ="DURING/AFTER" or CMENRF ="AFTER" or CMSTRF = "DURING")</li> <li>(CMSTRF = "BEFORE" or CMSTRF = "DURING" or CMENRF = "DURING/AFTER") and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(CMSTRF = "BEFORE" or CMSTRF ="DURING") and (CMENRF = "DURING/AFTER" or CMENRF = "AFTER")</li> <li>CMSTRF = "DURING"</li> <li>CMSTRF = "DURING"</li> </ul> |
| Post-treatment | <ul> <li>Conmed Start Date &gt; Study Treatment Last Dose Date + 28</li> <li>Conmed End Date &gt; Study Treatment Last Dose Date + 28</li> <li>CMENRF = "AFTER"</li> <li>CMENRF = "DURING/AFTER"</li> </ul> |
| All phases | Conmed start date is missing and CMSTRF is missing and conmed end date is missing and CMENRF is missing |

#### 1. NOTES:

- The duration of a single concomitant medication can extend over multiple study phases
- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### 12.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date + |
| Emergent | 28 days. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 28 days |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

#### 12.5.1. Reporting Process

# Software ■ The currently supported versions of SAS software will be used. Reporting Area HARP Server : uk1salx00175 HARP Compound : /arenv/arprod/gsk3772847/mid207597/

Additional information of reporting areas:

data\_look\_01

This is where the blinded dry run will take place.

final\_01:

This is where the end of treatment phase analysis will take place.

final 02:

This is where the end of study analysis will take place.

Details of the reporting efforts used for the iSRC analysis are detailed in the separate iSRC RAP.

#### **Analysis Datasets**

Analysis datasets will be created according to CDISC standards

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts

#### 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.

• The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| All unscheduled \ | All unscheduled visits will be included in listings. |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

#### 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 12.6.2. Study Population

#### Age

Date of birth will be set as YYYY where YYYY is the year of birth taken from the CRF. For participants who attended a screening visit, age will be calculated at the screening visit date. For pre-screen failures, age will be calculated at the pre-screening visit date.

#### **Body Mass Index (BMI)**

BMI = Weight (kg) / Height(m)<sup>2</sup>

#### **Treatment Misallocations**

To allocate treatment, the number of doses of GSK3772847 and Placebo that were given will be calculated, and the subject will be assigned to whichever treatment has the higher number. The only exception will be when both treatments were given equally, in which case the subject will be assigned their randomised treatment.

#### **Early Withdrawal from Study Treatment Date**

The eCRF captures the study treatment start and end, however this is the physical time and date of the infusion. The date of early withdrawal from study treatment is not captured and should therefore be calculated as follows:

- If the participant withdrew from treatment due to loss of asthma control then the date of early withdrawal from study treatment is set to the date of loss of asthma control.
- If the participant withdrew due to an AE/SAE/Death then withdrawal date is set to the AE/SAE onset date (all deaths should be reported as serious adverse events)
- If the participant withdrew from study treatment (for a reason other than those above) during the first 10 weeks of the study i.e. during the down titration of the background medications, then the FP/SAL or FP discontinuation date should be used as the date of withdrawal from study treatment.
- For participants who withdraw from study treatment (for a reason other than those above) between
  Week 10 and Week 16, there is no information on when they withdrew as they are no longer taking
  background medications. The date of early withdrawal from study treatment should therefore be set
  to the maximum of date of last dose of FP and date of last dose +1. This is because no more
  information is available other than the fact that they had not lost control prior to completing the
  down titration or prior to receiving their final dose of IP.

#### Treatment Compliance for Fluticasone Propionate (FP) and Salmeterol (SAL)

• Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)\*100

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are
  events of overdose. Cumulative compliance (since Day 1) by each background therapy will be
  calculated.
- Planned Treatment Duration is defined according to the schedule of activities.
- Compliance will be summarized by the following categories:

<80%.

 $\geq$  80% to < 95%,

 $\geq$ 95% to <105%,

≥ 105% to <120% and

≥120%

Date) + 29

#### **Extent of Exposure (Therapeutic Coverage)**

- IP is administered approximately every 4 weeks and each dose viewed as providing therapeutic coverage for 4 weeks (28 days).
- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Study Treatment Last Dose Date (Study Treatment First Dose
- The only exception to this will be when a participant dies in which case
  - Duration of Exposure in Days = Death Date (Study Treatment First Dose Date) + 1

#### **12.6.3.** Efficacy

#### **Loss of Asthma Control**

#### **Multiple Loss of Asthma Control**

If a participant reaches loss of control for multiple reasons then all reasons will be reported. For any
time to loss of asthma control analysis, the time of the earliest component of loss of control will be used.

#### **Date of Loss of Asthma Control**

Date of loss of control will be taken from the loss of control log page.

#### **Diary Data**

The vendor data captures the date on which the subject completes the diary (actual date of collection) rather than the date to which the questions relate. For example, in the morning diary subjects are asked 'Did you wake up due to asthma symptoms' and 'when you woke up due to your asthma symptoms did you use any rescue bronchodilator?' In the evening diaries subjects answer a question on daytime asthma symptoms and record the number of puffs of rescue medication used during the day. This means that the morning diary date in the raw data refers to the events during the previous night and that the evening diary relates to the events during the day time.

In order to ensure that correct observations are assigned to each four-week time period, measurements recorded in the morning diary will have 1 day removed in the analysis dataset to ensure that the date reflects the time period that the information related to. This adjustment is not required for evening diary as these are collected in the evening of the day to which they relate. Questions which this affects are those where the timepoint reference is MORNING:

- Was evening dose taken?
- Did you wake up due to asthma symptoms?
- When you woke up due to your asthma symptoms did you use any rescue bronchodilator?
- Number of puffs night time

PEF assessments will not have the adjustment made as these reflect the PEF as assessed (so the PEF recorded in the morning diary is the PEF at that time).

#### 12.6.4. Safety

#### **Adverse Events**

#### **Adverse Events of Special Interest (AESI)**

Systemic Allergic/Hypersensitivity and Non-allergic Reactions:

- Hypersensitivity (SMQ) [narrow]
- Anaphylactic reaction (SMQ) [narrow]
- Angioedema (SMQ) [narrow]

#### Alterations in immune response (infections)

All infections and serious infections reported under the MedDRA system organ class of 'Infections and Infestations'. Specific events of interest are opportunistic infections with preferred terms matching identified/pre-determined terms based on a published list of pathogens and/or presentations of specific pathogens to be considered as opportunistic infections in the setting of biologic therapy [Winthrop, 2015].

#### Alterations in immune response (malignancies):

All neoplasms reported under the MedDRA system organ class of 'Neoplasms, benign, malignant and unspecified (including cysts and polyps)'. Specific events of interest are malignancies which will be identified through matching of collected preferred terms with those from the following:

#### Sub-SMQs under the Malignancies SMQ:

- Malignant tumours sub-SMQ (narrow terms)
- Tumours of unspecified malignancy sub-SMQ (narrow terms)

#### Alterations in cardiovascular safety:

Cardiac disorders and serious cardiac disorders reported under the MedDRA system organ class of 'Cardiac Disorders'. Serious cardiac, vascular and thromboembolic (CVT) events, identified as all serious events classified under the MedDRA system organ classes of 'Cardiac Disorders' and of 'Vascular Disorders', and thromboembolic events identified through matching of collected preferred terms with those from the following:

#### Sub-SMQs under the Embolic and thrombotic events SMQ:

- Embolic and thrombotic events, arterial sub-SMQ (narrow terms)
- Embolic and thrombotic events, venous sub-SMQ (narrow terms)
- Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous sub-SMQ (narrow terms)

#### Sub-SMQs under the Ischaemic Heart Disease SMQ

- Myocardial infarction sub-SMQ (narrow terms)
- Other Ischaemic heart disease sub-SMQ (narrow terms)

#### Sub-SMQs under the Central Nervous System Vascular Disorders SMQ

- Ischaemic central nervous system vascular conditions sub-SMQ (narrow terms)
- Central nervous system vascular disorders, not specified as haemorrhagic or ischaemic sub-SMQ (narrow terms)
- Serious ischemic adverse events, a subset of the serious CVT events identified through matching of collected preferred terms with those from the following:

#### Local Injection Site Reactions

Local injection site reactions are identifying through preferred terms which had been selected by medical review of the MedDRA dictionary and are provided in a separate spreadsheet.

#### Rate of Events per 1000 Treatment Years

Rate of events per 1000 treatment years will be calculated using:

Rate = number of events \* 1000 / total treatment exposure in years where subjects can contribute more than one event.

This is equivalent to:

Rate = number of events \* 1000 / (number of subjects in treatment group \* mean treatment exposure in years).

#### Maximum/Minimum Definitions for Vital Signs Data

Maximum and Minimum: Maximum and Minimum post-randomisation value over all time-points (including scheduled and unscheduled assessments) will be presented.

#### FEV<sub>1</sub>

#### **Absolute Reversibility**

Absolute reversibility (mL) = (post-bronchodilator  $FEV_1$  – pre-bronchodilator  $FEV_1$ )

#### **Percent Reversibility**

Definition of Percentage Reversibility as a percentage of predicted  $FEV_1$  = ((post-bronchodilator  $FEV_1$ – pre-bronchodilator  $FEV_1$ ) / predicted  $FEV_1$ ) x 100%

Definition of Percentage Reversibility as a percentage of pre-bronchodilator  $FEV_1$  = ((post-bronchodilator  $FEV_1$ ) / pre-bronchodilator  $FEV_1$ ) x 100%

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as either completing the 16 week treatment period and three month safety follow up, or withdrawing from the treatment period early due to loss of asthma control and completing the three month safety follow up period. |
| | Withdrawn participants were not replaced in the study, unless the participants were withdrawn due to sites failing to comply with GCP. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Analysis | All missing data will be handled according to estimand of interest as described within the main body of the RAP. |
| ACQ | <ul> <li>If one of the five items in the ACQ is missing then the response from the four remaining items will be interpolated (pro-rata) to gain the overall response for the participant.</li> <li>If more than one item is missing then the ACQ will be considered missing.</li> </ul> |
| SGRQ | <ul> <li>Symptoms</li> <li>The Symptoms component will tolerate a maximum of 2 missed items. The weight for the missed item is subtracted from the total possible weight for the Symptoms component (662.5) and from the Total weight (3989.4)</li> <li>Activity</li> <li>The Activity component will tolerate a maximum of 4 missed items. The weight for the missed item is subtracted from the total possible weight for the Activity component (1209.1) and from the Total weight (3989.4)</li> <li>Impacts</li> <li>The Impacts component will tolerate a maximum of 6 missed items. The weight for the missed item is subtracted from the total possible weight for the Impacts component (2117.8) and from the Total weight (3989.4)</li> </ul> |
| | If any component has more missing items then mentioned above then the SGRQ will be considered missing. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

Values of potential clinical importance will not be used in this study, instead normal reference ranges of "Low", "Normal" and "High" will be used.

# 12.9. Appendix 9: Abbreviations & Trade Marks

# 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IgE | Immunoglobulin E |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| mIT | Modified Intent-to-Treat excluding GCP non-compliant subjects |
| mITT_LoC | Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of |
| | Control) |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomisation & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAFF_ALL | Safety including site including GCP non-compliant subjects |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

# 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

None

Trademarks not owned by the GlaxoSmithKline Group of Companies

NONMEM

SAS

#### 12.10. Appendix 10: List of Data Displays

All displays (Tables, Figures & Listings) will use the term 'Subjects' instead of "Participants".

#### 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic or Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic or Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 12.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| ETP [1] | End of Treatment Phase Statistical Analysis Complete |
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.10.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Subject Disposition | | | | |
| 1.1. | SAFF_ALL | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | ETP, SAC |
| 1.2. | SAFF_ALL | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 1.3. | SAFF_ALL | ES4 | Summary of Subject Disposition at Each Study Epoch | ICH E3 | ETP, SAC |
| 1.4. | ASE | ES6 | Summary of Screening/Run-in Status and Reasons for Screen/Run-in Failure | Journal Requirements | ETP, SAC |
| 1.5. | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | ETP, SAC |
| 1.6. | SAFF_ALL | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | ETP, SAC |
| Protoco | ol Deviation | | | | |
| 1.7. | SAFF_ALL | DV1 | Summary of Important Protocol Deviations | ICH E3 | ETP, SAC |
| 1.8. | SAFF_ALL | IE1 | Summary of Inclusion/ Exclusion Deviations | ICH E3 | ETP, SAC |
| Popula | tion Analysed | | | | |
| 1.9. | Enrolled | SP1 | Summary of Study Populations | IDSL | ETP, SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.10. | SAFF_ALL | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | ETP, SAC |
| 1.11. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | ETP, SAC |
| 1.12. | SAFF_ALL | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | ETP, SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.13. | SAFF_ALL | MH4 | Summary of Current Medical Conditions | ICH E3 | ETP, SAC |

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.14. | SAFF_ALL | MH4 | Summary of Past Medical Conditions | ICH E3 | ETP, SAC |
| 1.15. | SAFF_ALL | SP07 | Summary of Family History of Cardiovascular Disorders at Screening | | ETP, SAC |
| 1.16. | SAFF_ALL | POP_T01 | Summary of Disease Duration and Exacerbation History | | ETP, SAC |
| 1.17. | SAFF_ALL | SU1 | Summary of Smoking History at Screening | | ETP, SAC |
| 1.18. | SAFF_ALL | CM1 | Summary of Pre-treatment Non-Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| 1.19. | SAFF_ALL | CM1 | Summary of On-treatment Non-Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| 1.20. | SAFF_ALL | CM1 | Summary of Post-treatment Non-Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| 1.21. | SAFF_ALL | CM1 | Summary of On-treatment Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| 1.22. | SAFF_ALL | CM1 | Summary of Post-treatment Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| Pre-trea | tment Lung Fun | ction | | | |
| 1.23. | SAFF_ALL | POP_T02 | Summary of Screening Lung Function | Include Pre- and Post- albuterol (salbutamol) FEV <sub>1</sub> , FVC, FEV <sub>1</sub> /FVC and % Predicted Normal and post-BD at screening %predicted. Include overall and by treatment group. | ETP, SAC |
| 1.24. | SAFF_ALL | POP_T03 | Summary of Baseline Lung Function | FEV <sub>1</sub> , FVC, FEV <sub>1</sub> /FVC and % Predicted Normal. Include overall and by treatment group. | ETP, SAC |
| Exposu | re and Treatmen | t Compliance | | | |
| 1.25. | SAFF_ALL | EX1 | Summary of Exposure and Compliance to Background Therapy (FP and SAL) | ICH E3 | ETP, SAC |

# 12.10.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | re | | | | |
| 2.1. | SAFF_ALL | EX1 | Summary of Exposure to Study Treatment | ICH E3 | ETP, SAC |
| Primary | Endpoint: Los | ss of Asthma Con | trol Weeks 0-16 | | |
| 2.2. | mITT_LoC | EFF_T01 | Summary of Loss of Asthma Control | Include overall loss of control, each component and the combination of exacerbation or inability to titrate. | ETP, SAC |
| 2.3. | mITT_LoC | EFF_T02 | Summary of On-treatment Intercurrent Events | | ETP, SAC |
| 2.4. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | | ETP, SAC |
| 2.5. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | | ETP, SAC |
| 2.6. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | | ETP, SAC |
| 2.7. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | | ETP, SAC |
| Second | ary Endpoint: | Loss of Asthma C | ontrol Weeks 0-6 | | |
| 2.8. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | | ETP, SAC |
| 2.9. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | | ETP, SAC |
| 2.10. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | | ETP, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | | ETP, SAC |
| Second | lary Endpoints: | Time to Loss of | Asthma Control | | |
| 2.12. | mITT_LoC | EFF_T05 | Summary and Analysis of Time to Loss of Asthma Control (Primary Estimand) | | ETP, SAC |
| 2.13. | mITT_LoC | EFF_T05 | Summary and Analysis of Time to Loss of Asthma Control (Secondary Estimand) | | ETP, SAC |
| Second | lary Endpoints: | Hospitalisation a | and Emergency Room Visits | | |
| 2.14. | mITT | EFF_T06 | Summary and Rate of Asthma-Related On-treatment Hospitalisations and Emergency Room Visits (Primary Estimand) | | ETP, SAC |
| Second | lary Endpoint: | ACQ-5 and SGRQ | | | |
| 2.15. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in ACQ-5 Total Score (Primary Estimand) | | ETP, SAC |
| 2.16. | mITT | EFF_T07 | Summary of ACQ-5 Responders (Primary Estimand) | | ETP, SAC |
| 2.17. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in SGRQ Total Score (Primary Estimand) | | ETP, SAC |
| 2.18. | mITT | EFF_T07 | Summary of SGRQ-Responders (Primary Estimand) | | ETP, SAC |
| Second | Secondary Endpoint: FEV1 and PEF | | | | |
| 2.19. | mITT | EFF_T07 | Summary of Raw and Change from Baseline FEV <sub>1</sub> (Primary Estimand) | | ETP, SAC |
| 2.20. | mITT | EFF_T08 | Analysis of Change from Baseline in FEV <sub>1</sub> up to Week 4(Primary Estimand) | | ETP, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21. | mITT | EFF_T07 | Summary of Raw and Change from Baseline Fractional Exhaled Nitric Oxide (FeNO) (Primary Estimand) | | ETP, SAC |
| 2.22. | mITT | EFF_T08 | Analysis of Change from Baseline in Fractional Exhaled Nitric Oxide (FeNO) up to Week 4 (Primary Estimand) | | ETP, SAC |
| Second | Secondary Endpoint: Exacerbations | | | | |
| 2.23. | mITT | EFF_T09 | Summary of On-treatment Asthma Exacerbations | | ETP, SAC |
| Second | lary Endpoint: | Eosinophils | | | |
| 2.24. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in Eosinophils (Primary Estimand) | | ETP, SAC |
| 2.25. | mITT | EFF_T08 | Analysis of Eosinophils up to Week 4 (Primary Estimand) | | ETP, SAC |
| Second | lary Endpoint: | PEF, Daytime Syn | nptom Score, Night-time Symptom Score and Rescue Medication | on | |
| 2.26. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Morning Peak Expiratory Flow (PEF) | | ETP, SAC |
| 2.27. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Evening Peak Expiratory Flow (PEF) | | ETP, SAC |
| 2.28. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Daytime Asthma Symptom Score | | ETP, SAC |
| 2.29. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Night-Time Awakenings Due to Asthma Symptoms | | ETP, SAC |
| 2.30. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Rescue Medication use (Albuterol/Salbutamol) | | ETP, SAC |

# 12.10.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Endpoint: Los | s of Asthma Con | trol | | |
| 2.1. | mITT_LoC | | Plot of Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | Include overall and components of loss on control | ETP, SAC |
| 2.2. | mITT_LoC | | Plot of Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | Include overall and components of loss on control | ETP, SAC |
| 2.3. | mITT_LoC | | Cumulative Density Plot of the Posterior Distribution for Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | | ETP, SAC |
| 2.4. | mITT_LoC | | Cumulative Density Plot of the Posterior Distribution for Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | | ETP, SAC |
| 2.5. | mITT_LoC | | Plot of Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | Include overall and components of loss on control | ETP, SAC |
| 2.6. | mITT_LoC | | Plot of Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | Include overall and components of loss on control | ETP, SAC |
| 2.7. | mITT_LoC | | Cumulative Density Plot of the Posterior Distribution for Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | | ETP, SAC |
| 2.8. | mITT_LoC | | Cumulative Density Plot of the Posterior Distribution for Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | | ETP, SAC |
| Seconda | Secondary Endpoint: Time to Loss of Control | | | | |
| 2.9. | mITT_LoC | | Kaplan-Meir Plot of Time to Loss of Asthma Control (Primary Estimand) | | ETP, SAC |
| 2.10. | mITT_LoC | | Kaplan-Meir Plot of Time to Loss of Asthma Control (Secondary Estimand) | | ETP, SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | Secondary Endpoint: Secondary Analysis of Loss of Asthma Control | | | | |
| 2.11. | mITT_LoC | | Cumulative Density Plot of Eosinophils | | ETP, SAC |
| 2.12. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.13. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.14. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 2.15. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.16. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.17. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.18. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 2.19. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.20. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE by Treatment - Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.21. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.22. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.24. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.25. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.26. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 2.27. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| Second | ary Endpoint: | Exploratory Analy | rsis of FEV1 | | |
| 2.28. | mITT | | FEV1 at Week 4 vs Eosinophils by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.29. | mITT | | FEV1 at Week 4 vs Eosinophils – Fractional Polynomial Treatment Difference | | ETP, SAC |
| 2.30. | mITT | | FEV1 at Week 4 vs IgE by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.31. | mITT | | FEV1 at Week 4 vs IgE – Fractional Polynomial Treatment Difference | | ETP, SAC |
| 2.32. | mITT | | FEV1 at Week 4 vs FeNO by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.33. | mITT | | FEV1 at Week 4 vs FeNO – Fractional Polynomial Treatment Difference | | ETP, SAC |
# 12.10.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | SAFF_ALL | SAFE_T01 | Overview of On-treatment Adverse Events During the Study | | ETP, SAC |
| 3.2. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.3. | SAFF_ALL | AE1 | Summary of All Post-treatment Adverse Events by System<br>Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.4. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.5. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.6. | SAFF_ALL | AE1 | Summary of All On-treatment Fatal Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.7. | SAFF_ALL | AE3 | Summary of All On-treatment Common (>=3%) Adverse Events by Overall Frequency | ICH E3 | ETP, SAC |
| 3.8. | SAFF_ALL | AE1 | Summary of All On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.9. | SAFF_ALL | AE15 | Summary of All On-treatment Common (>=3%) Non-serious<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | FDAAA, EudraCT | ETP, SAC |
| 3.10. | SAFF_ALL | AE1 | Summary of All Pre-treatment Serious Adverse Events by System Organ Class and Preferred Term | | ETP, SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.11. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.12. | SAFF_ALL | AE1 | Summary of All Post-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.13. | SAFF_ALL | AE16 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Participants and Occurrences) | FDAAA, EudraCT | ETP, SAC |
| 3.14. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term | IDSL | ETP, SAC |
| 3.15. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | IDSL | ETP, SAC |
| Advers | e Events of Sp | ecial Interest (AES | Sis) | | · |
| 3.16. | SAFF_ALL | AE1 | Summary of On-treatment Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.17. | SAFF_ALL | AE1 | Summary of On-treatment Serious Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.18. | SAFF_ALL | AE1 | Summary of Post-treatment Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.19. | SAFF_ALL | AE1 | Summary of Post-treatment Serious Adverse Events of Special Interest | IDSL | ETP, SAC |
| Mexico | Specific Table | S | | | |
| 3.20. | SAFF_ALL | | Summary of Suspected Investigational Product Adverse Reaction (Mexican Participants Only) | | ETP, SAC |
| 3.21. | SAFF_ALL | | Summary of Suspected Investigational Product Adverse Reaction (Non-Mexican Participants) | | ETP, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | aboratory: Chemistry | | | | |
| 3.22. | SAFF_ALL | LB1 | Summary of Clinical Chemistry | ICH E3 | ETP, SAC |
| 3.23. | SAFF_ALL | LB1 | Summary of Change from Baseline in Clinical Chemistry | ICH E3 | ETP, SAC |
| 3.24. | SAFF_ALL | LB16 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | ETP, SAC |
| Labora | tory: Hematolo | gy and Cardiac M | arkers | | |
| 3.25. | SAFF_ALL | LB1 | Summary of Hematology and Cardiac Markers | ICH E3 | ETP, SAC |
| 3.26. | SAFF_ALL | LB1 | Summary of Changes from Baseline in Hematology and Cardiac Markers | ICH E3 | ETP, SAC |
| 3.27. | SAFF_ALL | LB16 | Summary of Worst Case Hematology and Cardiac Markers<br>Results Relative to Normal Range Post-Baseline Relative to<br>Baseline | ICH E3 | ETP, SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.28. | SAFF_ALL | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | ETP, SAC |
| 3.29. | SAFF_ALL | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | ETP, SAC |
| ECG | • | | | | |
| 3.30. | SAFF_ALL | | Summary of Antihistamine, Decongestant and Caffeine Use Prior to ECG assessments | | ETP, SAC |
| 3.31. | SAFF_ALL | EG1 | Summary of ECG Findings | IDSL | ETP, SAC |
| 3.32. | SAFF_ALL | EG2 | Summary of ECG Values by Visit | IDSL | ETP, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.33. | SAFF_ALL | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | ETP, SAC |
| 3.34. | SAFF_ALL | EG10 | Summary of Maximum QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | ETP, SAC |
| 3.35. | SAFF_ALL | EG11 | Summary of Maximum Increase in QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | ETP, SAC |
| Holter | | | | | |
| 3.36. | SAFF_ALL | HM1 | Summary of Holter Interpretations | IDSL | ETP, SAC |
| 3.37. | SAFF_ALL | HM2 | Summary of Holter Abnormalities | IDSL | ETP, SAC |
| 3.38. | SAFF_ALL | HM3 | Summary of Holter Values | IDSL | ETP, SAC |
| 3.39. | SAFF_ALL | HM3 | Summary of Change from Baseline in Holter Values | IDSL | ETP, SAC |
| 3.40. | SAFF_ALL | HM4 | Summary of Subjects with R-on-T Beats | IDSL | ETP, SAC |
| Vital Si | gns | | | | |
| 3.41. | SAFF_ALL | VS1 | Summary of Vital Signs | ICH E3 | ETP, SAC |
| 3.42. | SAFF_ALL | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | ETP, SAC |
| 3.43. | SAFF_ALL | VS1 | Summary of Change from Pre-dose to Post-dose in Vital Signs | ICH E3 | ETP, SAC |

# 12.10.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | ary: Pharmaco | kinetic | | | |
| 4.1. | PK | | Summary of PK Serum Concentrations of GSK3772847 | | SAC only |
| 4.2. | PK | | Summary of Incidence and Titres of Anti-GSK3772847<br>Antibodies | | SAC only |

# 12.10.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | dary: Pharmaco | odynamic | | | |
| 6.1. | mITT | | Summary of Raw and Percentage Change from Baseline in Free Soluble ST2 concentration (ug/L) (On-treatment) | Pre and Post dose. | ETP, SAC |
| 6.2. | mITT | | Analysis of Percentage Change from Baseline in Free Soluble ST2 concentration (ug/mL) (On-treatment) | Pre dose only. | ETP, SAC |
| 6.3. | mITT | | Summary of Raw and Percentage Change from Baseline in Free soluble ST2 concentration (ug/L) (Post-treatment) | | ETP, SAC |
| 6.4. | mITT | | Analysis of Percentage Change from Baseline in Free soluble ST2 concentration (ug/mL) (Post-treatment) | | ETP, SAC |
| 6.5. | mITT | | Summary of Raw and Percentage Change from Baseline in Total Soluble ST2 concentration (ug/L) (On-treatment) | Pre and Post dose. | ETP, SAC |
| 6.6. | mITT | | Analysis of Percentage Change from Baseline in Total Soluble ST2 concentration (ug/L) (On-treatment) | Pre dose only. | ETP, SAC |
| 6.7. | mITT | | Summary of Raw and Percentage Change from Baseline in Total Soluble ST2 concentration (ug/L) (Post-treatment) | | ETP, SAC |
| 6.8. | mITT | | Analysis of Percentage Change from Baseline in Total Soluble ST2 concentration (ug/L) (Post-treatment) | | ETP, SAC |
| Explor | atory: Biomark | ers | | | |
| 6.9. | mITT | | Summary and Change from Baseline in Induced Sputum Biomarkers (subset) at Weeks 8 and 16 | Include geometric mean and %CV | ETP, SAC |
| 6.10. | mITT | | Summary and Change from Baseline in Exploratory Serum Markers at Weeks 8 and 16 | Include geometric mean and %CV | ETP, SAC |

# 12.10.10. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | dary: Pharmaco | kinetic | | | |
| 6.1. | PK | | Plot of Serum Concentrations of GSK3772847 over Time | | ETP, SAC |
| 6.2. | PK | | Pre-dose Trough Concentration of GSK3772847 vs Eosinophils at Week 4 | | ETP, SAC |
| 6.3. | PK | | Pre-dose Trough Concentration of GSK3772847 vs FeNO at Week 4 | | ETP, SAC |
| 6.4. | PK | | Pre-dose Trough Concentration of GSK3772847 vs IgE at Week 4 | | ETP, SAC |

# 12.10.11. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | dary: Pharmaco | odynamic | | | |
| 6.5. | mITT | | Plot of Percentage Change from Baseline in Free Soluble ST2 levels (On-treatment) | | ETP, SAC |
| 6.6. | mITT | | Plot of Percentage Change from Baseline in Free soluble ST2 levels (Post-treatment) | | ETP, SAC |
| 6.7. | mITT | | Plot of Percentage Change from Baseline in Total Soluble ST2 levels (On-treatment) | | ETP, SAC |
| 6.8. | mITT | | Plot of Percentage Change from Baseline in Total Soluble ST2 levels (Post-treatment) | | ETP, SAC |
| 6.9. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Free soluble ST2 by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 6.10. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Free soluble ST2<br>Treatment Difference – Fractional Polynomial (Primary<br>Estimand) | | ETP, SAC |
| 6.11. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Free soluble ST2 by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 6.12. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Free soluble ST2 Treatment Difference – Fractional Polynomial (Secondary Estimand) | | ETP, SAC |

# **12.10.12. ICH Listings**

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen and Run-in Failure | Journal Guidelines | ETP, SAC |
| 2. | SAFF_ALL | ES2 / ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | ETP, SAC |
| 3. | SAFF_ALL | SD2/SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | ETP, SAC |
| 4. | SAFF_ALL | BL1 / BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | ETP, SAC |
| 5. | SAFF_ALL | TA1 / CP_RD1x | Listing of Planned and Actual Treatments | IDSL | ETP, SAC |
| Protoc | ol Deviations | <u> </u> | | l | 1 |
| 6. | SAFF_ALL | DV2 | Listing of Important Protocol Deviations | ICH E3 | ETP, SAC |
| 7. | SAFF_ALL | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | ETP, SAC |
| Popula | tions Analysed | | | | • |
| 8. | SAFF_ALL | | Listing of Participants Excluded from Any Population (GCP non compliance) | ICH E3. | ETP, SAC |
| Demog | raphic and Bas | seline Characteris | tics | ' | • |
| 9. | SAFF_ALL | DM2 | Listing of Demographic Characteristics | ICH E3 | ETP, SAC |
| 10. | SAFF_ALL | DM9 | Listing of Race | ICH E3 | ETP, SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | SAFF_ALL | CP_CM3 | Listing of Concomitant Medications | IDSL | ETP, SAC |
| Exposi | ire and Treatme | ent Compliance | | | |
| 12. | SAFF_ALL | EX3 | Listing of Exposure Data | ICH E3 | ETP, SAC |
| Advers | e Events | | | | |
| 13. | SAFF_ALL | AE8 | Listing of All Adverse Events | ICH E3 | ETP, SAC |
| 14. | SAFF_ALL | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | ETP, SAC |
| 15. | SAFF_ALL | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 16. | SAFF_ALL | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | ETP, SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 17. | SAFF_ALL | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | ETP, SAC |
| 18. | SAFF_ALL | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | ETP, SAC |
| 19. | SAFF_ALL | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | ETP, SAC |
| 20. | SAFF_ALL | AE8 | Listing of Serious Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 21. | SAFF_ALL | AE8 | Listing of Adverse Events of Special Interest | ICH E3 | ETP, SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hepato | biliary (Liver) | | | | |
| 22. | SAFF_ALL | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | ETP, SAC |
| 23. | SAFF_ALL | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | ETP, SAC |
| All Lab | oratory | | | | |
| 24. | SAFF_ALL | LB5 / LB6 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | ETP, SAC |
| 25. | SAFF_ALL | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | ETP, SAC |
| ECG | | | | | |
| 26. | SAFF_ALL | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | ETP, SAC |
| 27. | SAFF_ALL | EG5 | Listing of Abnormal ECG Findings | IDSL | ETP, SAC |
| Holter | | | | | |
| 28. | SAFF_ALL | MH6 | Listing of Holter R-on-T Beat Data | IDSL | ETP, SAC |
| 29. | SAFF_ALL | MH7 | Listing of Holter {Supraventricular} {Ventricular} Event Data | IDSL, Update title as appropriate based on data | ETP, SAC |
| 30. | SAFF_ALL | MH8 | Listing of Holter {Sustained} {Non-sustained} {Supraventricular} {Ventricular} Run | IDSL, Update title as appropriate based on data | ETP, SAC |
| 31. | SAFF_ALL | MH9 | Listing of Holter Atrial {Fibrillation} {Flutter} Data | IDSL, Update title as appropriate based on data | ETP, SAC |
| 32. | SAFF_ALL | MH10 | Listing of Holter Abnormalities | IDSL | ETP, SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 33. | SAFF_ALL | VS4 | Listing of All Vital Signs Data | IDSL | ETP, SAC |
| Primary | y Analysis Data | : Loss of Asthma | Control and Intercurrent Events | | |
| 34. | mITT_LoC | | Listing of Loss of Asthma Control | Include all reasons for loss of control and time to loss of asthma control | ETP, SAC |
| 35. | mITT_LoC | | Listing of Intercurrent Events | Include treatment subject was analysed as taking and treatment at time of loss of control | ETP, SAC |

# 12.10.13. Non-ICH Listings

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Stud | y Population | | | | |
| 36. | SAFF_ALL | SP2 | Listing of the Follow-up Contact | ng of the Follow-up Contact | |
| 37. | SAFF_ALL | TA1 | Listing of Treatment Misallocations | ng of Treatment Misallocations Change Centre ID to Investigator ID: xxxxxx and also Investigator at Centre: xxxxxx | |
| 38. | SAFF_ALL | SP4 | Listing of Overall Percentage Treatment<br>Compliance | | |
| Seco | ondary Efficac | y | | | |
| 39. | mITT | | Listing of Eosinophils | ing of Eosinophils Include randomisation and analysis strata | |
| 40. | mITT | SP10 | Listing of Lung Function Results at Screening | sting of Lung Function Results at Screening | |
| 41. | mITT | SP10 | Listing of Lung Function Results post-Screening | sting of Lung Function Results post-Screening | |
| 42. | mITT | S3 | Listing of Asthma Exacerbations | Include a column for severity | ETP, SAC |
| 43. | mITT | | Listing of Asthma Control Questionnaire (ACQ-5) | Listing of Asthma Control Questionnaire (ACQ-5) | |
| 44. | mITT | | Listing of St George's Respiratory Questionnaire (SGRQ) | | |
| 45. | mITT | | Listing of Peak Exploratory Flow (PEF) | | ETP, SAC |
| 46. | mITT | | Listing of Fractional Exhaled Nitric Oxide (FeNO) | | ETP, SAC |
| 47. | mITT | | Listing of Daytime and Night-time Asthma<br>Symptoms | isting of Daytime and Night-time Asthma | |
| 48. | mITT | | Listing of Rescue Medication Use | Listing of Rescue Medication Use ET | |
| 49. | mITT | | Listing of Hospitalisations and Emergency Room Visits | | |
| 50. | PK | | Listing of Serum GSK3772847 Concentration | | SAC Only |

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 51. | mlTT | | List of Free and Total Soluble ST2<br>Concentrations | | |
| Adve | erse Events | | | | |
| 52. | SAFF_ALL | | Listing of Clinical Chemistry | | ETP, SAC |
| 53. | SAFF_ALL | | Listing of Haematology and Cardiac Markers | | ETP, SAC |
| 54. | SAFF_ALL | | Listing of Anti-GSK3772847 Antibodies | | ETP, SAC |
| 55. | SAFF_ALL | ESI8 | Listing of AE Terms of Special Interest | IDSL | ETP, SAC |
| Expl | Exploratory Biomarker | | | | |
| 56. | mlTT | | Listing of Induced Sputum and Exploratory<br>Serum Biomarkers | | ETP, SAC |
| Med | ical History | | | | |
| 57. | SAFF_ALL | MH2 | Listing of Medical Conditions at Screening | | ETP, SAC |
| 58. | SAFF_ALL | SP5 | Listing of Family History of Cardiovascular<br>Disorders | | |
| 59. | SAFF_ALL | SP6 | Listing of Asthma History | | ETP, SAC |
| 60. | SAFF_ALL | SP7 | Listing of Smoking History and Smoking Status | | ETP, SAC |
| 61. | SAFF_ALL | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text | | |
| Live | r Events: Note | only produced if | there is a Liver Event | | |
| 62. | SAFF_ALL | LIVER5 | Listing of Liver Events | Listing of Liver Events | |
| 63. | SAFF_ALL | LIVER6 | Listing of Liver Event Information for RUCAM Score | Y I FIP | |
| 64. | SAFF_ALL | LIVER7 | Listing of Liver Biopsy | | ETP, SAC |

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 65. | SAFF_ALL | LIVER8 | Listing of Liver Imaging Details | | ETP, SAC |
| Card | liovascular Ev | ents: Note only pr | oduced if there is a Cardiovascular Event | | |
| 66. | SAFF_ALL | Patient Profile | Listing of Myocardial infarction/unstable angina | | ETP, SAC |
| 67. | SAFF_ALL | Patient Profile | Listing of Congestive heart failure | | ETP, SAC |
| 68. | SAFF_ALL | Patient Profile | Listing of Arrhythmias | | ETP, SAC |
| 69. | SAFF_ALL | Patient Profile | Listing of Valvulopathy | | ETP, SAC |
| 70. | SAFF_ALL | Patient Profile | Listing of Pulmonary hypertension | | ETP, SAC |
| 71. | SAFF_ALL | Patient Profile | Listing of Cerebrovascular events/stroke and transient ischemic attack | | |
| 72. | SAFF_ALL | Patient Profile | Listing of Peripheral arterial thromboembolism | Listing of Peripheral arterial thromboembolism | |
| 73. | SAFF_ALL | Patient Profile | Listing of Deep venous thrombosis/pulmonary embolism | | |
| 74. | SAFF_ALL | Patient Profile | Listing of Revascularisation | | |
| 75. | SAFF_ALL | Patient Profile | Listing of Deaths | | |

# 12.11. Appendix 11: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | GSK3772847 |
|---|---|---|
| Compound Number | : | Reporting and Analysis Plan for a randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma. |
| <b>Effective Date</b> | : | 20-DEC-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2017N311825\_02.
- This RAP is intended to describe the Efficacy, Safety, PK, PD and Biomarker analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the End of Treatment Phase (ETP) and Statistical Analysis Complete (SAC) deliverable.
- This study does have an internal safety review committee (iSRC) and all details of iSRC deliverable are documented in a separate iSRC RAP.

#### **Author's Name and Functional Area:**

| Approver | Date |
|-----------------------------------------------------------|-------------|
| PPD | 27 NOV 2010 |
| Principal Statistician (Respiratory, Clinical Statistics) | 27-NOV-2018 |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Review Confirmations** (Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Investigation Lead (Respiratory, HUP Clinical Development) | 27-NOV-2018 |
| Principal Programmer (Respiratory, Clinical Programming) | 27-NOV-2018 |
| Clinical Development Physician (Respiratory, MDC Global Clinical) | 27-NOV-2018 |
| Scientist (Respiratory, Value Evidence and Outcomes) 19-DEC-2018 | |
| Director (Respiratory, Value Evidence and Outcomes) | 29-NOV-2018 |
| Senior Director (Respiratory, Clinical Pharmacology Modelling and Simulation) | 27-NOV-2018 |
| Director of Clinical Development (Respiratory, MDC Global Clinical) | 18-DEC-2018 |
| Senior Scientific Director (Respiratory, RD AI DPU Head) | 18-DEC-2018 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| Senior Statistics Director (Respiratory, Clinical Statistics) | 20-DEC-2018 |
| Programming Manger (Respiratory, Clinical Programming) 20-DEC-2018 | |

## TABLE OF CONTENTS

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 6 |
| 2. | CLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | | | |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | 13 |
| 3. | PLAN | INED ANALYSES | 13 |
| ٠. | 3.1. | End of Treatment Phase Analyses | |
| | 3.2. | Final Analyses | |
| 4. | ΔΝΔΙ | YSIS POPULATIONS | 14 |
| т. | 4.1. | Protocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 16 |
| | | VENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | |
| | 5.5. | Multiple Comparisons and Multiplicity | 19 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 19 |
| 6. | STUE | DY POPULATION ANALYSES | 20 |
| | 6.1. | Overview of Planned Study Population Analyses | 20 |
| | 6.2. | Disposition | 20 |
| | 6.3. | Medical Conditions | <mark>20</mark> |
| | 6.4. | Concomitant Medications | 20 |
| 7. | EFFIC | CACY ANALYSES | 21 |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomisation) Events | |
| | | 7.1.5. Statistical Analyses / Methods | |
| | | • | |
| | 7.0 | | |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint and Summary Measure | |
| | | 7.2.2. Population of Interest | |
| | | 7.2.3. Strategy for Intercurrent (Post-Randomisation) Events | |
| | | 7.2.4. Statistical Analyses / Methods | |
| | | 7.2.4.1. Statistical Methodology Specification | 27 |
| Q | SVEE | TV ANALYSES | 30 |


207597

| | 8.1. | | Events Analyses | |
|---|---|---|---|---|
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | | ns, Electrocardiogram (ECG) and Holter | |
| | 8.4. | | Chemistry, Haematology and Cardiac Markers | |
| | 8.5. | | <del>9</del> \$ | |
| | 8.6. | Clinical L | aboratory Analyses | 32 |
| 9. | PHAR | MACOKIN | IETIC ANALYSES | 32 |
| | 9.1. | | ry Pharmacokinetic Analyses | |
| | | 9.1.1. | Endpoint / Variables | |
| | | 9.1.2. | Population of Interest | |
| | | 9.1.3. | Strategy for Intercurrent (Post-Randomisation) Events | |
| | | 9.1.4. | Statistical Analyses / Methods | |
| 10 | | MACODY | NAMIC AND BIOMARKER ANALYSES | 20 |
| 10. | 10.1. | | ry Pharmacodynamic Analyses | |
| | 10.1. | 10.1.1. | | |
| | | | • | |
| | | 10.1.2. | Summary Measure | |
| | | 10.1.3. | Population of Interest | |
| | | 10.1.4. | Strategy for Intercurrent (Post-Randomisation) Events | |
| | | 10.1.5. | Statistical Analyses / Methods | |
| | 10.2. | | ory Biomarker Analyses | |
| | | 10.2.1. | Endpoint / Variables | |
| | | 10.2.2. | Summary Measure | |
| | | 10.2.3. | Population of Interest | |
| | | 10.2.4. | Strategy for Intercurrent (Post-Randomisation) Events | 3 <mark>5</mark> |
| | | 10.2.5. | Statistical Analyses / Methods | 35 |
| 11. | REFE | RENCES. | | 36 |
| 12. | APPE | NDICES | | 37 |
| | 12.1. | | c 1: Protocol Deviation Management | |
| | 12.2. Appendix 2: Schedule of Activities | | | |
| | | | Protocol Defined Schedule of Events | |
| | 12.3. | | 3: Assessment Windows | |
| | 12.0. | 12.3.1. | Definitions of Assessment Windows for Analyses | |
| | 12.4. | - | 4: Study Phases and Treatment Emergent Adverse | |
| | 12.4. | | | 15 |
| | | 12.4.1. | | |
| | | 12.4.1. | Study Phases | |
| | | 40.40 | 12.4.1.1. Study Phases for Concomitant Medication | |
| | 40.5 | 12.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 12.5. | | 5: Data Display Standards & Handling Conventions | |
| | | 12.5.1. | Reporting Process | |
| | | 12.5.2. | Reporting Standards | |
| | 12.6. | | c 6: Derived and Transformed Data | |
| | | 12.6.1. | General | |
| | | 12.6.2. | Study Population | |
| | | 12.6.3. | Efficacy | |
| | | 12.6.4. | Safety | |
| | 12.7. | Appendix | 7: Reporting Standards for Missing Data | 53 |
| | | 12.7.1. | Premature Withdrawals | |
| | | 12.7.2. | Handling of Missing Data | |


| | 12.7.2.1. Handling of Missing and Partial Dates | <mark>54</mark> |
|---|---|---|
| 12.8. | Appendix 8: Values of Potential Clinical Importance | <mark>56</mark> |
| 12.9. | Appendix 9: Abbreviations & Trade Marks | 57 |
| | 12.9.1. Abbreviations | 57 |
| | 12.9.2. Trademarks | 58 |
| 12.10. | Appendix 10: List of Data Displays | |
| | 12.10.1. Data Display Numbering | |
| | 12.10.2. Mock Example Shell Referencing | |
| | 12.10.3. Deliverables | |
| | 12.10.4. Study Population Tables | |
| | 12.10.5. Efficacy Tables | |
| | 12.10.6. Efficacy Figures | |
| | 12.10.7. Safety Tables | 68 |
| | 12.10.8. Pharmacokinetic Tables | |
| | 12.10.9. Pharmacodynamic and Biomarker Tables | 74 |
| | 12.10.10. Pharmacokinetic Figures | 75 |
| | 12.10.11. Pharmacodynamic and Biomarker Figures | |
| | 12.10.12.ICH Listings | 77 |
| | 12.10.13. Non-ICH Listings | |
| 12.11. | Appendix 11: Example Mock Shells for Data Displays | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 207597:

| Protocol Revision Chronology: | | |
|---|---|---|
| 2017N311825_00 | 2017-MAR-06 | Original |
| 2017N311825_01 | 2017-JUN-02 | To address clarifications regarding the aim of the study, the eligibility criteria, the schedule of activities, the clinical assessments, and the recording of lab data and adverse events. The benefit: risk section was also updated based on the Part 2 results from study CNTO7160ASH1001. Also, a few typographical errors were corrected. |
| 2017N311825_02 | 2017-SEP-13 | To add more information on the risk: benefit section and the study design justification sections. To address clarifications regarding the unblinding of treatment in case of emergency. To clarify that rechallenge is not allowed once the treatment discontinuation criteria are met. Also, a few typographical errors were corrected. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Modified Intent to Treat population. | Modified Intent to Treat (Loss of Control), Modified Intent to Treat and Safety excluding GCP noncompliant subjects populations. | The Modified Intent to Treat (Loss of Control) was added to account for the intercurrent event when participants receive the wrong study treatment. Whilst the data from GCP non- compliant participants should not be used in the efficacy analysis, the participants were dosed with GSK3772847 or Placebo so all safety data (AEs, SAEs, ECGs etc.) should be reported. |
| Section 10.4.1 of the protocol describes a sensitivity analysis | A primary and secondary estimand have been defined to | The protocol was approved before the ICH E9 addendum on |

| Protocol Reporting & Analysis Plan | | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| where data is analysed as missing and worst case (loss of control) for participants who withdraw from the study for reasons other than loss of asthma control. Statistical analysis would be | capture where data is analysed as missing and worst case (loss of control) for various intercurrent events where participants withdraw from the study for reasons other than loss of asthma control. Bayesian analysis will include | estimands. The RAP is performing the same planned analysis as detailed in the Protocol however the terminology has been updated in accordance with ICH E9. Bayesian analysis will now |
| performed for each screening eosinophil strata separately. | screening eosinophil strata as a covariate instead of performing split analysis models. In addition, an exploratory analysis using fractional polynomials was added to examine the relationship between loss of control and screening eosinophils (continuous), IgE and FeNO. | include the same covariates as the frequentist analysis. By modelling eosinophils as a continuous endpoint, it will provide more information on the impact of varying screening eosinophil levels on the treatment effect. It will also provide additional information on the role of IgE and FeNO on loss of asthma control. |
| Mixed model repeated measures will be used to analyse the following endpoints. The baseline value of each endpoint will be included along with baseline*visit and treatment*visit interactions. Treatment differences, 95% confidence intervals and p-values will be presented. Change from baseline in ACQ-5 absolute score Change from baseline in SGRQ total score Change from baseline in Pre-bronchodilator FEV <sub>1</sub> Change from baseline in FeNO | FEV <sub>1</sub> and FeNO will only be analysed up until Week 4 (down titration of ICS), all data post Week 4 will be summarised descriptively only. In addition, an exploratory analysis using fractional polynomials was added to examine the relationship between FEV <sub>1</sub> at Week 4 with screening eosinophils (continuous), IgE and FeNO. Continuous ACQ-5 and SGRQ will only be summarised and will not be analysed. Responder analysis will still be performed. This will not impact any of the responder analysis in the primary or secondary endpoints. | FEV1 and FeNO are impacted by ICS, so including change from baseline post-down titration of ICS would be confounding change due to study treatment with change due to ICS. To better explore the data prior to down titration, the fractional polynomial analysis has been added to examine the relationship between FEV1 at Week 4 with screening eosinophils (continuous), IgE and FeNO. FEV1, FeNO, ACQ-5 and SGRQ analysed using an MMRM would be assuming that data is missing at random. In fact, participants could have withdrawn due to loss of asthma control which is related to study treatment, so the analysis assumptions would not have been valid. |
| Secondary endpoints listed as: Serum concentrations of GSK3772847 at weeks 2, 4, 8, 12, 16, 20, 24 and 28. Free and total soluble ST2 levels | Secondary endpoints listed as: Serum concentrations of GSK3772847 by nominal time. Free and total soluble ST2 | Endpoint updated to use nominal time so that all data collected is summarised. |


| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| at weeks 2, 4, 8, 12, 16, 20, 24<br>and 28. | levels in serum by nominal time. | |
| Proportion of participants with loss of asthma control assessed over Weeks 0-16 only. | Proportion of participants with loss of asthma control assessed over Weeks 0-16 and over Weeks 0-6. | An additional endpoint assessing loss of control between Weeks 0 and 6 was added to help support the time to loss of asthma control analysis. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of GSK3772847, compared with placebo, administered intravenously every 4 weeks for 12 weeks (Week 0 – Week 12, 4 doses in total) in participants with moderately severe asthma. | Primary – Proportion of participants with loss of asthma control over Weeks 0-16 where 'loss of asthma control' is defined as at least one of the following: • Asthma Control Questionnaire (ACQ-5) score increase from baseline (measured at the end of Run-in) ≥ 0.5 point or • Pre-bronchodilator Forced expiratory volume in 1 second (FEV1) decrease from baseline (measured at the end of Run-in) >7.5 % or • Inability to titrate inhaled corticosteroid according to the pre-defined schedule or • A clinically significant asthma exacerbation (requiring oral corticosteroid [OCS] and/or hospitalisation). |
| Secondary | |
| To evaluate other aspects of efficacy of GSK3772847 compared with placebo in participants with moderately severe asthma. | <ul> <li>Other efficacy endpoints (at or by Week 16): <ul> <li>Proportion of participants with a ≥0.5 point. ACQ-5 score increase from baseline.</li> <li>Proportion of participants who have prebronchodilator FEV1 decrease from baseline (measured at the end of Run-in) &gt;7.5 %.</li> <li>Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the pre-defined schedule.</li> <li>Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).</li> <li>Proportion of participants with loss of asthma control over Weeks 0-6</li> <li>Time to loss of asthma control.</li> <li>Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule</li> <li>The incidence, mean rate, and total number per participant of hospitalisations or Emergency Room (ER) visits during the study treatment period.</li> </ul> </li> </ul> |

| Objectives | Endpoints |
|---|---|
| Objectives | <ul> <li>Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.</li> <li>Proportion of participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16.</li> <li>Change from baseline in SGRQ total score at Weeks 4, 8, 12 and 16.</li> <li>Proportion of St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16.</li> <li>Change from baseline in pre-bronchodilator FEV1 at Weeks 2, 4, 6, 8, 10, 12, 14, 16.</li> <li>Change from baseline in mean morning</li> </ul> |
| | <ul> <li>peak expiratory flow (PEF) and mean evening PEF over each four weeks of the 16 week treatment period.</li> <li>Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period.</li> <li>Change from baseline in rescue medication use (albuterol/salbutamol): mean number of inhalations per day over each four weeks of the 16 week treatment period.</li> <li>Changes from baseline in night-time awakenings due to asthma symptoms requiring rescue medication use over each four weeks of the 16 week treatment period.</li> <li>Change from baseline in fractional exhaled nitric oxide (FeNO) at each</li> </ul> |
| To evaluate the safety and tolerability of GSK3772847, compared with placebo administered intravenously every 4 weeks for 12 weeks (Week 0-12, 4 doses in total) in participants with moderately severe asthma. | <ul> <li>week measured.</li> <li>Incidence and frequency of adverse events (AEs) and serious adverse events (SAEs).</li> <li>Change from baseline in vital signs at weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24 and 28.</li> <li>Change between post-dose and pre-dose in vital signs at weeks 0, 4, 8 and 12.</li> <li>Change from baseline in 12-lead electrocardiogram (ECG) measurements at weeks 4, 8, 12 and 16.</li> <li>Change between post-dose and pre-dose in 12-lead ECG measurements at weeks 0, 4, 8 and 12.</li> <li>Change from baseline in 24 hours Holter</li> </ul> |

| Objectives | Endnainte |
|---|---|
| Objectives | Endpoints |
| | measurements at weeks 4 and 12. |
| | <ul> <li>Change from baseline in clinical chemistry<br/>at weeks 2, 4, 8, 12, 16 and 28.</li> </ul> |
| | <ul> <li>Change from baseline in haematology and<br/>cardiac markers at weeks 1, 2, 4, 6, 8, 10,<br/>12, 14, 16 and 28.</li> </ul> |
| | <ul> <li>Incidence of and titres of anti- GSK3772847<br/>antibodies at weeks 2, 4, 8, 12, 16, 20, 24<br/>and 28.</li> </ul> |
| To evaluate the pharmacokinetics (PK) of<br>GSK3772847 in participants with moderately<br>severe asthma. | Serum concentrations of GSK3772847 by nominal time. |
| To evaluate the pharmacodynamics (PD) of<br>GSK3772847 in participants with moderately<br>severe asthma. | Free and total soluble ST2 levels in serum by nominal time. |
| Exploratory | |
| To compare the effect of GSK3772847 with placebo on biomarkers in serum and sputum. | <ul> <li>Changes from baseline in induced<br/>sputum biomarkers (subset) at weeks 8<br/>and 16.</li> </ul> |
| | <ul> <li>Changes from baseline in exploratory<br/>serum markers at weeks 8 and 16.</li> </ul> |

### 2.3. Study Design



| Overview | Overview of Study Design and Key Features |
|---|---|
| Interim<br>Analysis | The End of Treatment Phase Analysis will take place after all subjects have completed the week 16 visit, and will be considered an interim analysis for both efficacy and safety. There will be no modifications to dosing regimens, sample size or any other aspects of the trial based on this data, as all study assessments, apart from follow-up, will have already been completed. |
| | assessments, apart norm to low-up, will have already been completed. |

## 2.4. Statistical Hypotheses

The primary null hypothesis ( $H_0$ ) for this study is that the ratio of the proportions of subjects with loss of asthma control from randomisation to Week 16 between GSK3772847 and placebo is unity.

$$H_0$$
:  $\frac{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ GSK3772847}{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ Placebo}=1$ 

The alternative hypothesis  $(H_1)$  for this study is that the ratio of the proportions of subjects with loss of asthma control from randomisation to Week 16 between GSK3772847 and placebo is not unity.

$$H_1$$
:  $\frac{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ GSK3772847}{Proportion\ with\ loss\ of\ asthma\ control\ at\ Week\ 16\ on\ Placebo} 
eq 1$ 

#### 3. PLANNED ANALYSES

## 3.1. End of Treatment Phase Analyses

The End of Treatment Phase Analysis will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the Week 16 visit or the Early Withdrawal visit
- 2. All required database cleaning activities have been completed and database release has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

Due to an inability to lock log forms used for collection of exacerbation data, the end of treatment phase analysis will be considered an interim analysis for both efficacy and safety. Any safety data collected for participants who have completed clinic visits after Week 16 will also be cleaned and included in the analysis.

All participants will have completed the active treatment phase of the study by the time of the interim, so no modifications will be made to the study as a result of the End of Treatment Phase Analysis. The Final Analysis is intended to be an analysis of safety data collected in the Post-Treatment Follow-Up phase.

The sponsor will be unblinded to the results of the analysis.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- All subjects have completed the study.
- All required database cleaning activities for data after Week 16/ Early Withdrawal as well as data collected on log pages have been completed.
- Final database release and database freeze has been declared by Data Management.

No unblinding will take place as part of the final analysis as all participants will have already been unblinded during the End of Treatment Phase Analysis.

#### 4. ANALYSIS POPULATIONS

Some participants are being excluded from the efficacy analyses due to a failure at their site to follow GCP. As these participants received GSK3772847 or placebo during their period of participation, all safety data will be reported.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | The All Subjects Enrolled (ASE) population will consist of all participants who sign the ICF. | <ul><li>Study population</li><li>Reason for withdrawal prior to randomisation</li></ul> |
| Randomised | The randomised population will consist of all participants who were randomised. A participant who is recorded as a screen or run-in failure and also randomised will be considered to be randomised in error provided they have not performed any study assessments. | No formal analysis will<br>be performed on this<br>population |
| Modified Intent-to-<br>Treat excluding<br>GCP non-<br>compliant<br>subjects (Loss of<br>Control) | The Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of Control) (mITT_LoC) will consist of all randomised participants who take at least 1 dose of study treatment, excluding participants where an investigation by GSK has shown that good clinical practice has not been followed. Any participants excluded from this population will | •Efficacy (loss of control) |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | be identified as protocol deviations and listed in a separate output. Participants will be analysed according to the treatment they receive >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. For loss of asthma control, participants will be analysed according to the treatment they were receiving at the time of loss of control. | |
| Modified Intent-to-<br>Treat excluding<br>GCP non-<br>compliant<br>subjects | The Modified Intent-to-Treat excluding GCP non-compliant subjects (mITT) population will consist of all randomised participants who take at least 1 dose of study treatment, excluding participants where an investigation by GSK has shown that good clinical practice has not been followed. Any participants excluded from this population will be identified as protocol deviations and listed in a separate output. Participants will be analysed according to the treatment they receive >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. | Efficacy (all except loss of control) |
| Safety including<br>GCP non-<br>compliant<br>subjects | The Safety (SAFF_ALL) population will consist of all randomised participants who take at least 1 dose of study treatment. Participant will be analysed according to the treatment they receive >=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment. | Study population Inclusion, exclusion and randomisation criteria deviations Participant disposition Safety |
| Pharmacokinetic | The PK population will consist of all randomised participants who received at least one dose of study medication, and for whom at least one pharmacokinetic sample was obtained, analysed and was measurable. | •PK |

### NOTES:

- 1. Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.
- 2. If a participant is inadvertently given both study treatments they will be analysed according to the treatment that they received the more frequently.

#### 4.1. Protocol Deviations

All important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [21-Aug-2017 (Version 1) or later].

- ➤ Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- ➤ This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Note: Inclusion and exclusion criteria deviations are always reported as important.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description Order [1] | |
| G | GSK3772847 10 mg/kg | GSK3772847 | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

• Order represents treatments being presented in TFL, as appropriate.

Treatment comparisons will be displayed as follows using the descriptors as specified:

• GSK3772847 vs Placebo

There were four strata used for the randomisation depending on the participants baseline blood eosinophil count and whether they consented to the sputum sub-study:

- Sputum sub-study and baseline blood eosinophils < 150 cells/μL
- Sputum sub-study and baseline blood eosinophils >=150 cells/μL
- Not sputum sub-study and baseline blood eosinophils < 150 cells/μL
- Not sputum sub-study and baseline blood eosinophils  $\geq 150 \text{ cells/}\mu\text{L}$

Displays will be presented by combining data across all four strata to give the overall estimate of GSK3772847 versus placebo.

Sputum sub-study will not be accounted for within the statistical analysis as the sputum sub-study strata was for monitoring recruitment only.

An additional exploratory analysis using fractional polynomials has been added to further investigate the relationship between loss of control and screening eosinophils and summary statistics on eosinophils will also be provided.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Pre-<br>Screening | Screen<br>Run-in | Day 1<br>(Pre-Dose) | |
| Loss of Asthma Control | | | | |
| Pre-bronchodilator Forced expiratory volume in 1 second (FEV <sub>1</sub> ) | | X | Х | Day 1 |
| Asthma Control Questionnaire (ACQ-5) score | | Χ | X | Day 1 |
| Other Patient Reported Outcomes | 3 | | | |
| St. George's Respiratory Questionnaire (SGRQ) | | | Х | Day 1 |
| Peak Expiratory Flow (PEF) | | | | |
| Mean morning peak expiratory flow (PEF) | | Χ | X | Run-in [1] |
| Mean evening peak expiratory flow (PEF) | | Х | X | Run-in [1] |
| Fractional Exhaled Nitric Oxide (F | eNO) | | | |
| Fractional Exhaled Nitric Oxide (FeNO) | | | Х | Day 1 |
| Symptom Scores | | | | |
| Mean daytime asthma symptom score | | Х | Х | Run-in [1] |
| Night-time awakenings due to asthma symptoms requiring rescue medication | | X | Х | Run-in [1] |

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Pre-<br>Screening | Screen<br>Run-in | Day 1<br>(Pre-Dose) | |
| Rescue Medication | | | | |
| Rescue medication use | | Х | Х | Run-in [1] |
| Mean number of inhalations per day over each four weeks | | Х | Х | Run-in [1] |
| Safety | | | | |
| Vital Signs | | Х | Х | Day 1 |
| 12-lead Electrocardiogram (ECG) measurements | | Х | Х | Day 1 |
| 24 hours Holter measurements | | Х | | Screen/Run in |
| Clinical laboratory tests (haematology and chemistry) | | Х | Х | Day 1 |
| Biomarkers | | | | |
| Induced sputum biomarkers | | | Х | Day 1 |
| Serum biomarkers | | | Х | Day 1 |
| Exploratory serum markers | | | Х | Day 1 |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- [1] Mean over the last 7 days of the run-in period prior to V2. Participants must have at least 4 full days of data (morning and evening) in the last 7 days of run-in to be eligible.

### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site, country, and regions.

| Region | Countries |
|----------------|-----------------------------|
| North America | United States, Canada |
| Latin America | Mexico |
| Eastern Europe | Ukraine, Russian Federation |
| Oceania | Australia |

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Covariates |
|---|---|
| Screening eosinophils | At randomisation participants are stratified according to their baseline peripheral blood eosinophil. Screening eosinophils will be included in both primary and secondary analysis as a categorical variable (<150 cells/µL, >=150 cells/µL). An additional exploratory analysis of the primary endpoint using continuous eosinophils will also be examined. |
| | If the analysis models are unable to converge due to low number of participants with baseline blood eosinophils <150 cells/µL, then screening eosinophil will be re-categorised according to a cut point of 300 cells/µL instead i.e. <300 cells/µL and >=300 cells/µL |

# 5.5. Multiple Comparisons and Multiplicity

As there is a single primary treatment comparison, no adjustment is required for primary comparisons. No adjustments will be made for multiplicity for other endpoints.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety Population including GCP non-compliant subjects population (SAFF\_ALL), unless specified to be on the All Subjects Enrolled (ASE) population.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

## 6.2. Disposition

The study population summary will use the All Subjects Enrolled (ASE) population and show the number of subjects overall who were enrolled, the number of screen failures and the number with each reason for screen failure. It will also show the number of subjects who were randomised and who were in the modified Intent-to-treat (Loss of Control), modified Intent-to-treat, Safety including GCP non-compliant subjects, and PK populations.

For the Safety including GCP non-compliant subjects, reasons for withdrawal summary will show the number and percentage of subjects who completed the study, who withdrew prematurely from the study and who reported each primary and sub-reason for withdrawal.

#### 6.3. Medical Conditions

The number and percentage of subjects reporting each current medical condition will be presented. This table will include a subheading of 'Cardiovascular Risk Factors,' which will summarise the information taken from the cardiac disorders page in the eCRF. All medical conditions must be summarised on this table regardless of frequency. This will be repeated for past medical conditions.

#### 6.4. Concomitant Medications

Non-Asthma medications will be summarised by Anatomical-Therapeutic-Chemical (ATC) level 1 and ingredient. Asthma medications will be summarised by the latest version of the Respiratory Medication Class (RMC), and will be derived for each asthma concomitant medication. Multi-ingredient medications will be presented according to their combination ATC classification rather than the classifications of the ingredients.

Asthma and non-asthma medications will be listed separately. A listing of the relationship between ATC Level 1, ingredient and verbatim text will be produced for non-asthma medications only.
#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint

- Proportion of participants with loss of asthma control over Weeks 0-16
- Proportion of participants with loss of asthma control over Weeks 0-6 (Secondary)

# 7.1.2. Summary Measure

Bayesian Method (Primary): The posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.5 and 0.2 (i.e. a 0%, 25%, 50% and 80% reduction).

Frequentist Method (Supportive): Odds Ratio. The odds of having experienced loss of asthma control on GSK3772847 compared to the odds of having experienced loss of asthma control on placebo.

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the modified Intent to Treat (Loss of Control) population, unless otherwise specified.

## 7.1.4. Strategy for Intercurrent (Post-Randomisation) Events

| Intercurrent Event | Primary Estimand | Secondary Estimand |
|---|---|---|
| Treatment discontinuation due to AE/SAE (not related to loss of asthma control) | Set to missing. | <ul> <li>If the AE/SAE was deemed related to IP then set as an event (i.e. worst case scenario).</li> <li>If the AE/SAE was not deemed related to IP then set to missing.</li> </ul> |
| Death | Set to missing. | <ul> <li>If the death was deemed related to IP then set as an event (i.e. worst case scenario).</li> <li>If the death was not deemed related to IP then set to missing.</li> </ul> |
| Prohibited/ Concomitant medications that could impact patients' asthma control | Use data as is. | Set as an event (i.e. worst case scenario). |
| Non-compliance with FP/SAL, FP or study titration | Use data as is. | Set as an event (i.e. worst case scenario). |
| Continuation in the study after LOC criteria met | Use information from first loss of asthma control. | Use information from first loss of asthma control. |

#### Note:

• Identification of whether an event (AE/SAE/Death) is considered related to IP will be identified

- using the investigator tick box collected on the eCRF.
- If the intercurrent event occurs after loss of asthma control then all information on loss of asthma control will be used.
- Prohibited/ concomitant medications will be identified as protocol deviations within the prohibited/ concomitant medications category and will have text that start with "LoAC"
- Non-compliance FP/SAL, FP or study titration will be identified as compliance <80%, compliance</li>
   ≥ 120% or not changing from FP/SAL or FP doses according to the predetermined schedule.

If any of the following intercurrent events occurs, then all data will be accepted:

Pregnancy
 Accidental unblinding

Whilst it's possible that site staff were unable to administer study drug as they were unable to find a suitable vein, the team felt this would not be caused by the randomised study treatment and the visit would be rescheduled. Therefore, if this occurs all data will be accepted and treated as any other out of window assessment.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Proportion of participants with loss of asthma control over Weeks 0-16
- Proportion of participants with loss of asthma control over Weeks 0-6 (Secondary)

#### **Model Specification**

• The primary endpoint proportion of subjects with loss of asthma control will be analysed for the Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of Control) population using both Bayesian (primary) and Frequentist (supportive) methods.

Bayesian Method (Primary):

- Proc MCMC will be used in order to gain the posterior distribution of the study data combined with a non-information beta(1,1) prior, and screening eosinophil strata included as a covariate.
   Note: This prior is equivalent to one event on both GSK3772847 and Placebo treatment arms.
- Three MCMC chains should be run, with all parameters in the model being assessed for convergence. Each chain will have 10,000 simulations (using a burn-in of 500) and will start with a set seed of 207597 to enable comparison between the main and qc.
- The posterior probabilities that the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo is less than 1.0, 0.75, 0.5 and 0.2 (i.e. a 0%, 25%, 50% and 80% reduction) will be calculated along with the estimated ratio and associated 95%

- credible interval. The 95% credible interval will use the highest posterior density where possible, and if this isn't possible then the 2.5% and 97.5% credible intervals will be reported.
- The posterior median and standard deviation will also be reported together with a 95% credible interval.
- In addition to summary tables a plot of the posterior distribution for the ratio of the proportion of subjects with loss of asthma control on GSK3772847 compared with placebo, along with the proportion of subjects with loss of asthma control on GSK3772847 and placebo separately will be generated.
- This analysis will be repeated for loss of asthma control between Weeks 0 and 6.

#### Frequentist Method (Supportive):

 The proportion of participants with loss of asthma control will be analysed using logistic regression allowing for screening eosinophils strata. It will include fixed effects terms for treatment and screening eosinophil strata.

Fractional Polynomials (Exploratory Analysis for Loss of Control Over Weeks 0-16):

- Screening blood eosinophil count will be transformed using a fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by eosinophil covariate interaction will also be included in the model to allow the magnitude of the interaction (but not the order of the fractional polynomial transformation) to differ with each treatment group). The best fitting model will be selected based on likelihood. The selected best fitting model will be plotted as continuous eosinophil count versus loss of asthma control in each treatment arm. The fit of the model to the raw data will be assessed visually.
- The role of baseline IgE and baseline FeNO (separately) on the effectiveness of GSK3772847 with respect to loss of asthma control will be investigated in a similar way.

#### **Model Checking & Diagnostics**

Bayesian Method (Primary):

- The Markov chain standard error (MCSE) should be compared to the standard deviation of the distribution (SD) to make sure that MCSE/SD ≤ 0.01 for all parameters in the mode.
- The Geweke diagnostic test will be used to check whether the mean estimates have converged by comparing means from the early and later part of the Markov chain using a z-score t-test.
   Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.
- Gelman & Rubin diagnostic checks should be used to assess if the Markov chains have mixed.
- Visual checks on diagnostic plots will be performed to assess:
  - O Has the Markov chain settled down?
  - Are sufficient simulations being run?
  - o Is there sufficient burn-in?
  - o Is the effective sample size large enough?

#### Frequentist Method (Supportive):

None.

#### **Model Results Presentation**

Bayesian Method (Primary):


207597

• The proportions of participants experience loss of asthma control on GSK3772847, Placebo and the ratio of GSK3882747/Placebo will be presented along with their 95% credible interval for all participants combined.

## Frequentist Method (Supportive):

The odds of experiencing loss of asthma control on GSK3772947, Placebo and the odds ratio
will be presented along with the 95% confidence intervals and p-value. This will be presented
for all participants combined.

## Fractional Polynomials (Exploratory Analysis):

 A plot of the relationship between the probability of experiencing loss of control on each treatment as well as the odds ratio versus continuous eosinophils will be produced.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Endpoint and Summary Measure

| Endpoint | Summary Measure |
|---|---|
| Individual Components of Loss of Asthma | |
| <ul> <li>Proportion of participants with a ≥0.5 point. ACQ-5 score increase from baseline.</li> <li>Proportion of participants who have pre-bronchodilator FEV1 decrease from baseline (measured at the end of Run-in) &gt;7.5 %.</li> <li>Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the predefined schedule.</li> <li>Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).</li> <li>Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule</li> </ul> | Frequentist Method (Supportive): Odds Ratio. For each endpoint listed, the odds of having experienced loss of asthma control on GSK3772847 compared to the odds of having experienced loss of asthma control on placebo will be produced. |
| Time to loss of asthma control. | Median and lower and upper quartiles (only calculable if>= 50%, 25%, 75% subjects lose control for each treatment respectively) for time to loss of asthma control |
| The incidence, mean rate, and total number per participant of hospitalisations or Emergency Room (ER) visits during the study treatment period. | Summary statistics and study treatment exposure (no statistical analysis required). |
| Responder Analysis: • Proportion of participants with ≥0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16. • Proportion of St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16. | Odds Ratio. The odds of being a responder on GSK3772847 compared to the odds of being a responder on placebo. |
| Change from Baseline Analysis: Change from baseline in pre-bronchodilator FEV1 at Weeks 2, 4, 6, 8, 10, 12, 14, 16. Change from baseline in fractional | Mean change from baseline |

| Endpoint | Summary Measure |
|---|---|
| exhaled nitric oxide (FeNO) at each week measured. | |
| <ul> <li>Change from Baseline Analysis:</li> <li>Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.</li> <li>Change from baseline in SGRQ total score at Weeks 4, 8, 12 and 16.</li> </ul> | Mean change from baseline |
| <ul> <li>Change from baseline in mean morning peak expiratory flow (PEF) and mean evening PEF for each four week period of the overall 16 week treatment period.</li> <li>Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period.</li> <li>Changes from baseline in night-time awakenings due to asthma symptoms requiring rescue medication use over each four weeks of the 16 week treatment period.</li> <li>Change from baseline in rescue medication use (albuterol/salbutamol): mean number of inhalations per day over each four weeks of the 16 week treatment period.</li> </ul> | Change from baseline (summary statistics only) |

# 7.2.2. Population of Interest

The secondary efficacy analyses will be based on the modified Intent to Treat population, unless otherwise specified.

# 7.2.3. Strategy for Intercurrent (Post-Randomisation) Events

For components of Loss of Asthma Control see Section 7.1.4.

For SGRQ and ACQ Responders primary and secondary estimands as table below:

| Intercurrent Event | Primary Estimand | Secondary Estimand |
|---|---|---|
| to AE/SAE (not related to loss | _ | If the AE/SAE was deemed related to IP then set as non-responder. |
| of asthma control) | | <ul> <li>If the AE/SAE was not deemed related to IP<br/>then set to missing.</li> </ul> |

| Intercurrent Event | Primary Estimand | Secondary Estimand |
|---|---|---|
| Death | Set to missing. | <ul> <li>If the death was deemed related to IP then set as non-responder.</li> <li>If the death was not deemed related to IP then set to missing.</li> </ul> |
| Prohibited/ Concomitant medications that could impact patients' asthma control | Use data as is. | Set as non-responder. |
| Non-compliance with FP/SAL, FP or study titration | Use data as is. | Set as non-responder. |

#### Note:

- Identification of whether an event (AE/SAE/Death) is considered related to IP will be identified
  using the investigator tick box collected on the eCRF.
- If the intercurrent event occurs after loss of asthma control then all information on loss of asthma control will be used.
- Prohibited/ concomitant medications will be identified as protocol deviations within the prohibited/ concomitant medications category and will have text that start with "LoAC"
- Non-compliance FP/SAL, FP or study titration will be identified as compliance <80%, compliance ≥ 120% or not changing from FP/SAL or FP doses according to the predetermined schedule.

## 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Proportion of participants with a ≥0.5 point. ACQ-5 score increase from baseline.
- Proportion of participants who have pre-bronchodilator FEV1 decrease from baseline (measured at the end of Run-in) >7.5 %.
- Proportion of participants where inhaled corticosteroids (ICS) cannot be titrated in accordance with the pre-defined schedule.
- Proportion of participants who have a significant asthma exacerbation (requiring OCS and/or hospitalisation).
- Proportion of participants with a clinically significant asthma exacerbation or inability to titrate ICS according to the pre-defined schedule

## Strategy for Intercurrent (Post-Randomisation) Events

Both primary and secondary estimands (Section 7.1.4) will be examined. It is important to assess both estimands as data is set to missing after withdrawal or loss of asthma control. This could produce biased estimands, as loss of control and therefore missing data is related to study treatment, and so the secondary estimand where missing data is set as non-responders must also be considered.

#### **Model Specification**

See Section 7.1.5.1.

# **Model Checking & Diagnostics**

• See Section 7.1.5.1

#### **Model Results Presentation**

See Section 7.1.5.1

## **Endpoint / Variables**

- Proportion of participants with ≥ 0.5 point ACQ-5 score decrease from baseline (responder) at each week from Week 1 to Week 16.
- Proportion of St. George's Respiratory Questionnaire (SGRQ) responders (at least a 4 unit improvement from baseline) at Weeks 4, 8, 12 and 16.

#### Strategy for Intercurrent (Post-Randomisation) Events

Both primary and secondary estimands (Section 7.2.3) will be examined. It is important to assess both estimands as data is missing after withdrawal or loss of asthma control. This could produce biased estimands, as loss of control and therefore missing data is related to study treatment, and so the secondary estimand where missing data is set as non-responders must also be considered.

#### **Model Specification**

- The proportion of participants who were responders will be analysed using logistic regression allowing for screening eosinophils strata.
- A responder on ACQ-5 is defined as participants with a ≥ 0.5 point decrease from baseline whilst a responder on SGRQ is defined as a ≥ 4 point decrease from baseline.
- This endpoint will be analysed using logistic regression. Treatment, eosinophil strata will be fixed effects.

#### **Model Checking & Diagnostics**

None

#### **Model Results Presentation**

• The odds of being a responder (as defined above) on GSK3772947, Placebo and the odds ratio will be presented along with the 95% confidence intervals and p-value.

#### **Endpoint / Variables**

Time to loss of asthma control.

## Strategy for Intercurrent (Post-Randomisation) Events

Both primary and secondary estimands (Section 7.1.4) will be examined. It is important to
assess both estimands as data is missing after withdrawal or loss of asthma control. This
could produce biased estimands, as loss of control and therefore missing data is related to
study treatment, and so the secondary estimand where missing data is set as nonresponders must also be considered.

## **Model Specification**

Time to loss of asthma control will be analysed on the Modified Intent-to-Treat excluding GCP

non-compliant subjects (Loss of Control) population using Kaplan-Meier analysis (Proc lifetest). Within the Kaplan Meier plot participants will either be counted as an event or they will be censored.

#### Events:

Participants who experience loss of asthma control during the study.

#### Censoring:

- Participants who discontinue investigational product for reasons other than loss of asthma control.
- Participants who successfully complete the 16 week treatment period will be censored at 113 days (16 weeks + 1 day).

Time to loss of asthma control = Date of loss of asthma control – Treatment start date + 1. If participants experience multiple reasons for loss of control then the earliest date will be used as described in Section 12.6.3.

#### **Model Checking & Diagnostics**

None

#### **Model Results Presentation**

- Kaplan-Meier plots of the probability of a participant experiencing loss of asthma control by treatment will be produced.
- In addition, a summary table will be produced showing the probability of experiencing loss of asthma control after 4, 8, 12 and 16 weeks along with the median time (this will be NA if <50% of participants on a treatment lose control) to loss of asthma control on both treatment arms.

#### **Endpoint / Variables**

- Change from baseline in pre-bronchodilator FEV<sub>1</sub> at Weeks 2, 4, 6, 8, 10, 12, 14, 16.
- Change from baseline in fractional exhaled nitric oxide (FeNO) at each week measured.
- Change from baseline in blood eosinophils

#### **Strategy for Intercurrent (Post-Randomisation) Events**

No intercurrent events are considered for this endpoint. All data will be used as collected.

#### Model Specification

Only data until Week 4 (down titration of ICS) will be analysed, all data post Week 4 will be summarised descriptively only.

Data up to and include Week 4 (down titration of ICS):

A repeated measures model with terms for treatment, visit, visit by treatment and screening eosinophil strata will be included along with the screening eosinophil strata\*visit and treatment\*visit interactions.

FEV<sub>1</sub> at Weeks 4 Only - Fractional Polynomials (Exploratory Analysis):

 Screening blood eosinophil count will be transformed using a fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by eosinophil covariate interaction will also be included in the model to allow the magnitude of the interaction (but not the order of the fractional polynomial transformation) to differ with each treatment group). The best fitting model will be selected based on likelihood. The selected best fitting model will be plotted as continuous eosinophil count versus loss of asthma control in each treatment arm. The fit of the model to the raw data will be assessed visually.

• The role of baseline IgE and baseline FeNO (separately) on the effectiveness of GSK3772847 with respect to FEV<sub>1</sub> at Weeks 4 will be investigated in a similar way.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

• The estimates of the mean and difference for each treatment group from the model will be produced, along with 95% confidence intervals and p-values for treatment comparisons.

The following endpoints will be summarised descriptively only. No analysis will be performed and all data will be reported as collected (no intercurrent events will be considered) using the modified Intent to Treat population:

- Change from baseline in ACQ-5 absolute score at each week from Week 1 to Week 16.
- Change from baseline in SGRQ total score at Weeks 4, 8, 12 and 16.
- Change from baseline in mean morning peak expiratory flow (PEF) and mean evening PEF over each four weeks of the 16 week treatment period.
- Change from baseline in mean daytime asthma symptom score over each four weeks of the 16 week treatment period.
- Changes from baseline in night-time awakenings due to asthma symptoms requiring rescue medication use over each four weeks of the 16 week treatment period.
- Change from baseline in rescue medication use (albuterol/salbutamol): mean number of inhalations per day over each four weeks of the 16 week treatment period.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety including GCP non-compliant subjects population, unless otherwise specified. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards.

# 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.

# 8.3. Vital Signs, Electrocardiogram (ECG) and Holter

Summary statistics for vital signs at baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24 and 28 will be produced along with change from baseline summaries for each post baseline timepoint. In addition, the change between post-dose and pre-dose vital signs measurements will be summarised at weeks 0, 4, 8 and 12.

Similar 12-lead electrocardiogram (ECG) measurements at baseline, weeks 4, 8, 12 and 16 will be produced along with change from baseline summaries for each post baseline timepoint, and changes between post-dose and pre-dose in 12-lead ECG measurements at weeks 0, 4, 8 and 12.

24 hour Holter measurements collected at baseline, weeks 4 and 12 will be summarised along with change from baseline at weeks 4 and 12. Only participants with at least 16hrs worth of data will be included in any tables however all data will be listed.

# 8.4. Clinical Chemistry, Haematology and Cardiac Markers

Summaries of clinical chemistry results at baseline, weeks 2, 4, 8, 12, 16 and 28 along with change from baseline for all post-baseline measurements will be produced.

Similarly, haematology and cardiac markers at baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28 along with change from baseline for all post-baseline measurements will also be produced.

#### 8.5. Antibodies

Summaries of the incidence of and titres of anti- GSK3772847 antibodies at weeks 0\*, 2, 4\*, 8\*, 12\*, 16, 20, 24 and 26.

<sup>\* =</sup> Pre-dose only

## 8.6. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of liver function tests will be based on GSK Core Data Standards.

#### 9. PHARMACOKINETIC ANALYSES

Due to the time required to analyse PK samples, no PK outputs will be included in the end of treatment phases analysis.

# 9.1. Secondary Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

Serum concentrations of GSK3772847 by nominal time.

## 9.1.2. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 9.1.3. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

## 9.1.4. Statistical Analyses / Methods

- No statistical analysis will be performed.
- Serum concentration will be summarised descriptively with summary figures being produced.
- Scatter plots of trough serum concentration vs FeNO, trough serum concentration vs blood eosinophils, and trough serum concentration vs IgE at Week 4 only will also be produced.

#### 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

# 10.1. Secondary Pharmacodynamic Analyses

#### 10.1.1. Endpoint / Variables

Free and total soluble ST2 levels in serum

## 10.1.2. Summary Measure

Free soluble ST2: Summary statistics and percentage change from baseline

Total soluble ST2: Summary statistics and change from baseline

Only pre-dose trough sST2 will be used for analysis. Post-dose trough sST2 will be summarised only.

# 10.1.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the modified Intent to Treat population, unless otherwise specified.

## 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

# 10.1.5. Statistical Analyses / Methods

#### **Endpoint / Variables**

- Percentage change from baseline in free sST2 (On-treatment)
- Percentage change from baseline in free sST2 (Post-treatment)

## Strategy for Intercurrent (Post-Randomisation) Events

No intercurrent events are considered for this endpoint. All data will be used as collected.

#### Model Specification

- The ratio of post-baseline sST2 values to baseline sST2 values will be log transformed prior to analysis. Note: Log(post baseline sST2 /baseline sST2) is equivalent to log(post baseline sST2) – log(baseline sST2).
- A repeated measures model with terms for treatment, visit, visit by treatment, the logarithm of baseline sST2, the logarithm of baseline sST2 by visit and screening eosinophil strata will be fitted.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

• The estimated treatment ratios together with 95% CIs (back-transformed from the differences on the log-scale).

#### **Endpoint / Variables**

- Change from baseline in free sST2 (On-treatment)
- Change from baseline in free sST2 (Post-treatment)

#### **Strategy for Intercurrent (Post-Randomisation) Events**

No intercurrent events are considered for this endpoint. All data will be used as collected.

#### **Model Specification**

 A repeated measures model with terms for treatment, visit, visit by treatment, baseline sST2, baseline sST2 by visit and screening eosinophil strata will be fitted.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analysis will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
values (i.e. checking the normality assumption and constant variance assumption of the model
respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

• The estimates of the mean and difference for each treatment group from the model will be produced, along with 95% confidence intervals and p-values for treatment comparisons.

## Fractional Polynomials (Exploratory Analysis)

The role of free sST2 on the effectiveness of GSK3772847 with respect to loss of asthma control will be investigated, using the modified intent to treat population. The number of participants experiencing loss of control will be predicted at each level of baseline free sST2 based on a model including a free sST2 main effect term and an interaction with treatment term.

Baseline free sST2 will be transformed using a fractional polynomial term which will be included in the model as a continuous covariate. A treatment group by free sST2 covariate interaction will also be included in the model to allow the magnitude of the interaction (but not the order of the fractional polynomial transformation) to differ with each treatment group. The best fitting model will be selected based on likelihood. The selected best fitting model will be plotted as continuous free sST2 versus loss of asthma control in each treatment arm. The fit of the model to the raw data will be assessed visually.

# 10.2. Exploratory Biomarker Analyses

# 10.2.1. Endpoint / Variables

- Changes from baseline in induced sputum biomarkers (subset) at weeks 8 and 16.
- Changes from baseline in exploratory serum markers at weeks 8 and 16.

#### 10.2.2. Summary Measure

Change from baseline

## 10.2.3. Population of Interest

The exploratory biomarker analyses will be based on the modified Intent to Treat population, unless otherwise specified.

## 10.2.4. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

# 10.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Induced sputum biomarkers and exploratory serum markers at weeks 8 and 16 will be summarised using descriptive statistics, including the geometric mean and CV as well as listed.

No statistical analysis will be performed on this data.

## 11. REFERENCES

Charter for the Internal Safety Review Commitee (iSRC), Protocol 207597 Title: A randomised, double-blind, parallel group, multicenter, stratified study assessing the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with severe asthma, 26 June 2017

GlaxoSmithKline Document Number 2017N311825\_02, Protocol: A randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma, 13 September 2017

Internal Safety Review Commitee (iSRC) Reporting and Analysis Plan for a randomised, double-blind, parallel group, multicenter, stratified study evaluating the efficacy and safety of repeat doses of GSK3772847 compared with placebo in participants with moderately severe asthma, 20 July 2018

Protocol Deviation Management Plan (PDMP), Version 01, 21 August 2017

Winthrop et al, 2015, Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance, Annals of the Rheumatoid Arthritis Disease, doi: 10.1136/annrheumdis-2015-207841. Epub 2015 Sep 22

# 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management

The full list of protocol deviations collected on the eCRF is in the PDMP. Please refer to this document for current guidance.

There is no per protocol population in this study.

# 12.2. Appendix 2: Schedule of Activities

# 12.2.1. Protocol Defined Schedule of Events

| Procedure | Pre-<br>Screen | Scree<br>n Run- | FOILOW IID MOLLOGE | | | | | | | eriod <sup>2</sup> | Notes | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | 0 1 23 3 4 5 6 7 8 9 10 (ETP or EW) | 1111 | 1 | £ 2 day | s | | | | ± 3 da | ays | | | | ± 3 day | | Notes |
| Visit | | 12 | 13 | 14 | Pre-screening and screening can occur on the same day FU period to start 4 weeks after ETP or EW visit. | | | | | | | | | | | |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | <i>u j.</i> |
| Informed consent<br>(ICF) | х | | | | | | | | | | | 31 | | | | |
| Genetic ICF | | X | | | | | | | | | | 4. | 4 | | | |
| F for sputum X | X | 07 | | | | | | | | | | ļ | | | | |
| Inclusion and exclusion criteria | | Х | | | | | | | | | | | | | | |
| Randomisation<br>Criteria | | | X | | | | | | | | 20 | | | | | |
| Demography | X | | | | | | | | | | | | | | | |
| Full physical exam<br>including height and<br>weight | | х | | | | | | | | | | | | | | |
| Medical history<br>(includes substance<br>abuse) | | х | | | | | | | | | | | | | | Substances [Drugs, Alcohol,<br>tobacco] and family history of<br>premature CV disease]):<br>[including cardiovascular<br>medical history] |

| December | Pre- | Scree | | | | Tr | eatme | nt Per | iod | | | | Follo | ow-up F | eriod <sup>2</sup> | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screen<br>ing <sup>1</sup> | n Run-<br>in | 4 | 2 day | s | | | | ± 3 da | ays | | | | ± 3 day | (s) | Notes | |
| | 11 (570) | 12 | 13 | 14 | 1.Pre-screening and screening<br>can occur on the same day 2. FU period to start 4 weeks<br>after ETP or EW visit. 2. Nort 3 - Day 4 (first doos of | | | | | | | | | | | | |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 24 2 | 20 24 | 20 24 | 28 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | <i>j.</i> | |
| Laboratory<br>assessments | | X1, 2 | Χı | х | Χ¹ | Χ¹ | х | Χ¹ | х | Χ¹ | х | Χ¹ | | | Xı | Haematology (including eosinophil count) and cardiac markers measured at all clinic visits. 1. Clinical chemistry (including liver chemistry). 2. Routine urinalysis at screening (Visit 1) | |
| Pregnancy test <sup>1</sup> | х | ē. | X3 | | | X3 | | X3 | | X3 | | х | х | х | х | 1. Test for women with child bearing potential. 2. Serum pregnancy test at V0/V1. 3. Test to be performed predose during the treatment period. | |
| [HIV, Hep B and Hep<br>C screen] | | х | | | | | | | | | | | | XI. | | A confirmatory negative Hepatitis C RNA test must be obtained, to be able to enrol participants with positive Hepatitis C antibody due to prior resolved disease. If test has been performed within 3 months prior to first dose of study treatment, testing at screening is not required. | |

| Describes | Pre- | Scree | Treatment Period | | | | | | | Follo | ow-up l | Period <sup>2</sup> | Notes | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screen<br>ing <sup>1</sup> | n Run- | 1 | 2 day | s | | | | ± 3 da | ays | | | 10 | (± 3 da | ys) | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 8 9 10 (ETP or 12 13 14 can occur on the 2. FU period to after ETP or EV | | 1.Pre-screening and screening can occur on the same day 2. FU period to start 4 weeks after ETP or EW visit. | | | | | | |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 24 | 20 24 28 | 0 24 | 3. Visit 2 = Day 1 (first dose of IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | 1F). |
| Genetic blood sample<br>– Pre dose | | | | | | | - | х | | | 23.1 | EN: | | | | Pharmacogenetic sample may<br>be drawn any time from Visit 2<br>onwards. Informed consent for<br>optional substudies e.g.<br>genetics must be obtained<br>before collecting a sample |
| Sputum sample collection | | | Х | | | | | x | | | | х | | | | Pre-dose collection and in a<br>sub-set of participants (~50 %)<br>at selected sites; also collected<br>for EW participants |
| PK, target<br>engagement and<br>immunogenicity<br>assessments | | | X | х | Х | х | | x | | х | | х | χ | x | х | See SoA Table 2 for details |
| Exploratory<br>Biomarkers | | | X | | | | | X | | | | Х | | | | Pre dose collection |
| Efficacy | | ġ ; | 0 - 3 | | | 3 3 | | i 8 | - 1 | | 3 | 3 | | 9 | ğ | <u> </u> |
| Spirometry | | Х | Χ | | Х | Х | Х | X | Х | Х | χ | Х | | | | Test to be performed pre-dose<br>during the Treatment period |
| Reversibility | | X | | | - 3 | | | | 3 | | | | | | | |
| FeNO | | | X | Х | Х | Х | Х | X | Х | Х | Х | Х | | | 8 | Test to be performed pre-dose |
| Review loss of<br>asthma control<br>criteria | | | | х | Х | х | Х | х | Х | Х | Х | х | | | | It will include review of data to<br>determine loss of asthma<br>control. See Section 9.1.5. |
| Dispense eDiary | | Х | | | | | | | * | | 20 | * | 0.0 | | | |

| Procedure | Pre-<br>Screen | Scree<br>n Run- | ( S | | | Tr | eatme | nt Per | riod | | | | Follo | Follow-up Period <sup>2</sup> | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ingt | in | <u>, 4</u> | 2 day | s | | | v - v: | ± 3 da | ays | 53 | 53 | | ±3 da | ys) | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | 1.Pre-screening and screening can occur on the same day 2. FU period to start 4 weeks after ETP or EW visit. 3. Visit 2 = Day 1 (first dose of |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | IF). |
| Collect eDiary | | | 8 3 | | 3 | | | | 3 | | | X | | | | |
| Review eDiary | | | X | Х | Х | Х | Х | X | Х | Х | Х | X | ). | | | Į. |
| Safety | 20 | | | | | | · | | | | | 22- | vii. | 410 | | • The Research 1997 |
| 12-lead ECG | | х | Χ¹ | | | X1 | | X1 | | X¹ | | х | | | | Test to be performed pre-<br>dose and post-dose within 30<br>mins after end of infusion. |
| 24 hrs Holter | | х | Хі | | | Χ¹ | | | | Χ¹ | | | | | | Holter monitor needs to be returned to clinic at end of 24-hour recording (i.e. the next day). 1. Place the Holter 30-60 mins prior to dosing. |
| Vital signs | | х | Χ¹ | х | Х | Х1 | х | Χı | Х | X1 | Х | х | Х | х | х | Test to be performed pre-<br>dose prior to spirometry and<br>post-dose prior the 12 -lead<br>ECG. |
| Dispense paper<br>Medical<br>Problems/Medication<br>s Taken worksheet | | х | X | X | x | х | х | x | Х | х | х | Х | х | х | | |
| Review paper<br>Medical<br>Problems/Medication<br>s Taken worksheet | | | х | х | х | х | Х | х | х | х | х | х | х | х | х | |

| Procedure | Pre-<br>Screen | Scree<br>n Run- | | Treatment Period | | | | | | | | Follo | ow-up | Period <sup>2</sup> | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ing <sup>1</sup> | | in | 4 | 2 day | s | | | | ± 3 da | ays | | | | (± 3 da | ys) | Notes |
| Visit | 0 | 1 | 23 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11<br>(ETP<br>or<br>EW) | 12 | 13 | 14 | 1.Pre-screening and screening can occur on the same day 2. FU period to start 4 weeks after ETP or EW visit. 3. Visit 2 = Day 1 (first dose of |
| Week | -4~-2 | -2 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | IP). |
| Study Day | -28~-14 | -14 | 1 | 8 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | | | | 11 J. |
| AE/SAE review | Χ¹ | Χ¹ | | <b>←===</b> | | | | | | | | <b>&gt;</b> | х | х | х | At V0 and V1 collect only<br>SAEs considered as related to<br>study participation. |
| Concomitant<br>medication review | X | Х | | <b>←===</b> | | | | | | | | <b>→</b> | Х | Х | Х | |
| Questionnaires | 8 1 | 8 3 | | | | | | | | | | | 565<br>10. | \$6<br>10. | Š | ë |
| ACQ-5 | | х | | | | | 2 | X | | | | | | | | After randomization, ACQ5 will<br>be completed by the<br>participants every 7 days. |
| SGRQ | | | X | | | X | | X | | X | 88 | Х | | | | |
| Study Treatment | 40 0 | | | | | | | | | 50.10. | -01 | -51 | A11 | 40 | - | |
| Double blind Study<br>Treatment (IP) | | | х | | | х | | х | | х | | | | | | Patients will remain in the clinic<br>for monitoring for at least 2<br>hours after the end of infusion. |
| FP/Sal (500/50)<br>dispensing | | х | Х | | | | | | | | | | | | | |
| FP (mcg) dispensing | | | | | 500 | 250 | 100 | 50 | | | | | 0. | | | |
| Dispense albuterol<br>(as needed) | | X. | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | | | 175 | |

| Dragadura | | | -0 | 0 | Treatn | nent Peri | od | | | | F | ollow-up | ) <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | ± 2 days | 5 | 4 | | | ±3 day | | ± 3 days | Notes | | | | |
| Visit | 21 3 4 5 6 7 | 8 | 8 9 | 10 | 11<br>(ETP<br>or EW) | 12 | 13 | 14 | Visit 2 = Day 1 (first dose of IP). FU period to start | | | | | |
| Week | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 20 | 24 | 28 | 4 weeks after ETP of<br>EW visit. |
| Study Day | 1 | 8 | 15 | 29 | 43 | 49 | 71 | 85 | 99 | 113 | | | | EVV VISIL |
| Double blind<br>Study<br>Treatment<br>(IP) | X | | | X | | х | | x | | | | | | |
| PK sample | X2 | X | X | X3 | | X3 | | χ1 | | X | X | X | X | 1. Pre dose and |
| Free and total<br>sST2 | X1 | Х | Х | X3 | | X3 | | X1 | | X | Х | Х | X | post dose. 2. Post dose only. |
| Immunogenicit<br>y sam <mark>p</mark> le | X3 | | X | Χ3 | | Хз | | Х3 | | X | х | х | х | 3. Pre dose only. Pre-dose samples within 2 hours from the planned dosing time. Post-dose samples as soon as possible after end of infusion but must be taken within 4 hours. |

# 12.3. Appendix 3: Assessment Windows

# 12.3.1. Definitions of Assessment Windows for Analyses

Nominal visits will be used and no windowing will be applied for analysis.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 28 days |
| Post-Treatment | Date > Study Treatment Stop Date + 28 days |

Completion of study epoch's will be defined as the following:

| Study Phase | Definition of Completion |
|---|---|
| Run-in | Randomised into study and received first dose of study treatment |
| Treatment | Completed Week 16 visit or withdrew from treatment phase due to loss of asthma control |
| Follow up | Completed 12 week follow-up period |

# 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| Pre-Treatment | <ul> <li>Conmed Start Date &lt; Study Treatment First Dose Date</li> <li>Conmed End Date &lt; Study Treatment First Dose Date</li> <li>CMSTRF = "BEFORE"</li> <li>Randomisation date is missing i.e. subject was not randomised</li> </ul> |
| On-Treatment | <ul> <li>Study Treatment First Dose Date &lt;= Conmed Start Date &lt;= Study Treatment Last Dose Date + 28</li> <li>Study Treatment First Dose Date &lt;= Conmed End Date &lt;= Study Treatment Last Dose Date + 28</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (CMENRF ="DURING/AFTER" or CMENRF ="AFTER" or CMSTRF = "DURING")</li> <li>(CMSTRF = "BEFORE" or CMSTRF = "DURING" or CMENRF = "DURING/AFTER") and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(CMSTRF = "BEFORE" or CMSTRF ="DURING") and (CMENRF = "DURING/AFTER" or CMENRF = "AFTER")</li> <li>CMSTRF = "DURING"</li> <li>CMSTRF = "DURING/AFTER"</li> </ul> |

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| Post-Treatment | <ul> <li>Conmed Start Date &gt; Study Treatment Last Dose Date + 28</li> <li>Conmed End Date &gt; Study Treatment Last Dose Date + 28</li> <li>CMENRF = "AFTER"</li> <li>CMENRF = "DURING/AFTER"</li> </ul> |
| All phases | Conmed start date is missing and CMSTRF is missing and conmed end date is missing and CMENRF is missing |

#### NOTES:

- The duration of a single concomitant medication can extend over multiple study phases
- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 12.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date + |
| Emergent | 28 days. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 28 days |

#### NOTES:

If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

# 12.5.1. Reporting Process

## Software

The currently supported versions of SAS software will be used.

#### **Reporting Area**

HARP Compound : /arenv/arprod/gsk3772847/mid207597/

Additional information of reporting areas:

data\_look\_01

This is where the blinded dry run will take place.

final 01:

This is where the end of treatment phase analysis will take place.

final 02:

This is where the end of study analysis will take place.

Details of the reporting efforts used for the iSRC analysis are detailed in the separate iSRC RAP.

#### **Analysis Datasets**

Analysis datasets will be created according to CDISC standards

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts

## 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be

adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| 7 til driserieddied visits will be friedded i'r fistirigs. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |

Refer to IDSL Statistical Principals 7.01 to 7.13.

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 12.3.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 12.6.2. Study Population

#### Age

Date of birth will be set as YYYY where YYYY is the year of birth taken from the CRF. For participants who attended a screening visit, age will be calculated at the screening visit date. For pre-screen failures, age will be calculated at the pre-screening visit date.

#### **Body Mass Index (BMI)**

BMI = Weight (kg) / Height(m)<sup>2</sup>

#### **Treatment Misallocations**

To allocate treatment, the number of doses of GSK3772847 and Placebo that were given will be calculated, and the subject will be assigned to whichever treatment has the higher number. The only exception will be when both treatments were given equally, in which case the subject will be assigned their randomised treatment.

#### Treatment Compliance for Fluticasone Propionate (FP) and Salmeterol (SAL)

• Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)\*100

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are
  events of overdose. Cumulative compliance (since Day 1) by each background therapy will be
  calculated.
- Planned Treatment Duration is defined according to the schedule of activities.
- Compliance will be summarized by the following categories:
  - <80%,
  - $\geq$  80% to < 95%,
  - $\geq$ 95% to <105%,
  - ≥ 105% to <120% and
  - ≥120%

#### **Extent of Exposure (Therapeutic Coverage)**

- IP is administered approximately every 4 weeks and each dose viewed as providing therapeutic coverage for 4 weeks (28 days).
- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Study Treatment Last Dose Date (Study Treatment First Dose Date) + 29
- The only exception to this will be when a participant dies in which case
   Duration of Exposure in Days = Death Date (Study Treatment First Dose Date) + 1

## **12.6.3.** Efficacy

#### **Loss of Asthma Control**

#### **Multiple Loss of Asthma Control**

• If a participant reaches loss of control for multiple reasons then all reasons will be reported. For any time to loss of asthma control analysis, the time of the earliest component of loss of control will be used.

#### Time of Loss of Asthma Control

Time to loss of control will be taken from the loss of control log page.

#### 12.6.4. Safety

#### **Adverse Events**

#### **Adverse Events of Special Interest (AESI)**

Systemic Allergic/Hypersensitivity and Non-allergic Reactions:

Systemic allergic/hypersensitivity and non-allergic reactions are identifying through preferred terms which had been selected by medical review of the MedDRA dictionary and are provided in a separate spreadsheet.

Alterations in immune response (infections)

All infections and serious infections reported under the MedDRA system organ class of 'Infections and Infestations'. Specific events of interest are opportunistic infections with preferred terms matching identified/pre-determined terms based on a published list of pathogens and/or presentations of specific pathogens to be considered as opportunistic infections in the setting of biologic therapy [Winthrop, 2015].

Alterations in immune response (malignancies):

All neoplasms reported under the MedDRA system organ class of 'Neoplasms, benign, malignant and unspecified (including cysts and polyps)'. Specific events of interest are malignancies which will be identified through matching of collected preferred terms with those from the following:

Sub-SMQs under the Malignancies SMQ:

- Malignant tumours sub-SMQ (narrow terms)
- Tumours of unspecified malignancy sub-SMQ (narrow terms)

Alterations in cardiovascular safety:

Cardiac disorders and serious cardiac disorders reported under the MedDRA system organ class of 'Cardiac Disorders'. Serious cardiac, vascular and thromboembolic (CVT) events, identified as all serious events classified under the MedDRA system organ classes of 'Cardiac Disorders' and of 'Vascular Disorders', and thromboembolic events identified through matching of collected preferred terms with those from the following:

Sub-SMQs under the Embolic and thrombotic events SMQ:

- Embolic and thrombotic events, arterial sub-SMQ (narrow terms)
- Embolic and thrombotic events, venous sub-SMQ (narrow terms)
- Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous sub-SMQ (narrow terms)

Sub-SMQs under the Ischaemic Heart Disease SMQ

- Myocardial infarction sub-SMQ (narrow terms)
- Other Ischaemic heart disease sub-SMQ (narrow terms)

Sub-SMQs under the Central Nervous System Vascular Disorders SMQ

- Ischaemic central nervous system vascular conditions sub-SMQ (narrow terms)
- Central nervous system vascular disorders, not specified as haemorrhagic or ischaemic sub-SMQ (narrow terms)
- Serious ischemic adverse events, a subset of the serious CVT events identified through matching of collected preferred terms with those from the following:

Local Injection Site Reactions

Local injection site reactions are identifying through preferred terms which had been selected by medical review of the MedDRA dictionary and are provided in a separate spreadsheet.

#### Rate of Events per 1000 Treatment Years

Rate of events per 1000 treatment years will be calculated using:

Rate = number of events \* 1000 / total treatment exposure in years where subjects can contribute more than one event.

This is equivalent to:

Rate = number of events \* 1000 / (number of subjects in treatment group \* mean treatment exposure in years).

#### Maximum/Minimum On-Treatment Definitions for Vital Signs Data

Maximum and Minimum on-treatment: Maximum and Minimum on-treatment value over all time-points (including scheduled and unscheduled assessments) will be presented.

#### FEV<sub>1</sub>

#### **Absolute Reversibility**

Absolute reversibility (mL) = (post-bronchodilator  $FEV_1$  – pre-bronchodilator  $FEV_1$ )

#### **Percent Reversibility**

Definition of Percentage Reversibility as a percentage of predicted  $FEV_1$  = ((post-bronchodilator  $FEV_1$ – pre-bronchodilator  $FEV_1$ ) / predicted  $FEV_1$ ) x 100%

Definition of Percentage Reversibility as a percentage of pre-bronchodilator  $FEV_1$  = ((post-bronchodilator  $FEV_1$ ) / pre-bronchodilator  $FEV_1$ ) x 100%

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as either completing the 16 week treatment period and three month safety follow up, or withdrawing from the treatment period early due to loss of asthma control and completing the three month safety follow up period. |
| | <ul> <li>Withdrawn participants were not replaced in the study, unless the participants were<br/>withdrawn due to sites failing to comply with GCP.</li> </ul> |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | <ul> <li>Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be<br/>summarised as withdrawal visits.</li> </ul> |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated by the use of a "blank" in subject listing displays. |
| | Unless all data for a specific visit are missing in which case the data is excluded from the table. |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Analysis | <ul> <li>All missing data will be handled according to estimand of interest as described<br/>within the main body of the RAP.</li> </ul> |
| ACQ | If one of the five items in the ACQ is missing then the response from the four remaining items will be interpolated (pro-rata) to gain the overall response for the participant. |
| | If more than one item is missing then the ACQ will be considered missing. |
| SGRQ | The SGRQ questionnaire has three components; symptoms, activity and impact. |
| | Symptoms |
| | The Symptoms component will tolerate a maximum of 2 missed items. The weight for the missed item is subtracted from the total possible weight for the Symptoms component (662.5) and from the Total weight (3989.4) |
| | Activity |
| | <ul> <li>The Activity component will tolerate a maximum of 4 missed items. The weight for the missed item is subtracted from the total possible weight for the Activity component (1209.1) and from the Total weight (3989.4)</li> </ul> |
| | Impacts |
| | The Impacts component will tolerate a maximum of 6 missed items. The weight for the missed item is subtracted from the total possible weight for the Impacts component (2117.8) and from the Total weight (3989.4) |
| | If any component has more missing items then mentioned above then the SGRQ will be considered missing. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | Missing Start Day: First of the month will be used unless this is before the start<br>date of study treatment; in this case the study treatment start date will be used and<br>hence the event is considered On-treatment as per Appendix 4: Study Phases and<br>Treatment Emergent Adverse Events. |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

## CONFIDENTIAL

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

Values of potential clinical importance will not be used in this study, instead normal reference ranges of "Low", "Normal" and "High" will be used.
## 12.9. Appendix 9: Abbreviations & Trade Marks

#### 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| mIT | Modified Intent-to-Treat excluding GCP non-compliant subjects |
| mITT_LoC | Modified Intent-to-Treat excluding GCP non-compliant subjects (Loss of |
| | Control) |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomisation & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAFF_ALL | Safety including site including GCP non-compliant subjects |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

#### 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| None | NONMEM |
| _ | SAS |

#### 12.10. Appendix 10: List of Data Displays

All displays (Tables, Figures & Listings) will use the term 'Subjects' instead of "Participants".

#### 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic or Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic or Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 12.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| ETP [1] | End of Treatment Phase Statistical Analysis Complete |
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.10.4. Study Population Tables

| Study F | Population Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | SAFF_ALL | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | ETP, SAC |
| 1.2. | SAFF_ALL | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 1.3. | SAFF_ALL | ES4 | Summary of Subject Disposition at Each Study Epoch | ICH E3 | ETP, SAC |
| 1.4. | ASE | ES6 | Summary of Screening/Run-in Status and Reasons for Screen/Run-in Failure | Journal Requirements | ETP, SAC |
| 1.5. | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | ETP, SAC |
| 1.6. | SAFF_ALL | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | ETP, SAC |
| Protoco | ol Deviation | | | | |
| 1.7. | SAFF_ALL | DV1 | Summary of Important Protocol Deviations | ICH E3 | ETP, SAC |
| 1.8. | SAFF_ALL | IE1 | Summary of Inclusion/ Exclusion Deviations | ICH E3 | ETP, SAC |
| Popula | tion Analysed | | | | |
| 1.9. | Enrolled | SP1 | Summary of Study Populations | IDSL | ETP, SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.10. | SAFF_ALL | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | ETP, SAC |
| 1.11. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | ETP, SAC |
| 1.12. | SAFF_ALL | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | ETP, SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.13. | SAFF_ALL | MH4 | Summary of Current Medical Conditions | ICH E3 | ETP, SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.14. | SAFF_ALL | MH4 | Summary of Past Medical Conditions | ICH E3 | ETP, SAC |
| 1.15. | SAFF_ALL | SP07 | Summary of Family History of Cardiovascular Risk Factors at Screening | | ETP, SAC |
| 1.16. | SAFF_ALL | POP_T01 | Summary of Disease Duration and Exacerbation History | | ETP, SAC |
| 1.17. | SAFF_ALL | SU1 | Summary of Smoking History at Screening | | ETP, SAC |
| 1.18. | SAFF_ALL | CM1 | Summary of Pre-Treatment Concomitant Medications | ICH E3 | ETP, SAC |
| 1.19. | SAFF_ALL | CM1 | Summary of On-Treatment Concomitant Medications | ICH E3 | ETP, SAC |
| 1.20. | SAFF_ALL | CM1 | Summary of Post-Treatment Concomitant Medications | ICH E3 | ETP, SAC |
| 1.21. | SAFF_ALL | CM1 | Summary of On-Treatment Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| 1.22. | SAFF_ALL | CM1 | Summary of Post-Treatment Asthma Concomitant Medications | ICH E3 | ETP, SAC |
| Pre-Trea | atment Lung Fun | ection | | | |
| 1.23. | SAFF_ALL | POP_T02 | Summary of Screening Lung Function | Include Pre- and Post- albuterol (salbutamol) FEV <sub>1</sub> , FVC, FEV <sub>1</sub> /FVC and % Predicted Normal and post-BD at screening %predicted. Include overall and by treatment group. | ETP, SAC |
| 1.24. | SAFF_ALL | POP_T03 | Summary of Baseline Lung Function | FEV <sub>1</sub> , FVC, FEV <sub>1</sub> /FVC and % Predicted Normal. Include overall and by treatment group. | ETP, SAC |
| Exposu | exposure and Treatment Compliance | | | | |
| 1.25. | SAFF_ALL | EX1 | Summary of Exposure and Compliance to Background Therapy (FP and SAL) | ICH E3 | ETP, SAC |

## 12.10.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | ire | | | | |
| 2.1. | SAFF_ALL | EX1 | Summary of Exposure to Study Treatment | ICH E3 | ETP, SAC |
| Prima | ry Endpoint: l | Loss of Asthma | Control Weeks 0-16 | | |
| 2.2. | mITT_LoC | EFF_T01 | Summary of Loss of Asthma Control | Include overall loss of control, each component and the combination of exacerbation or inability to titrate. | ETP, SAC |
| 2.3. | mITT_LoC | EFF_T02 | Summary of Intercurrent Events | | ETP, SAC |
| 2.4. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | | ETP, SAC |
| 2.5. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-16 (Primary Estimand) | | ETP, SAC |
| 2.6. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | | ETP, SAC |
| 2.7. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-16 (Secondary Estimand) | | ETP, SAC |
| Second | lary Endpoint | : Loss of Asthm | a Control Weeks 0-6 | | |
| 2.8. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | | ETP, SAC |
| 2.9. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-6 (Primary Estimand) | | ETP, SAC |
| 2.10. | mITT_LoC | EFF_T03 | Bayesian Analysis of Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | | ETP, SAC |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | mITT_LoC | EFF_T04 | Frequentist Analysis of Loss of Asthma Control Over Weeks 0-6 (Secondary Estimand) | | ETP, SAC |
| Second | dary Endpoint | s: Components | of Loss of Asthma Control | | |
| 2.12. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an ACQ increase from Baseline >= 0.5 (Primary Estimand) | | ETP, SAC |
| 2.13. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an ACQ increase from Baseline >= 0.5 (Secondary Estimand) | | ETP, SAC |
| 2.14. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an FEV1 decrease from Baseline > 7.5% (Primary Estimand) | | ETP, SAC |
| 2.15. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an FEV1 decrease from Baseline > 7.5% (Secondary Estimand) | | ETP, SAC |
| 2.16. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an Inability to Titrate According to the Pre-Defined Schedule (Primary Estimand) | | ETP, SAC |
| 2.17. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with an Inability to Titrate According to the Pre-Defined Schedule (Secondary Estimand) | | ETP, SAC |
| 2.18. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with a Significant Asthma Exacerbation (Primary Estimand) | | ETP, SAC |
| 2.19. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with a Significant Asthma Exacerbation (Secondary Estimand) | | ETP, SAC |
| 2.20. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with a Significant Asthma Exacerbation or Inability to Titrate According to the Pre-Defined Schedule (Primary Estimand) | | ETP, SAC |
| 2.21. | mITT_LoC | EFF_T03 | Analysis of Proportion of Subjects with a Significant Asthma Exacerbation or Inability to Titrate According to the Pre-Defined Schedule (Secondary Estimand) | | ETP, SAC |

| Effica | cy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | dary Endpoint | ts: Time to Loss | of Asthma Control | | |
| 2.22. | mITT_LoC | EFF_T05 | Summary and Analysis of Time to Loss of Asthma Control (Primary Estimand) | | ETP, SAC |
| 2.23. | mITT_LoC | EFF_T05 | Summary and Analysis of Time to Loss of Asthma Control (Secondary Estimand) | | ETP, SAC |
| Second | lary Endpoint | ts: Hospitalisatio | on and Emergency Room Visits | | |
| 2.24. | mITT | EFF_T06 | Summary and Rate of Asthma-Related On-Treatment<br>Hospitalisations and Emergency Room Visits (Primary<br>Estimand) | | ETP, SAC |
| Second | lary Endpoint | :: ACQ-5 | | | |
| 2.25. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in ACQ-5 Total Score (Primary Estimand) | | ETP, SAC |
| 2.26. | mITT | EFF_T04 | Analysis of Proportion of Subjects with an ACQ-5 Total Score increase from Baseline >= 0.5 (Primary Estimand) | | ETP, SAC |
| 2.27. | mITT | EFF_T04 | Analysis of Proportion of Subjects with an ACQ-5 Total Score increase from Baseline >= 0.5 (Secondary Estimand) | | ETP, SAC |
| Second | lary Endpoint | :: SGRQ | | | |
| 2.28. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in SGRQ Total Score (Primary Estimand) | | ETP, SAC |
| 2.29. | mITT | EFF_T04 | Analysis of Proportion of Subjects with an SGRQ Total Score increase from Baseline >= 4 (Primary Estimand) | | ETP, SAC |
| 2.30. | mITT | EFF_T04 | Analysis of Proportion of Subjects with an SGRQ Total Score decrease from Baseline >= 4 (Secondary Estimand) | | ETP, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | lary Endpoint | : FEV <sub>1</sub> and PEI | F | | |
| 2.31. | mITT | EFF_T07 | Summary of Raw and Change from Baseline FEV <sub>1</sub> (Primary Estimand) | | ETP, SAC |
| 2.32. | mITT | EFF_T08 | Analysis of Change from Baseline in FEV <sub>1</sub> up to Week 4(Primary Estimand) | | ETP, SAC |
| 2.33. | mITT | EFF_T07 | Summary of Raw and Change from Baseline Fractional Exhaled Nitric Oxide (FeNO) (Primary Estimand) | | ETP, SAC |
| 2.34. | mITT | EFF_T08 | Analysis of Change from Baseline in Fractional Exhaled Nitric Oxide (FeNO) up to Week 4 (Primary Estimand) | | ETP, SAC |
| Second | lary Endpoint | : Exacerbations | | | |
| 2.35. | mITT | EFF_T09 | Summary of On-Treatment Asthma Exacerbations | | ETP, SAC |
| Second | lary Endpoint | : Eosinophils | | | |
| 2.36. | mITT | EFF_T07 | Summary of Raw and Change from Baseline in Eosinophils (Primary Estimand) | | ETP, SAC |
| 2.37. | mITT | EFF_T08 | Analysis of Eosinophils (Primary Estimand) | | ETP, SAC |
| Second | lary Endpoint | : PEF, Daytime | Symptom Score, Night-time Symptom Score and Rescue | Medication | |
| 2.38. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Morning Peak Expiratory Flow (PEF) | | ETP, SAC |
| 2.39. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Evening Peak Expiratory Flow (PEF) | | ETP, SAC |
| 2.40. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Daytime Asthma Symptom Score | | ETP, SAC |
| 2.41. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Night-Time<br>Awakenings Due to Asthma Symptoms | | ETP, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.42. | mITT | EFF_T010 | Summary of Raw and Change from Baseline in Mean Rescue Medication use (Albuterol/Salbutamol) | | ETP, SAC |

# 12.10.6. Efficacy Figures

| Efficacy | r: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Endpoint: Los | ss of Asthma Con | trol | | |
| 2.1 | mITT_LoC | | Plot of Loss of Asthma Control (Primary Estimand) | Include Show overall and components of loss on control | ETP, SAC |
| 2.2 | mITT_LoC | | Plot of Loss of Asthma Control (Secondary Estimand) | Include Show overall and components of loss on control | ETP, SAC |
| Second | ary Endpoint: | Time to Loss of C | ontrol | | |
| 2.1. | mITT_LoC | | Kaplan-Meir Plot of Time to Loss of Asthma Control (Primary Estimand) | | ETP, SAC |
| 2.2. | mITT_LoC | | Kaplan-Meir Plot of Time to Loss of Asthma Control (Secondary Estimand) | | ETP, SAC |
| Second | ary Endpoint: | Eosinophils | | | |
| 2.3. | mITT_LoC | | Cumulative Density Plot of Eosinophils | | ETP, SAC |
| 2.4. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.5. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.6. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.7. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs Eosinophils – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.8. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.9. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.10. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 2.11. | mITT_LoC | | Loss of Control Over Weeks 0-6 vs Eosinophils – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| Seconda | ary Endpoints: | IgE and FeNO Ov | ver Weeks 0-16 | <u>, </u> | |
| 2.12. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE by Treatment - Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.13. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.14. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 2.15. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs IgE – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.16. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 2.17. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO – Fractional Polynomial Treatment Difference (Primary Estimand) | | ETP, SAC |
| 2.18. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | mITT_LoC | | Loss of Control Over Weeks 0-16 vs FeNO – Fractional Polynomial Treatment Difference (Secondary Estimand) | | ETP, SAC |
| 2.20. | mITT | | FEV1 at Week 4 vs Eosinophils by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.21. | mITT | | FEV1 at Week vs Eosinophils – Fractional Polynomial Treatment Difference | | ETP, SAC |
| 2.22. | mITT | | FEV1 at Week 4 vs IgE by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.23. | mITT | | FEV1 at Week vs IgE – Fractional Polynomial Treatment Difference | | ETP, SAC |
| 2.24. | mITT | | FEV1 at Week 4 vs FeNO by Treatment – Fractional Polynomial Model | | ETP, SAC |
| 2.25. | mITT | | FEV1 at Week vs FeNO – Fractional Polynomial Treatment Difference | | ETP, SAC |

## 12.10.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events (AEs) | | | | |
| 3.1. | SAFF_ALL | SAFE_T01 | Overview of On-treatment Adverse Events During the Study | | ETP, SAC |
| 3.2. | SAFF_ALL | AE1 | Summary of All Pre-treatment Adverse Events by System Organ Class and Preferred Term | | ETP, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.4. | SAFF_ALL | AE1 | Summary of All Post-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.5. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.6. | SAFF_ALL | AE1 | Summary of All On-treatment Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.7. | SAFF_ALL | AE1 | Summary of All On-treatment Fatal Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.8. | SAFF_ALL | AE3 | Summary of All On-treatment Common (>=3%) Adverse Events by Overall Frequency | ICH E3 | ETP, SAC |
| 3.9. | SAFF_ALL | AE1 | Summary of All On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.10. | SAFF_ALL | AE15 | Summary of All On-treatment Common (>=3%) Non-serious<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | FDAAA, EudraCT | ETP, SAC |
| 3.11. | SAFF_ALL | AE1 | Summary of All Pre-treatment Serious Adverse Events by System Organ Class and Preferred Term | | ETP, SAC |
| 3.12. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | ICH E3 | ETP, SAC |
| 3.13. | SAFF_ALL | AE1 | Summary of All Post-treatment Serious Adverse Events by System Organ Class and Preferred Term | ICH E3 | ETP, SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.14. | SAFF_ALL | AE16 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Participants and Occurrences) | FDAAA, EudraCT | ETP, SAC |
| 3.15. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term | IDSL | ETP, SAC |
| 3.16. | SAFF_ALL | AE1 | Summary of All On-treatment Serious Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | IDSL | ETP, SAC |
| Advers | e Events of Sp | ecial Interest (AES | Sis) | | |
| 3.17. | SAFF_ALL | AE1 | Summary of On-treatment Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.18. | SAFF_ALL | AE1 | Summary of On-treatment Serious Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.19. | SAFF_ALL | AE1 | Summary of Post-treatment Adverse Events of Special Interest | IDSL | ETP, SAC |
| 3.20. | SAFF_ALL | AE1 | Summary of Post-treatment Serious Adverse Events of Special Interest | IDSL | ETP, SAC |
| Mexico | Specific Table | S | | | |
| 3.21. | SAFF_ALL | | Summary of Suspected Investigational Product Adverse Reaction (Mexican Participants Only) | | ETP, SAC |
| 3.22. | SAFF_ALL | | Summary of Suspected Investigational Product Adverse Reaction (Non-Mexican Participants) | | ETP, SAC |
| Labora | tory: Chemistry | / | | | |
| 3.23. | SAFF_ALL | LB1 | Summary of Clinical Chemistry | ICH E3 | ETP, SAC |
| 3.24. | SAFF_ALL | LB1 | Summary of Change from Baseline in Clinical Chemistry | ICH E3 | ETP, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.25. | SAFF_ALL | LB16 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | ETP, SAC |
| Labora | tory: Hematolo | gy and Cardiac M | arkers | | · |
| 3.26. | SAFF_ALL | LB1 | Summary of Hematology and Cardiac Markers | ICH E3 | ETP, SAC |
| 3.27. | SAFF_ALL | LB1 | Summary of Changes from Baseline in Hematology and Cardiac Markers | ICH E3 | ETP, SAC |
| 3.28. | SAFF_ALL | LB16 | Summary of Worst Case Hematology and Cardiac Markers<br>Results Relative to Normal Range Post-Baseline Relative to<br>Baseline | ICH E3 | ETP, SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | · |
| 3.29. | SAFF_ALL | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | ETP, SAC |
| 3.30. | SAFF_ALL | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | ETP, SAC |
| ECG | • | | | | • |
| 3.31. | SAFF_ALL | | Summary of Antihistamine, Decongestant and Caffeine Use Prior to ECG assessments | | ETP, SAC |
| 3.32. | SAFF_ALL | EG1 | Summary of ECG Findings | IDSL | ETP, SAC |
| 3.33. | SAFF_ALL | EG2 | Summary of ECG Values by Visit | IDSL | ETP, SAC |
| 3.34. | SAFF_ALL | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | ETP, SAC |
| 3.35. | SAFF_ALL | EG10 | Summary of Maximum QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | ETP, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.36. | SAFF_ALL | EG11 | Summary of Maximum Increase in QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | ETP, SAC |
| Holter | | | | | |
| 3.37. | SAFF_ALL | HM1 | Summary of Holter Interpretations | IDSL | ETP, SAC |
| 3.38. | SAFF_ALL | HM2 | Summary of Holter Abnormalities | IDSL | ETP, SAC |
| 3.39. | SAFF_ALL | HM3 | Summary of Holter Values | IDSL | ETP, SAC |
| 3.40. | SAFF_ALL | HM3 | Summary of Change from Baseline in Holter Values | IDSL | ETP, SAC |
| 3.41. | SAFF_ALL | HM4 | Summary of Subjects with R-on-T Beats | IDSL | ETP, SAC |
| Vital Sig | gns | | | | |
| 3.42. | SAFF_ALL | VS1 | Summary of Vital Signs | ICH E3 | ETP, SAC |
| 3.43. | SAFF_ALL | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | ETP, SAC |
| 3.44. | SAFF_ALL | VS1 | Summary of Change from Pre-dose to Post-dose in Vital Signs | ICH E3 | ETP, SAC |

#### 12.10.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | |
|---|---|---|---|
| No. Population IDSL / Example Shell Title Programming Notes Deliverabl [Priority] | | | |
| Second | Secondary: Pharmacokinetic | | |
| 4.1. | PK | Summary of PK Serum Concentrations | SAC only |

## 12.10.9. Pharmacodynamic and Biomarker Tables

| rnanni | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | dary: Pharmaco | dynamic | | | |
| 6.1. | mITT | | Summary of Raw and Percentage Change from Baseline in Free Soluble ST2 concentration (ng/mL) (On-treatment) | Pre and Post dose. | ETP, SAC |
| 6.2. | mITT | | Analysis of Percentage Change from Baseline in Free Soluble ST2 concentration (ng/mL) (On-treatment) | Pre dose only. | ETP, SAC |
| 6.3. | mITT | | Summary of Raw and Percentage Change from Baseline in Free soluble ST2 concentration (ng/mL) (Post-treatment) | | ETP, SAC |
| 6.4. | mITT | | Analysis of Percentage Change from Baseline in Free soluble ST2 concentration (ng/mL) (Post-treatment) | | ETP, SAC |
| 6.5. | mITT | | Summary of Raw and Change from Baseline in Total Soluble ST2 concentration (ng/mL) (On-treatment) | Pre and Post dose. | ETP, SAC |
| 6.6. | mITT | | Analysis of Change from Baseline in Total Soluble ST2 concentration (ng/mL) (On-treatment) | Pre dose only. | ETP, SAC |
| 6.7. | mITT | | Summary of Raw and Change from Baseline in Total Soluble ST2 concentration (ng/mL) (Post-treatment) | | ETP, SAC |
| 6.8. | mITT | | Analysis of Change from Baseline in Total Soluble ST2 concentration (ng/mL) (Post-treatment) | | ETP, SAC |
| Explora | atory: Biomark | ers | | | |
| 6.9. | mITT | | Summary and Change from Baseline in Induced Sputum Biomarkers (subset) at Weeks 8 and 16 | Include geometric mean and %CV | ETP, SAC |
| 6.10. | mITT | | Summary and Change from Baseline in Exploratory Serum Markers at Weeks 8 and 16 | Include geometric mean and %CV | ETP, SAC |

# 12.10.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | Secondary: Pharmacokinetic | | | | |
| 6.1. | PK | | Plot of Serum Concentrations | | ETP, SAC |
| 6.2. | PK | | Pre-dose Trough Concentration vs Eosinophils at Week 4 | | ETP, SAC |
| 6.3. | PK | | Pre-dose Trough Concentration vs FeNO at Week 4 | | ETP, SAC |
| 6.4. | PK | | Pre-dose Trough Concentration vs IgE at Week 4 | | ETP, SAC |

# 12.10.11. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Secondary: Pharmacokinetic | | | | | |
| 6.5. | mITT | | Plot of Percentage Change from Baseline in Free Soluble ST2 levels (On-treatment) | | ETP, SAC |
| 6.6. | mITT | | Plot of Percentage Change from Baseline in Free soluble ST2 levels (Post-treatment) | | ETP, SAC |
| 6.7. | mITT | | Plot of Change from Baseline in Total Soluble ST2 levels (Ontreatment) | | ETP, SAC |
| 6.8. | mITT | | Plot of Change from Baseline in Total Soluble ST2 levels (Post-treatment) | | ETP, SAC |
| 6.9. | mITT_LoC | | Loss of Control vs Free soluble ST2 by Treatment – Fractional Polynomial Model (Primary Estimand) | | ETP, SAC |
| 6.10. | mITT_LoC | | Loss of Control vs Free soluble ST2 Treatment Difference – Fractional Polynomial (Primary Estimand) | | ETP, SAC |
| 6.11. | mITT_LoC | | Loss of Control vs Free soluble ST2 by Treatment – Fractional Polynomial Model (Secondary Estimand) | | ETP, SAC |
| 6.12. | mITT_LoC | | Loss of Control vs Free soluble ST2 Treatment Difference – Fractional Polynomial (Secondary Estimand) | | ETP, SAC |

## 12.10.12. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen and Run-in Failure | Journal Guidelines | ETP, SAC |
| 2. | SAFF_ALL | ES2 / ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | ETP, SAC |
| 3. | SAFF_ALL | SD2/SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | ETP, SAC |
| 4. | SAFF_ALL | BL1 / BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | ETP, SAC |
| 5. | SAFF_ALL | TA1 / CP_RD1x | Listing of Planned and Actual Treatments | IDSL | ETP, SAC |
| Protoc | ol Deviations | | | , | |
| 6. | SAFF_ALL | DV2 | Listing of Important Protocol Deviations | ICH E3 | ETP, SAC |
| 7. | SAFF_ALL | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | ETP, SAC |
| 8. | SAFF_ALL | | Listing of Subjects excluded for GCP non-compliance | | |
| Popula | tions Analysed | | | | • |
| 9. | SAFF_ALL | SP3 | Listing of Participants Excluded from Any Population | ICH E3. | ETP, SAC |
| Demog | raphic and Bas | eline Characterist | tics | · | |
| 10. | SAFF_ALL | DM2 | Listing of Demographic Characteristics | ICH E3 | ETP, SAC |
| 11. | SAFF_ALL | DM9 | Listing of Race | ICH E3 | ETP, SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | Prior and Concomitant Medications | | | | |
| 12. | SAFF_ALL | CP_CM3 | Listing of Concomitant Medications | IDSL | ETP, SAC |
| Exposi | ire and Treatmo | ent Compliance | | | |
| 13. | SAFF_ALL | EX3 | Listing of Exposure Data | ICH E3 | ETP, SAC |
| Advers | e Events | | | | |
| 14. | SAFF_ALL | AE8 | Listing of All Adverse Events | ICH E3 | ETP, SAC |
| 15. | SAFF_ALL | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | ETP, SAC |
| 16. | SAFF_ALL | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 17. | SAFF_ALL | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | ETP, SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 18. | SAFF_ALL | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | ETP, SAC |
| 19. | SAFF_ALL | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | ETP, SAC |
| 20. | SAFF_ALL | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | ETP, SAC |
| 21. | SAFF_ALL | AE8 | Listing of Serious Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | ETP, SAC |
| 22. | SAFF_ALL | AE8 | Listing of Other Significant Adverse Events | ICH E3 | ETP, SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hepato | Hepatobiliary (Liver) | | | | |
| 23. | SAFF_ALL | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | ETP, SAC |
| 24. | SAFF_ALL | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | ETP, SAC |
| All Lab | oratory | | | | |
| 25. | SAFF_ALL | LB5 / LB6 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | ETP, SAC |
| 26. | SAFF_ALL | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | ETP, SAC |
| ECG | | | | | |
| 27. | SAFF_ALL | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | ETP, SAC |
| 28. | SAFF_ALL | EG5 | Listing of Abnormal ECG Findings | IDSL | ETP, SAC |
| Holter | | | | | |
| 29. | SAFF_ALL | MH6 | Listing of Holter R-on-T Beat Data | IDSL | ETP, SAC |
| 30. | SAFF_ALL | MH7 | Listing of Holter {Supraventricular} {Ventricular} Event Data | IDSL, Update title as appropriate based on data | ETP, SAC |
| 31. | SAFF_ALL | MH8 | Listing of Holter {Sustained} {Non-sustained} {Supraventricular} {Ventricular} Run | IDSL, Update title as appropriate based on data | ETP, SAC |
| 32. | SAFF_ALL | MH9 | Listing of Holter Atrial {Fibrillation} {Flutter} Data | IDSL, Update title as appropriate based on data | ETP, SAC |
| 33. | SAFF_ALL | MH10 | Listing of Holter Abnormalities | IDSL | ETP, SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 34. | SAFF_ALL | VS4 | Listing of All Vital Signs Data | IDSL | ETP, SAC |
| Primary | Analysis Data | : Loss of Asthma | Control and Intercurrent Events | | |
| 35. | mITT_LoC | | Listing of Loss of Asthma Control | Include all reasons for loss of control and time to loss of asthma control | ETP, SAC |
| 36. | mITT_LoC | | Listing of Intercurrent Events | Include treatment subject was analysed as taking and treatment at time of loss of control | ETP, SAC |

## 12.10.13. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study I | Population | | | | |
| 37. | SAFF_ALL | SP2 | Listing of the Follow-up Contact | | ETP, SAC |
| 38. | SAFF_ALL | TA1 | Listing of Treatment Misallocations | Change Centre ID to Investigator ID: xxxxxx and also Investigator at Centre: xxxxxx | ETP, SAC |
| 39. | SAFF_ALL | SP4 | Listing of Overall Percentage Treatment Compliance | | ETP, SAC |
| Second | dary Efficacy | | | | |
| 40. | mITT | | Listing of Eosinophils | Include randomisation and analysis strata | ETP, SAC |
| 41. | mITT | SP10 | Listing of Lung Function Results including FEV <sub>1</sub> | | ETP, SAC |
| 42. | mITT | S3 | Listing of Asthma Exacerbations | Include a column for severity | ETP, SAC |
| 43. | mITT | | Listing of Asthma Control Questionnaire (ACQ-5) | | ETP, SAC |
| 44. | mITT | | Listing of St George's Respiratory Questionnaire (SGRQ) | | ETP, SAC |
| 45. | mITT | | Listing of Peak Exploratory Flow (PEF) | | ETP, SAC |
| 46. | mITT | | Listing of Fractional Exhaled Nitric Oxide (FeNO) | | ETP, SAC |
| 47. | mITT | | Listing of Daytime and Night-time Asthma Symptoms | | ETP, SAC |
| 48. | mITT | | Listing of Rescue Medication Use | | ETP, SAC |
| 49. | mITT | | Listing of Hospitalisations and Emergency Room Visits | | ETP, SAC |
| 50. | PK | | Listing of Serum Concentration | | SAC Only |
| 51. | PD | | List of Free and Total Soluble ST2 Levels | | |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | • | |
| 52. | SAFF_ALL | | Listing of Clinical Chemistry | | ETP, SAC |
| 53. | SAFF_ALL | | Listing of Haematology and Cardiac Markers | | ETP, SAC |
| 54. | SAFF_ALL | | Listing of Anti-GSK3772847 Antibodies | | ETP, SAC |
| 55. | SAFF_ALL | ESI8 | Listing of AE Terms of Special Interest | IDSL | ETP, SAC |
| Explor | atory Biomarke | r | | | |
| 56. | mITT | | Listing of Induced Sputum and Exploratory Serum Biomarkers | | ETP, SAC |
| Medica | l History | | | | |
| 57. | SAFF_ALL | MH2 | Listing of Medical Conditions at Screening | | ETP, SAC |
| 58. | SAFF_ALL | SP5 | Listing of Family History of Cardiovascular Risk Factors | | ETP, SAC |
| 59. | SAFF_ALL | SP6 | Listing of Asthma History | | ETP, SAC |
| 60. | SAFF_ALL | SP7 | Listing of Smoking History and Smoking Status | | ETP, SAC |
| 61. | SAFF_ALL | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text for Bone Mineral Density and Other Medications | | ETP, SAC |
| Liver E | vents: Note on | ly produced if the | re is a Liver Event | | |
| 62. | SAFF_ALL | VS4 | Listing of Liver Events | | ETP, SAC |
| 63. | SAFF_ALL | VS4 | Listing of Liver Event Information for RUCAM Score | | ETP, SAC |
| 64. | SAFF_ALL | VS4 | Listing of Liver Biopsy | | ETP, SAC |
| 65. | SAFF_ALL | VS4 | Listing of Liver Imaging Details | | ETP, SAC |
| Cardio | vascular Events | s: Note only produ | uced if there is a Cardiovascular Event | | |
| 66. | SAFF_ALL | VS4 | Listing of Myocardial infarction/unstable angina | | ETP, SAC |
| 67. | SAFF_ALL | VS4 | Listing of Congestive heart failure | | ETP, SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 68. | SAFF_ALL | VS4 | Listing of Arrhythmias | | ETP, SAC |
| 69. | SAFF_ALL | VS4 | Listing of Valvulopathy | | ETP, SAC |
| 70. | SAFF_ALL | VS4 | Listing of Pulmonary hypertension | | ETP, SAC |
| 71. | SAFF_ALL | VS4 | Listing of Cerebrovascular events/stroke and transient ischemic attack | | |
| 72. | SAFF_ALL | VS4 | Listing of Peripheral arterial thromboembolism | | |
| 73. | SAFF_ALL | VS4 | Listing of Deep venous thrombosis/pulmonary embolism | | |
| 74. | SAFF_ALL | VS4 | Listing of Revascularisation | | |
| 75. | SAFF_ALL | VS4 | Listing of Deaths | | |

## 12.11. Appendix 11: Example Mock Shells for Data Displays

Available upon request